## **Statistical Analysis Plan**

**Study ID:** 213360 (PR-30-5020-C)

**Official Title of Study:** A Phase 2, Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of Niraparib in Patients with Advanced, Relapsed, High-Grade Serous Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Who Have Received Three or Four Previous Chemotherapy Regimens

**Date of Document:** 21-JUL-2021

#### STATISTICAL ANALYSIS PLAN

A Phase 2, Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of Niraparib in Patients with Advanced, Relapsed, High-Grade Serous Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Who Have Received Three or Four Previous Chemotherapy Regimens

### Protocol PR-30-5020-C

Protocol Number: PR-30-5020-C

Protocol Version and Date: Version 8.0: 21 December 2017 (Amendment 5)

Version 7.0: 07 April 2017 (Amendment 4)

Version 6.0: 14 September 2016 (Amendment 3.2) Version 5.0: 07 September 2016 (Amendment 3.1)

Version 4.0: 29 July 2016 (Amendment 3) Version 3.0: 24 May 2016 (Amendment 2) Version 2.0: 30 October 2015 (Amendment 1) Version 1.0: 17 December 2014 (Original)

Name of Test Drug: Niraparib ([3S]-3-[4-{7-(aminocarbonyl)-2H-indazol-2-yl}

phenyl] piperidine [tosylate monohydrate salt])

Phase: Phase 2

Methodology: Open-Label, Single-Arm

Sponsor: TESARO, Inc.

1000 Winter Street Waltham MA 02451

Tel: PPD

Sponsor Representative: Romnee Clark, MD

Senior Medical Director

Analysis Plan Date: 21 July 2021

Analysis Plan Version: Version 4.0

### **Confidentiality Statement**

The information contained herein is confidential and the proprietary property of TESARO, Inc., and any unauthorized use or disclosure of such information without the prior written authorization of TESARO, Inc., is expressly prohibited.


# APPROVAL SIGNATURE PAGE

| Protocol Title: | A Phase 2, Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of Niraparib in Patients with Advanced, Relapsed, High-Grade Serous Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Who Have Received Three or Four Previous Chemotherapy Regimens |
|---|---|
| Protocol Number: PR-30-5020-C | |
| Sponsor: | TESARO, Inc.<br>1000 Winter Street<br>Waltham MA 02451 |
| Author: | Veristat, LLC<br>118 Turnpike Road<br>Southborough, MA 01772 |
| Author Signatory: | |
| PPD | Signature: |
| Principal Biostatisti | cian Date: |
| Sponsor Approval: | |
| the planned statistic<br>analyses are approp<br>are consistent with t | ament, I acknowledge that I have read the document and approve of all analyses described herein. I agree that the planned statistical riate for this study, are in accordance with the study objectives, and the statistical methodology described in the protocol, clinical and all applicable regulatory guidances and guidelines. |
| I have discussed any biostatistical author | y questions I have regarding the contents of this document with the |
| described herein, ma | at any subsequent changes to the planned statistical analyses, as ay have a regulatory impact and/or result in timeline adjustments. All ned analyses will be described in the clinical study report. |
| Sponsor Signatory: | |
| Romnee Clark, MD | |
| Senior Medical Dire | Date: |
| Yong Li, PhD | Signature: |
| Director, Biostatisti | cs Date: |


# TABLE OF CONTENTS

| 1. | INFC | RMATIC | ON FROM THE STUDY PROTOCOL | 10 |
|---|---|---|---|---|
| | 1.1. | Introdu | ction and Objectives | 10 |
| | | 1.1.1. | Introduction | 10 |
| | | 1.1.2. | Study Objectives | 10 |
| | 1.2. | Study I | Design | 12 |
| | | 1.2.1. | Synopsis of Study Design | 12 |
| | | 1.2.2. | Randomization Methodology | 13 |
| | | 1.2.3. | Stopping Rules and Unblinding | 13 |
| | | 1.2.4. | Study Procedures | 13 |
| | | 1.2.5. | Efficacy, Pharmacokinetic, and Safety Parameters | 17 |
| | | | 1.2.5.1. Efficacy Parameters | 17 |
| | | | 1.2.5.2. Pharmacokinetic Parameters | 17 |
| | | | 1.2.5.3. Safety Parameters | 17 |
| 2. | PATI | ENT PO | PULATION | 19 |
| | 2.1. | Populat | tion Definitions | 19 |
| | 2.2. | Protoco | ol Deviations | 19 |
| 3. | GEN | ERAL ST | TATISTICAL METHODS | 20 |
| | 3.1. | Sample Size Justification | | |
| | 3.2. | General Methods | | |
| | 3.3. | Computing Environment | | |
| | 3.4. | Baseline Definitions | | |
| | 3.5. | Methods of Pooling Data | | |
| | 3.6. | Adjustments for Covariates | | |
| | 3.7. | Multipl | Multiple Comparisons/Multiplicity | |
| | 3.8. | | | |
| | | 3.8.1. | Prior Lines of Chemotherapy | 22 |
| | | 3.8.2. | Response to the Last Platinum-Based Therapy | 23 |
| | | 3.8.3. | Prior PARP Treatment | 23 |
| | | 3.8.4. | Biomarker Subpopulations | 23 |
| | | | 3.8.4.1. Biomarker Definitions | 23 |
| | | | 3.8.4.2. Study-Specific Biomarker Populations | 24 |


| | 3.9. | Withdra | awals, Drop | oouts, Loss to Follow-up | 25 |
|---|---|---|---|---|---|
| | 3.10. | Missing | g Data | | 25 |
| | 3.11. | Visit W | indows | | 26 |
| | 3.12. | Admini | strative Int | erim Analyses | 26 |
| 4. | STUD | Y ANAI | LYSES | | 27 |
| | 4.1. | Patient | Disposition | 1 | 27 |
| | 4.2. | Demog | raphics, Ba | seline Characteristics, and Medical History | 27 |
| | 4.3. | Efficac | y Evaluatio | n | 28 |
| | | 4.3.1. | | Variables for Primary and Key Secondary | 28 |
| | | 4.3.2. | Secondar | y Efficacy Variables | 32 |
| | | | 4.3.2.1. | Duration of Response | 32 |
| | | | 4.3.2.2. | Disease Control Rate | 33 |
| | | | 4.3.2.3. | Progression-Free Survival | 33 |
| | | | 4.3.2.4. | Time to First Subsequent Therapy | 34 |
| | | | 4.3.2.5. | Overall Survival | 34 |
| | | | 4.3.2.6. | Pharmacokinetic Evaluations | 34 |
| | 4.4. | Safety A | Analyses | | 34 |
| | | 4.4.1. | Study Tr | eatment Exposure | 34 |
| | | 4.4.2. | Study Tr | eatment Compliance | 35 |
| | | 4.4.3. | Adverse | Events | 36 |
| | | | 4.4.3.1. | Overview | 36 |
| | | | 4.4.3.2. | Adverse Events of Special Interest | 38 |
| | | | 4.4.3.3. | Other Adverse Events of Interest | 39 |
| | | | | Examination of Adverse Events Controlling Duration of Drug Exposure | |
| | | | 4.4.3.5. | Examination of Duration of Adverse Events | 41 |
| | | 4.4.4. | Laborato | ry Data | 41 |
| | | 4.4.5. | Vital Sig | ns and Physical Examination | 42 |
| | | 4.4.6. | Electroca | ırdiogram | 42 |
| | | 4.4.7. | Concomi | tant Medications | 43 |
| 5. | CHAN | NGES TO | ) PLANNE | D ANALYSES | 45 |
| 6 | REEE | RENCES | 2 | | 16 |


| 7. | APPI | ENDIX | 47 |
|----|------|-------------------------------------------------------|-----|
| | 7.1. | MedDRA Preferred Terms for Adverse Events of Speci | |
| | 7.2. | | |
| | 7.3. | SMQ Terms for Pregnancy and Neonatal Topics | 136 |
| | 7.4. | SMQ Terms for Hypertension | 207 |
| | 7.5. | List of Per-Protocol Chemotherapy Regimens in Preferr | |
| 8. | STA | TISTICAL OUTPUT SHELLS | 216 |
| 9. | REV | ISION HISTORY | 217 |


# TABLES INCLUDED IN THE TEXT

| Table 1-1 | Schedule of Assessments. | 14 |
|---|---|---|
| Table 3-1 | Evaluation Intervals | 26 |
| Table 4-1 | Overall Response for Patients with Measureable Disease at Study Entry | 29 |
| Table 4-2: | Best Overall Response when Confirmation of CR and PR Required | 30 |
| Table 4-3: | Censoring Rules used in Duration of Response Analysis | 32 |
| Table 4-4: | Censoring Rules used in Progression-Free Survival Analysis | 33 |
| Table 4-5: | Adverse Events of Special Interest and Other Grouped Events | 40 |


# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation | Definition |
|----------------------|-------------------------------------------------------|
| AE | Adverse event |
| AESI | Adverse event(s) of special interest |
| ALT | Alanine aminotransferase |
| AML | Acute myeloid leukemia |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BER | Base excision repair |
| BMI | Body mass index |
| BRCA | Breast cancer gene |
| CA-125 | Cancer antigen 125 |
| CBC | Complete blood count |
| CI | Confidence interval |
| CR | Complete response |
| CSR | Clinical study report |
| CT | Computed tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DCR | Disease control rate |
| DNA | Deoxyribonucleic acid |
| DOR | Duration of response |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic case report form |
| EOT | End of treatment |
| FDA | (United States) Food and Drug Administration |
| FIGO | International Federation of Gynecology and Obstetrics |
| FISH | Fluorescence in situ hybridization |
| gBRCA <sup>mut</sup> | Germline breast cancer gene mutation |
| GCIG | Gynecologic Cancer Intergroup |
| GCP | Good Clinical Practice |
| GGT | Gamma glutamyl transferase |
| $H_0$ | Null hypothesis |
| $H_1$ | Alternative hypothesis |
| HEENT | Head, Eyes, Ears, Neck, and Throat |
| HRD | Homologous recombination deficiency |
| ICF | Informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |


| Abbreviation | Definition |
|---|---|
| IRB | Institutional Review Board |
| ITT | Intent-to-treat |
| KM | Kaplan-Meier |
| LLN | Lower limit of normal |
| MDS | Myelodysplastic syndrome |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic resonance imaging |
| NCI | National Cancer Institute |
| ORR | Objective response rate |
| OS | Overall survival |
| PARP | Poly(ADP-ribose) polymerase |
| PD | Progressive disease (in the context of disease evaluation) or protocol deviation |
| PEY | Patient-exposure year |
| PFI | Platinum-free interval |
| PFS | Progression-free survival |
| PK | Pharmacokinetic |
| PP | Per-protocol |
| PR | Partial response |
| PT | Preferred Term (MedDRA) |
| $Q_1$ | First quartile |
| $Q_3$ | Third quartile |
| QD | Once daily |
| QTc | QT interval corrected for heart rate |
| QTcB | QT interval corrected for heart rate using Bazett's formula |
| QTcF | QT interval corrected for heart rate using Fridericia's formula |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE | Serious adverse event |
| SAF | Safety |
| SAP | Statistical analysis plan |
| sBRCA <sup>mut</sup> | Somatic breast cancer gene mutation |
| SD | Stable disease (in the context of disease evaluation) or standard deviation (in the context of statistics) |
| SOC | System Organ Class (MedDRA) |
| tBRCAmut | Tumor breast cancer gene mutation |
| tBRCAwt | Tumor breast cancer gene wild-type |
| TEAE | Treatment-emergent adverse event |
| TFST | Time to first subsequent therapy |
| ULN | Upper limit of normal |


| Abbreviation | Definition |
|--------------|-------------------------------------------|
| WHO | World Health Organization |
| WHODD | World Health Organization Drug Dictionary |


### 1. INFORMATION FROM THE STUDY PROTOCOL

## 1.1. Introduction and Objectives

#### 1.1.1. Introduction

Niraparib is a potent, orally active poly(ADP-ribose) polymerases (PARP)-1 and -2 inhibitor being developed as an agent for tumors with defects in the homologous recombination deoxyribonucleic acid (DNA) repair pathway or that are driven by PARP-mediated transcription factors.

PARP-1 and -2 are zinc-finger DNA-binding enzymes that play a crucial role in DNA repair. Upon formation of DNA breaks, PARP binds at the end of broken DNA strands, a process that activates its enzymatic activity. Activated PARP catalyzes addition of long polymers of ADP-ribose onto PARP and several other proteins associated with chromatin, including histones and various DNA repair proteins. This results in chromatin relaxation, fast recruitment of DNA repair proteins, and efficient repair of DNA breaks. In this manner, PARP plays a key role in sensing DNA damage and converting it into intracellular signals that activate the base excision repair (BER) and single-strand break repair pathways.

Clinical studies have shown that PARP inhibitors are active for recurrent ovarian cancer.[1, 2, 3, 4, 5, 6, 7] Clinical anti-cancer activity has been observed in patients with and without germline breast cancer gene (BRCA) mutation (gBRCA<sup>mut</sup>) and in patients who are platinum-sensitive and platinum-resistant. PARP inhibition appears to be most active in patients with gBRCA<sup>mut</sup> platinum-sensitive disease.[1, 3, 5] Additionally, maintenance therapy in patients with relapsed, platinum-sensitive ovarian cancer appears promising, [6] Of patients with a BRCA mutation, median progression-free survival (PFS) was significantly longer in the PARP inhibitor group than in the placebo group (11.2 months vs 4.3 months; hazard ratio: 0.18; p < 0.0001). Similar findings were noted for patients with wild-type BRCA, although the difference between groups was smaller (7.4 months vs 5.5 months; hazard ratio: 0.54; p = 0.007). Patient-reported outcomes, including Functional Assessment of Cancer Therapy – Ovarian Symptom Index, did not show a significant difference between the placebo and treatment groups, suggesting that maintenance treatment did not decrease functioning or quality of life in these patients. Patient-reported outcome data beyond progression was not captured, and therefore quality of life effects related to subsequent chemotherapy treatments (likely to occur sooner in the placebo group) could not be used to assess the benefit of extending PFS on patient-reported outcomes for patients treated with a PARP inhibitor vs placebo.

#### 1.1.2. Study Objectives

In this document, "ovarian cancer" refers to high-grade serous epithelial cancers of the ovary, fallopian tube, or primary peritoneal cancer. As detailed in Section 3.8, "sensitivity to platinum-based therapy" is defined by platinum-free interval (PFI) following the first platinum-based therapy (required for eligibility) or the last platinum-based therapy (defines patient population for primary and key secondary objectives). Homologous recombination deficiency (HRD) status is based upon the Myriad MyChoice HRD test and/or a centralized gBRCA test.

The primary objective of the study is to evaluate the Objective Response Rate (ORR) of niraparib in HRD-positive patients with advanced, relapsed, high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer, who have received 3 or 4 prior lines of


anti-cancer therapy and are platinum-sensitive to the last platinum-based therapy (excluding patients with prior PARP treatment).

The key secondary objectives of the study are as follows:

- To evaluate the ORR of niraparib in all patients with advanced, relapsed, high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer, who have received 3 or 4 prior lines of anti-cancer therapy and are platinum-sensitive to the last platinum-based therapy (excluding patients with prior PARP treatment).
- To evaluate the ORR of niraparib in all patients with advanced, relapsed, high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer, who have received 3 or 4 prior lines of anti-cancer therapy and are platinum-sensitive or platinum-resistant to the last platinum-based therapy (excluding patients with prior PARP treatment).
- To evaluate the ORR of niraparib in all patients with advanced, relapsed, high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer.

Other secondary objectives of the study are as follows:

- To evaluate the efficacy (duration of response [DOR], disease control rate [DCR], PFS, time to first subsequent therapy [TFST] and overall survival [OS]) of niraparib in patients who have received 3 or 4 prior lines of anti-cancer therapy.
- To evaluate the efficacy (DOR, DCR, PFS, TFST and OS) of niraparib in all patients regardless of prior lines of anti-cancer therapy.
- To evaluate the safety and tolerability of niraparib.

The exploratory objectives of the study are as follows:

- To evaluate the efficacy and safety of niraparib in all patients who are platinum-refractory to the last platinum-based therapy.
- To evaluate the efficacy and safety of niraparib in all patients with prior PARP treatment.
- To evaluate QT interval corrected for heart rate (QTc) in a subset of niraparib-treated ovarian cancer patients.
- To assess population pharmacokinetics (PK) and estimate PK parameters for niraparib and its major metabolite.
- To explore potential biomarkers related to ovarian cancer and poly(ADP-ribose) polymerase (PARP) inhibition (eg, DNA repair pathways).

This statistical analysis plan (SAP) is designed to outline the methods to be used in the analyses of study data in order to answer the study objectives. Patient populations to be used for analyses, data handling rules, statistical methods, and formats for data presentation are identified and provided. The statistical analyses and summary tabulations described in this SAP will provide the basis for the results sections of the clinical study report (CSR) for this trial.

This SAP will also outline any differences in the currently planned analytical objectives relative to those planned in the study protocol.

The SAP is based upon the following study documents:


- Study Protocol v8.0 dated 21 December 2017
- Electronic Case Report Form (eCRF) v.1.184 dated 23 October 2017
- Analyses of PK data are described in a separate SAP, but all data will be displayed in the listings associated with this SAP.

## 1.2. Study Design

### 1.2.1. Synopsis of Study Design

This study is a multicenter, open-label, single-arm, Phase 2 study evaluating the safety and efficacy of niraparib in patients with recurrent ovarian cancer who experienced a response lasting at least 6 months to first-line platinum-based therapy and who previously treated with 3 or 4 lines of anti-cancer therapy (including, but not limited to, gemcitabine, doxorubicin, topotecan, carboplatin, oxaliplatin, cisplatin, bevacizumab, or PARP inhibitors as single agents or in combination per standard of care). Study objectives are discussed in Section 1.1.2.

In order to determine eligibility, a tumor sample will be sent to a centralized laboratory for immediate HRD testing. Archival or fresh tissue is required in order to enroll in the study. The sample may be sent in advance of the protocol-defined screening period in order to facilitate the screening and enrollment process. Patients must wait for the results from the on-study centralized HRD testing prior to enrollment, unless they have previously detected gBRCA mutation. Blood samples also will be collected for all patients during screening for determination of gBRCAmut status. If HRD status is known, then it is not necessary to wait for HRD testing results for enrollment into the study, however confirmatory HRD testing still needs to be performed.

In order to evaluate tumor markers, an optional fresh biopsy may be done at screening and at the end of treatment (EOT) visit.

Niraparib 300 mg will be administered orally QD continuously beginning on Day 1 and every cycle (28 days) thereafter until the patient discontinues study treatment. Three capsules of 100 mg strength will be taken at each dose administration. Dose interruption (no longer than 28 days) and dose reductions to 2 capsules daily (200 mg), and subsequently to 1 capsule daily (100 mg), will be allowed (no further dose reductions will be allowed). Dose interruption and/or reduction may be implemented at any time for any grade toxicity considered intolerable by the patient. The timing of efficacy or safety evaluations should not be affected by dose interruptions or reductions. Patients will continue on study medication until disease progression as long as in the Investigator's opinion they are benefiting from treatment and do not meet any other discontinuation criteria.

Blood samples for measurements of plasma levels of niraparib and its major metabolite will be obtained on Cycle 1/Day 1 predose and 2 hours postdose, Cycle 2/Day 1 predose and 2 hours postdose, Cycle 4/ Day 1 predose, and Cycle 8/ Day 1 predose. At selected sites, a subset of approximately 12 patients will undergo intensive, triplicate ECG monitoring to coincide with PK evaluation on Cycle1/Day 1. Triplicate ECGs should be performed between 2 and 5 minutes apart and should be performed prior to blood draws for PK. These patients will have triplicate ECGs and PK samples taken predose and at 1, 2, 4, 6, and 8 hours postdose. Patients will be supine and rested for approximately 2 minutes before ECGs are recorded. The average of the triplicate measures will be used for analysis. This subset of patients will undergo all other


assessments in the study. As of 09 February 2016, the PK QTc sub-study had reached the enrollment target of 12 patients and is now closed to enrollment.

Blood samples will be collected for all patients at screening for the exploratory evaluation of circulating biomarkers.

Clinic visits will be weekly during Cycle 1 and then every 4 weeks (±3 days) for subsequent cycles. Response Evaluation Criteria in Solid Tumors (RECIST; v.1.1) tumor assessment via CT or MRI of the abdomen/pelvis and clinically indicated areas is required every 8 weeks ( $\pm 7$  days) from Cycle 1/Day 1 for 6 months and then every 12 weeks until progression. Copies of scans will be collected for future central evaluation if needed. Cycle timing will not be delayed for treatment interruptions, and tumor assessment should occur according to this schedule regardless of whether study treatment is interrupted. All AEs and serious adverse events (SAEs) will be collected and recorded for each patient from the day of signing the screening informed consent form (ICF) until the EOT visit. New SAEs (including deaths) will be collected for 30 days after the last dose of study treatment. All AEs and SAEs experienced by a patient, irrespective of the suspected causality, will be monitored until the AE or SAE has resolved, any abnormal laboratory values have returned to baseline or normalized, until there is a satisfactory explanation for the changes observed, until the patient is lost to follow-up, or until the patient has died. The Adverse Events of Special Interest (AESIs) for this study are myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), and secondary cancers (new malignancies other than MDS/AML, pneumonitis, and embryo-fetal toxicity. AESIs must be reported to the Sponsor as soon as the Investigator becomes aware of them (per Section 6.2.5.3 of the protocol).

Approximately 500 patients will be enrolled in the study at approximately 60 sites. The study will be conducted in conformance with Good Clinical Practice (GCP).

#### 1.2.2. Randomization Methodology

Not applicable as this is a single-arm study.

### 1.2.3. Stopping Rules and Unblinding

There are no pre-specified stopping rules for the study. Unblinding is not applicable as this is a single-arm, open-label study.

#### 1.2.4. Study Procedures

The schedule of assessments, as outlined in the study protocol, is provided in Table 1-1.


**Table 1-1** Schedule of Assessments

| Cycle <sup>a</sup> | Screening <sup>b</sup> | ening <sup>b</sup> 1 | | | | Subsequent<br>Cycles <sup>a</sup> | EOT (within 7 days of last | Post-<br>Treatment |
|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 22 | Cycle n, Day 1 | dose) | Assessments |
| Informed consent <sup>b, c</sup> | X | | | | | | | |
| Demographics | X | | | | | | | |
| Medical, surgical, cancer, and medication history | X | | | | | | | |
| Sample collection (tumor) for centralized <i>tBRCA</i> <sup>mut</sup> /HRD testing <sup>c</sup> | X <sup>c</sup> | | | | | | | |
| Sample collection (whole blood) for <i>gBRCA</i> <sup>mut</sup> testing | X | | | | | | | |
| Tumor sample (optional) d | X | | | | | | X | |
| Blood sample for exploratory biomarker analysis <sup>e</sup> | X | | | | | | | |
| Blood sample for PK <sup>f</sup> | | X | | | | X | | |
| Tumor assessment (RECIST) <sup>g</sup> | X | | | | | Xg | X | Xg |
| Chest CT/MRI <sup>h</sup> | X | | | | | | | |
| Pregnancy test <sup>i</sup> | X | | | | | X | | |
| Serum chemistry | X | $\mathbf{X}^{\mathrm{j}}$ | | X | | X | X | |
| $CBC^k$ | X | $\mathbf{X}^{\mathrm{j}}$ | X <sup>l</sup> | X | X <sup>l</sup> | X | X | |
| Serum CA-125 <sup>j</sup> | X | Xg | | | | X <sup>g</sup> | X | X |
| ECG <sup>m</sup> | X <sup>m</sup> | | | | | | | |
| Physical examination | X | | | | | | | |
| Symptom-directed physical examination | | X | | X | | X <sup>n</sup> | X | |
| Vital signs, height, weight <sup>o</sup> | X | X | | X | | X | X | |


| Cycle <sup>a</sup> | Screening <sup>b</sup> | 1 | 1 | | | Subsequent<br>Cycles <sup>a</sup> | EOT (within 7 days of last | Post-<br>Treatment |
|---|---|---|---|---|---|---|---|---|
| Day | -28 to -1 | 1 | 8 | 15 | 22 | Cycle n, Day 1 | dose) Assessments | |
| ECOG performance status | X | | | | | X <sup>n</sup> | X | |
| Bone marrow aspirate and biopsy <sup>p</sup> | | Xp | | | | | | |
| Concomitant medication | X | X | | X | | X | X | |
| Adverse event monitoring | X | X | | X | | X | Xq | X |
| Study treatment dispensed/collected | | X | | | | X | X | |
| Survival assessment <sup>r</sup> | | | | | | | | X |

Abbreviations: AE = adverse event; AML = acute myloid leukemia; BP = blood pressure; CA-125 = cancer antigen 125; CBC = complete blood count; CT = computed tomography; ECG = electrocardiogram; ECOG = Eastern Cooperative Oncology Group; EOT = end of treatment;  $gBRCA^{mut}$  = germline breast cancer gene mutation; HRD = homologous recombination deficiency; ICF = informed consnt form; MDS = myelodysplastic syndrome; MRI = magnetic resonance imaging; PK = pharmacokinetics; RECIST = Response Evaluation Criteria in Solid Tumors; SAE = serious adverse event;  $tBRCA^{mut}$  = tumor breast cancer gene mutation.

- <sup>a</sup> Treatment cycles are 28 days long, with visits on Day 1 of each cycle unless otherwise specified. Visits (other than Cycle 1) continue every 28 days until study treatment discontinuation. All visits have a window of ±3 days (calculated in reference to Cycle 1/Day 1).
- b Screening tests that could be considered standard of care (ie, CT/MRI, physical examination, vital signs, height, weight, and assessment of serum chemistry, CBC, pregnancy testing, and serum CA-125) that were performed within the protocol-required timelines (ie, within the 28-day screening window; within 72 hours prior to first dose [ie, Cycle 1/Day 1] where required) but prior to informed consent being obtained may be used as part of the patient's screening assessment.
- <sup>c</sup> For patients who do not have archival tissue, tissue from a fresh biopsy must be obtained prior to study treatment initiation. Centralized HRD testing of tumor sample must be completed with results reported prior to enrollment. The sample may be sent in advance of the protocol-defined screening period in order to facilitate the screening and enrollment process. A separate ICF may be signed prior to the screening period for HRD testing in order to facilitate early testing. Depending on local site requirements, patients may sign a screening study ICF prior to the screening period to facilitate early HRD testing only. All other study tests and procedures must be done in the screening window (Day -28 to Day -1). For patients who do not have archival tissue, tissue from a fresh biopsy must be obtained.
- d Formalin-fixed, paraffin-embedded tumor sample consisting of a total of 100-micron thickness of sections (≥80-micron minimum) or unsectioned paraffin block.
- e Blood samples will be collected for all patients during screening for the exploratory evaluation of circulating markers of efficacy. The sponsor may discontinue the blood collection when samples have been collected from an adequate number of patients.
- f Blood samples for PK may be collected on Cycle 1/Day 1 predose (within 30 minutes) and 2 hours (± 15 minutes) postdose, on Cycle 2/ Day 1 predose (within 30 minutes) and 2 hours (± 15 minutes) postdose, on Cycle 4/Day 1 predose (within 30 minutes), and on Cycle 8/Day 1 predose (within 30 minutes). At selected sites, a subset of patients (approximately 12) will undergo triplicate ECG monitoring to coincide with PK evaluation on Cycle 1/Day 1 predose and at 1, 2, 4, 6, and 8 hours postdose. Note: The exact time of the PK blood draw will be recorded, and ECG monitoring is to be completed prior to the PK blood draw or other laboratory evaluations.


- EXECIST tumor assessment via CT or MRI of abdomen/pelvis and clinically indicated areas required at screening, every 8 weeks (±7 days) from Cycle 1/Day 1 (ie, Cycle 3, Cycle 5, Cycle 7) for 6 months, and then every 12 weeks (ie, Cycle 10, Cycle 13, Cycle 16, etc) until progression. Positron emission tomography/CT may be used according to RECIST guidelines. Cycle timing will not be delayed for treatment interruptions, and tumor assessment should occur according to this schedule regardless of whether study treatment is interrupted. If a patient discontinues treatment for a reason other than disease progression as defined in the protocol or death, withdrawal of consent, or loss to follow-up, then scans and CA-125 testing should continue at the specified intervals (until the start of subsequent anticancer treatment). If a patient had a CT/MRI of the abdomen/pelvis and clinically indicated areas within the 28-day screening window before Cycle 1/Day 1 but prior to signing the main ICF, the patient is not required to complete an additional CT/MRI scan for study screening. CT/MRI scans completed during screening prior to signing the main ICF must have been performed and be able to be submitted per the image acquisition guidelines.
- h Chest CT/MRI if not done as part of RECIST tumor assessment at screening. If the chest CT/MRI is clear at screening, repeat chest imaging is not required in the absence of lesions to be followed or in the absence of clinical indication requiring follow-up.
- Negative serum pregnancy test required within 72 hours from first dose of study treatment (ie, Cycle 1/Day 1) for females of childbearing potential; repeated every 3 months for duration of study (ie, Cycle 4, Cycle 7, etc).
- <sup>j</sup> If screening laboratory testing (serum chemistry, CBC, CA-125) performed within 72 hours of Day 1, repeat testing is not required.
- k If dose interruption or modification is required at any point on study because of hematologic toxicity, weekly blood draws for CBC will be monitored until the AE resolves, and to ensure safety of the new dose, weekly blood draws for CBC will be also required for an additional 4 weeks after the AE has been resolved to the specified levels, after which monitoring every 4 weeks may resume.
- Collection of blood for the Cycle 1/Day 8 and Day 22 CBC may be done at the study center's local laboratory or at a laboratory local to the patient, if approved by the Principal Investigator as an adequate laboratory. The laboratory must have the capability to provide results to the Principal Investigator electronically or by fax within 24 hours of blood collection.
- m Patients will undergo a single ECG monitoring assessment at screening, prior to laboratory evaluations. At selected sites, a subset of patients (approximately 12) will undergo triplicate ECG monitoring to coincide with PK evaluation on Cycle 1/Day 1 predose and at 1, 2, 4, 6, and 8 hours postdose. Triplicate ECGs should be performed between 2 and 5 minutes apart and should be performed prior to blood draws for PK or other laboratory evaluations.
- <sup>n</sup> Symptom-directed physical examination is to be conducted at every visit and ECOG assessed every 12 weeks (±7 days) until EOT.
- <sup>o</sup> Vital signs include BP, pulse, and temperature. Height obtained at screening only.
- P For any suspected MDS/AML case reported while a patient is receiving treatment or being followed for post-treatment assessments, bone marrow aspirate and biopsy testing must be completed by a local hematologist. A whole blood sample will also be collected for cytogenetic analysis (mutations of select myeloid-associated genes). Testing completed as part of standard of care is sufficient as long as the methods are acceptable to the Sponsor's Medical Monitor. The study site must receive a copy of the hematologist's report of aspirate/biopsy findings (which must include a classification according to World Health Organization criteria) and other sample testing results related to MDS/AML.
- <sup>q</sup> New SAEs recorded up to 30 days after last dose of study treatment administration.
- Every 90 (±7) days after treatment discontinuation. In addition to survival, this assessment also includes outcomes for subsequent anticancer therapies including any new malignancy information.


### 1.2.5. Efficacy, Pharmacokinetic, and Safety Parameters

### 1.2.5.1. Efficacy Parameters

Protocol-specified efficacy parameters include:

- ORR, which is defined as the proportion of patients achieving confirmed complete response (CR) or partial response (PR) as assessed by the Investigator per RECIST (v1.1).
- DOR, which is defined as the time from first documentation of CR or PR until the earlier date of first documentation of progressive disease (PD) or death by any cause in the absence of progression as assessed by the Investigator per RECIST (v1.1).
- DCR, which is defined as the proportion of patients achieving best overall response of CR, PR, or stable disease (SD) as assessed by the Investigator per RECIST (v1.1).
- PFS, which is defined as the time from the date of first dose of study treatment to the earlier date of assessment of progression or death by any cause in the absence of progression as assessed by the Investigator per RECIST (v1.1).
- OS, which is defined as the time from the date of first dose to the date of death for any cause.
- TFST, which is defined as the time from the date of first dose of study treatment to the date of first dose of first subsequent therapy or death, whichever occurs first.

#### 1.2.5.2. Pharmacokinetic Parameters

A separate analysis plan will describe PK parameters and analyses; considering that the PK analyses of the trial takes place during COVID-19 pandemic, as a result of which some of the trial procedures could be impacted in terms of missing visits and/or assessments. Missing protoctol required data/visits due to COVID-19 must be noted in participant notes and recorded as a COVID-19-related protocol deviations. A summary of the following COVID-19 assessments will be produced: case diagnosis, COVID-19 test performed, and results of the COVID-19 test. In addition, a separate listing defining "Important" GSK protocol deviations related to COVID-19 will be presented.

### 1.2.5.3. Safety Parameters

Safety parameters evaluated during the conduct of the study include: treatment-emergent AEs (TEAEs), clinical laboratory (hematology, chemistry, coagulation, and urinalysis), vital signs, ECG, physical examination, Eastern Cooperative Oncology Group (ECOG) performance status, and use of concomitant medications. The safety endpoints are:

- TEAEs
- Clinical laboratory:
  - Complete blood count (CBC): hemoglobin, platelets, mean platelet volume (optional), mean corpuscular volume, white blood cell count, differential white cell count (absolute lymphocyte count, percent lymphocytes, absolute neutrophil count, and percent neutrophils)


- Serum chemistry assessments for safety include: sodium, potassium, calcium, magnesium, chloride, glucose, creatinine, total bilirubin, gamma glutamyltransferase (GGT), alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), urea or blood urea nitrogen, total protein, albumin, lactate dehydrogenase, amylase
- o Serum CA-125
- Serum pregnancy testing
- Physical examination, which includes assessments of the following body systems:
  - General Appearance
  - Dermatologic
  - o Head, Eyes, Ears, Nose, and Throat (HEENT)
  - o Thyroid
  - Lymph Nodes
  - Respiratory
  - Cardiovascular
  - Gastrointestinal
  - Extremities
  - Musculoskeletal
  - o Psychiatric
- Vital signs:
  - Height (at screening only)
  - Weight
  - Blood pressure
  - o Pulse
  - Temperature
- ECOG performance status
- ECG (all patients at screening, PK QTc sub-study patients at all time points)
- Concomitant medications

Additional safety parameters include study treatment exposure and compliance.


#### 2. PATIENT POPULATION

# 2.1. Population Definitions

The following patient populations will be evaluated and used for presentation and analysis of the data:

- Safety (SAF) population is defined as all patients who receive at least 1 dose of study drug.
- Intent-to-Treat (ITT) population is defined as all dosed patients with measurable disease at baseline. Measurable disease at baseline is determined by the existence of at least 1 target lesion at baseline tumor scan.
- Response-Evaluable (RE) population is defined as all ITT patients with at least 1 evaluable post-baseline tumor scan.

Given the single arm study design, the SAF population will be used to summarize the patient disposition and baseline characteristics in this study. The ITT population is the primary population for the analysis of efficacy endpoints. The SAF population is the primary population for the analysis of safety endpoints. The RE population will be used in supportive analyses when applicable.

### 2.2. Protocol Deviations

Protocol Deviations (PD) will be assessed as important or significant per Sponsor's SOP.

- A PD is classified as important if there is the potential to impact the completeness, accuracy, and/or reliability of the study data, or affect a patient's rights, safety, or wellbeing.
- An important PD is classified as significant if it is confrrmed to adversely impact the completeness, accuracy, and/or reliability of the study data, or affect a patient's rights, safety, or well-being.

All PDs will be identified and finalized prior to database lock.

The following protocol deviation summaries will be provided:

- Number and percentage of patients with a significant protocol deviation by type of deviation.
- Number and percentage of patients with an important protocol deviation by type of deviation.
- A listing of all protocol deviations.

Per-protocol analysis that excludes patients with significant protocol deviations will not be performed.


### 3. GENERAL STATISTICAL METHODS

## 3.1. Sample Size Justification

The study protocol initially allowed enrollment of all patients with at least 3 prior lines of anticancer therapy. In the subsequent protocol amendments, the study enrollment was adjusted to allow only HRD-positive patients with 3 or 4 prior lines of anti-cancer therapy. This adjustment was made in consideration of the evolving role of PARP inhibitors in ovarian cancer treatment based on external data. Overall, approximately 500 patients are expected in the study. The study enrollment is also expected to include a minimum number of tBRCAmut patients ( $\geq$ 50) and HRD-positive patients ( $\geq$ 150).

For the primary efficacy endpoint of ORR in HRD-positive patients who have received 3 or 4 prior lines of anti-cancer therapy and are platinum-sensitive to the last platinum-based therapy, an alternative hypothesis of ORR  $\geq$ 30% is considered against a null hypothesis of ORR  $\leq$ 10%.

For the key secondary efficacy endpoints of ORR tested in broader subgroups to include platinum-resistant patients and/or HRD-negative/unknown patients, an alternative hypothesis of ORR  $\geq$ 25% is considered against a null hypothesis of ORR  $\leq$ 10%.

It is estimated that 45 patients would provide 90% power for testing the primary efficacy analyses. Statistical power for various sample sizes are presented below to provide guidance for the key secondary hypotheses when tested individually (regardless of sequential testing) using 1-sided alpha 0.025. The power is calculated by assuming the exact binomial distribution using East® software Version 6.4.

| n | Statistical Power* |
|----|--------------------|
| 45 | 72% |
| 60 | 85% |
| 75 | 92% |
| 90 | 96% |

<sup>\*</sup> Ho: ORR <10% vs Ha: ORR >25%

As of August 2017, approximately 450 patients were dosed in the study. Approximately 320 patients had 3 or 4 prior lines of anti-cancer therapy (~150 HRD positive). Based on a preliminary calculation of the platinum-sensitivity to the last platinum-based therapy, the number of enrolled patients for the primary endpoint and the key secondary efficacy endpoints are considered adequate to ensure sufficient power for the planned analysis.

### 3.2. General Methods

All safety data listings that contain an evaluation date will also contain a relative study day. Pre-treatment and on-treatment study days are numbered relative to the day of the first dose of study drug which is designated as Day 1. The preceding day is Day -1, the day before that is Day -2, etc. The last day of study drug is designated with an "L" (eg, Day 14L). Post-treatment study days are numbered relative to the last dose and are designated as Day +1, Day +2, etc. In addition to relative day, cycle and day of treatment within cycle will be calculated and presented.


All output will be incorporated into Microsoft Word or Excel files or Adobe Acrobat PDF files, sorted and labeled according to the International Conference on Harmonisation (ICH) recommendations[8], and formatted to the appropriate page size(s).

Tabulations will be produced for appropriate demographic, baseline, efficacy, and safety parameters. Unless otherwise stated, all tabulations will be summarized for patients with 3 or 4 previous chemotherapy regimens,  $\geq 5$  previous chemotherapy regimens, and overall (all lines of prevous chemotherapy regimens including  $\leq 2$  lines).

For categorical variables, summary tabulations of the number and percentage of patients within each category of the parameter will be presented. Percentages will be based on the patients with a non-missing parameter. Percentages will be reported to 1 decimal place. Percentages will not be presented for zero counts.

For continuous variables, the number of patients, mean, standard deviation (SD), median, first quartile  $(Q_1)$ , third quartile  $(Q_3)$ , minimum, and maximum values will be presented. Mean, median,  $Q_1$ , and  $Q_3$  will be reported to 1 more decimal place than the raw data, while the SD will be reported to 2 more decimal places than the raw data.

Time-to-event data will be summarized using Kaplan-Meier (KM) methodology using 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles with associated 2-sided 95% confidence intervals (CIs), as well as percentage of censored observations.

Formal statistical hypothesis testing will be performed on the primary efficacy endpoint as described in the sections below.

#### In addition:

- P-values greater than or equal to 0.001, in general, will be presented to 3 decimal places; p-values less than 0.001 will be presented as "<0.001"
- CIs will be presented to 1 more decimal place than the raw data
- Weeks will be calculated as Number of days divided by 7
- Months will be calculated as Number of days divided by 30.4375
- Years will be calculated as Number of days divided by 365.25
- Day 1 will be considered as the first day of treatment
- End of Study is defined as the last available study assessment
- All tables, figures, and listings will include footers at the bottom of the page reflecting the path and date of the datasets, datasets used to generate the tables, figures, and listings, and date and time of the generation of the output

**Note regarding COVID-19:** COVID-19 pandemic may impact the conduct of clinical studies. Challenges may arise from quarantines, site closures, travel limitations interruptions to the supply chain for the investigational product or other considerations if site personnel or patients become infected with COVID-19. These challenges may lead to difficulties in meeting protocol specified procedures, including administering or using the investigational product or adhering to protocol-mandated visits and laboratory/diagnostic testing.


# 3.3. Computing Environment

All statistical analyses will be performed using SAS statistical software v9.4 or later, unless otherwise noted. Medical history and AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) v20.0 or later. Laboratory parameter changes will be described using shift tables, relative to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03. Concomitant medications will be coded using the latest version of the World Health Organization's (WHO) Anatomical Therapeutic Chemical (ATC) classification.

### 3.4. Baseline Definitions

For all analyses except ECG, baseline is defined as the most recent measurement prior to the first administration of study drug. For ECG analyses, baseline will be defined as the average of the closest triplicate (if triplicates were collected) readings prior to dosing on the first day that study drug is administered.

# 3.5. Methods of Pooling Data

Data will be pooled across study sites.

## 3.6. Adjustments for Covariates

No formal statistical analyses that adjust for possible covariate effects are planned for the efficacy or safety endpoints. Formal analyses adjusting for possible covariate effects for the PK endpoints are contained in a separate SAP.

# 3.7. Multiple Comparisons/Multiplicity

Multiplicity is controlled by conducting a hierarchical testing of the primary endpoint and the key secondary endpoints.

# 3.8. Subpopulations

### 3.8.1. Prior Lines of Chemotherapy

The reported cancer therapy regmens from eCRF page (Ovarian Cancer Treatment) will be checked with the per-protocol list of chemotherapy regimens to determine patients with 3 or 4 previous chemotherapy regimens consistent with the protocol inclusion criteria #5:

• Patients must have completed 3 or 4 previous chemotherapy regimens (eg, gemcitabine, doxorubicin, topotecan, carboplatin, oxaliplatin, cisplatin, bevacizumab, or PARP inhibitors as single agents or in combination per standard of care).

A list of the per-protocol chemotherapy regimens is provided in the Appendix (Section 7.5).

Patients will be classified by  $\leq 2$ , 3-4, and  $\geq 5$  previous chemotherapy regimens based on the perprotocol chemotherapy regimens, and summarized by:

- Number and percentage by the number of prior chemotherapy regimens
- Duration (in months) between the end date of the last chemotherapy regimen and the date of first dose of study treatment


### 3.8.2. Response to the Last Platinum-Based Therapy

Platinum-free interval (PFI) to the last platinum-based therapy will be determined between the reported stop date of the last platinum-based therapy and the reported date of disease progression following the last platinum-based therapy.

- Platinum-sensitive: PFI ≥6 months (180 days) after the end date of last platinum-based therapy
- Platinum-resistant: PFI >4 weeks (28 days) and <6 months (180 days) after the end date of last platinum-based therapy
- Platinum-refractory: PFI ≤4 weeks (28 days) after the end date of last platinum-based therapy
- Response-unknown: PFI is missing. PFI is missing if both dates are completely missing. Partial dates will be handled according to Section 3.10

The per-protocol platinum-based therapies are determined using the list in the Appendix (Section 7.5).

Patients will be summarized by:

- Number and percentage by the number of prior platinum-based therapies
- Duration (in months) between the end date of the last platinum-based therapy and the date of first dose of study treatment

#### 3.8.3. Prior PARP Treatment

Patients with any PARP treatment prior to the first dose of study treatment will be identified and analyzed for exploratory purpose.

The list of prior PARP treatment includes: nirapariab, olaparib, rucaparib, and veliparib.

#### 3.8.4. Biomarker Subpopulations

### 3.8.4.1. Biomarker Definitions

BRCA mutation (BRCA-mut): A deleterious or suspected deleterious BRCA1 or BRCA2 mutation found in a tumor and/or in blood. In this document, BRCA-mut refers to patients with either germline or somatic mutation.

- Germline BRCA mutation (gBRCA-mut): A germline BRCA mutation is an inherited deleterious or suspected deleterious mutation in either a BRCA1 or BRCA2 tumor suppressor gene found in blood.
- Somatic BRCA mutation (sBRCA-mut): A somatic BRCA mutation is a deleterious or suspected deleterious alteration in the BRCA1 or BRCA2 genes that is acquired after conception (not hereditary). sBRCA-mut can be determined by the presence of tumor BRCA mutation (tBRCA-mut) but the absence of gBRCA-mut in blood.

BRCA wild type (BRCA-wt): A tumor and/or blood does not possess either a deleterious or suspected deleterious germline or a somatic BRCA mutation. In this document, BRCA-wt refers to patients without gBRCA-mut and sBRCA-mut.


Homologous recombination deficiency (HRD) – Dysregulation in the homologous recombination pathway (due to genetic mutations or alterations) leading to cellular genomic instability and an inability to efficiently repair damaged DNA.

HRD positive (HRD-pos): HRD positive status may be determined by the myChoice HRD test. Any tumor that scores ≥42 or has a deleterious or suspected deleterious BRCA mutation would be considered HRD positive.

HRD negative (HRD-neg): HRD negative status may be determined by the myChoice HRD test. Any tumor that scores <42 and does not possess a deleterious or suspected deleterious BRCA mutation would be considered HRD negative.

### 3.8.4.2. Study-Specific Biomarker Populations

In this study, tumor BRCA and HRD status are determined by tumor samples at screening via the myChoice HRD test. The gBRCA status is determined by a central test of blood samples at screening and recorded in the eCRF BRCA form.

All patients will be classified by BRCA mutation status as follows:

- BRCA-mut:
  - gBRCA-mut: patients with any variant or large rearrangement found in BRCA1/2 that is either positive for a deleterious mutation or genetic variant for suspected deleterious
  - o sBRCA-mut: patients with tBRCA-mut but without gBRCA-mut
- BRCA-wt: patients without gBRCA-mut and sBRCA-mut
- BRCA unknown (BRCA-unk): None of tBRCA and gBRCA test results available (eg, test canceled, incomplete/inconclusive, or data missing for a patient).

All patients will be summarized by HRD status in the following subgroups:

- HRD-pos:
  - o BRCA-mut
  - o (BRCA-wt or BRCA-unk) and HRD test score ≥42
- HRD-neg: (BRCA-wt or BRCA-unk) and HRD test score <42
- HRD unknown (HRD-unk): HRD test result not available (eg, test canceled, incomplete/inconclusive, or data missing for a patient)

In addition, the tBRCA-mut patients will also be summarized based on the reported BRCA variants found in tumor:

- BRCA1 variant
- BRCA2 variant

The gBRCAmut patients will also be summarized based on the reported BRCA variants found in blood and recorded in the eCRF BRCA form:

- BRCA1 variant
- BRCA2 variant


• Large rearrangement in BRCA1/2

If applicable, other exploratory biomarker subpopulations may be further defined and analyzed.

# 3.9. Withdrawals, Dropouts, Loss to Follow-up

Patients who are withdrawn or discontinue from the study will not be replaced.

# 3.10. Missing Data

In general, there will be no substitutions made to accommodate missing data points. All data recorded on the eCRF will be included in data listings that will accompany the CSR.

When calculating PFI to the last platinum-based therapy, partial dates of the last platinum-based therapy and the disease progression following the last platinum-based therapy will be handled as follows. If the day of the month is missing, the day will be set to the first day of the month. If the day and month are both missing, the day and month will be assumed to be January 1. If the imputed date of the disease profession following the last platinum-based therapy is earlier than the end date of the last platinum-based therapy, the imputed date of the disease progression will be set equal to the end date of the last platinum-based therapy. Imputation of partial dates is used only to estimate PFI; data listings will present the partial date as recorded in the eCRF.

When tabulating AE data, partial dates will be handled as follows. If the day of the month is missing, the onset day will be set to the first day of the month unless it is the same month and year as study treatment. In this case, in order to conservatively report the event as treatment-emergent, the onset date will be assumed to be the date of treatment. If the onset day and month are both missing, the day and month will be assumed to be January 1, unless the event occurred in the same year as the study treatment. In this case, the event onset will be coded to the day of treatment in order to conservatively report the event as treatment-emergent. A missing onset date will be coded as the day of treatment. If the resulting onset date is after a reported date of resolution, the onset date will be set equal to the date of resolution. Imputation of partial dates is used only to determine whether an event is treatment-emergent; data listings will present the partial date as recorded in the eCRF.


### 3.11. Visit Windows

**Table 3-1** Evaluation Intervals

| Evaluation | Protocol-Specified Interval | Interval for Analysis |
|---|---|---|
| Screening | Day -28 to Day -1 | Day -28 to Day -1 |
| Cycle 1, Day 1 | Day 1 | Day 1 |
| Cycle 1, Day 8 | Day 5 to Day 11 | Day 5 to Day 11 |
| Cycle 1, Day 15 | Day 12 to Day 18 | Day 12 to Day 18 |
| Cycle 1, Day 22 | Day 19 to Day 25 | Day 19 to Day 25 |
| Cycle n, Day 1 | Day $28(n-1) - 3$ to Day $28(n-1) + 3*$ | Day $28(n-1) - 3$ to Day $28(n-1) + 3*$ |
| End of Treatment | Within 7 days of last dose, except for AEs which will be collected for up to 30 days after the date of the last dose | Within 7 days of last dose, except for AEs which will be collected for up to 30 days after the date of the last dose |

Abbreviations: AE = adverse event; ECOG = Eastern Cooperative Oncology Group; RECIST = Response Evaluation Criteria in Solid Tumors.

Note: Day 25 is contained within both the Cycle 1 Day 22 and the Cycle 2 Day 1 visit windows. Visits occurring on Day 25 will be classified based on the purpose of the visit.

It is expected that all visits should occur according to the protocol schedule. By-visit summaries and analyses will be by nominal visit (all data will be tabulated per the evaluation visit as recorded on the eCRF even if the assessment is outside of the visit window for analysis). In data listings, the relative day of all dates will be presented.

# 3.12. Administrative Interim Analyses

Safety data from this study collected through 20 May 2016 was analyzed to write an interim CSR and for inclusion as part of the integrated summaries of safety in the niraparib submission in the second half of 2016. Efficacy data from this study were not analyzed.


<sup>\*</sup> Symptom-directed physical examination and ECOG performance status are required every 12 weeks (±7 days), serum pregnancy tests are required at 3-month intervals from screening (Cycles 4, 7, etc), and RECIST (v1.1) tumor assessments (as clinically indicated) are required every 8 weeks (±7 days) for 6 months and then every 12 weeks (±7 days) until progression. Therefore, the symptom-directed physical examinations and ECOG performance status are required at Cycle 4, Cycle 7, etc, with a protocol-specified interval and an interval for analysis of Day 28(*n*-1) – 7 to Day 28(*n*-1) + 7 (where *n* is the cycle number). RECIST tumor assessments are required at Cycles 3, 5, 7, 10, 13, etc, with a protocol-specified interval and an interval for analysis of Day 28(*n*-1) – 7 to Day 28(*n*-1) + 7 (where *n* is the cycle number).

### 4. STUDY ANALYSES

## 4.1. Patient Disposition

Patient disposition will be tabulated and include the numbers of screened patients (who have signed informed consent) and the numbers of patients in each patient population for analysis, the numbers who discontinued treatment and discontinued study and reason(s) for withdrawal, and the number of patients who died.

Tables will be summarized by 3-4 prior lines, ≥5 prior lines, and Overall. A by-patient data listing of study completion information including the reasons for treatment discontinuation and/or study discontinuation will be presented.

# 4.2. Demographics, Baseline Characteristics, and Medical History

Demographics, baseline characteristics, and medical history information will be summarized using descriptive statistics. Tables will be summarized by 3-4 prior lines, ≥5 prior lines, and Overall. No formal statistical comparisons will be performed.

Demographic and baseline data for each patient will be provided in data listings.

The demographic and baseline characteristics tables will include the following variables:

- Region (US, Canada)
- Age at time of screening (years) calculated as date of screening minus date of birth / 365.25, unless local regulations prevent the collection of date of birth, in which case age, as reported on the eCRF, will be used
- Age categories (18 to <65, 65 to <75,  $\ge 75$ ; and  $\ge 65$ )
- Reproductive status (childbearing/non-childbearing potential)
- Race (White, Black, Asian, American Indian/Alaska native, native Hawaiian or other Pacific Islander, other, unknown, and not reported)
- Ethnicity (Hispanic, non-Hispanic, unknown, and not reported)
- Time from first diagnosis to first dose (years)
- Primary tumor site (ovarian, primary peritoneal, or fallopian tube)
- International Federation of Gynecology and Obstetrics (FIGO) stage at time of initial diagnosis
- Baseline weight (in kilograms, last value prior to first dose; if weight is reported in pounds, convert to kilograms by dividing by 2.2)
- Baseline height (in centimeters, last value prior to first dose; if height is reported in inches, convert to centimeters by multiplying by 2.54)
- Baseline body mass index (BMI) (kg/m<sup>2</sup>), calculated using the patient's height and weight at Baseline [BMI (kg/m<sup>2</sup>) = weight (kg) / height (m)<sup>2</sup>]
- ECOG performance status at baseline
- History of myelosuppression (thrombocytopenia, leukopenia, anemia, or neutropenia) within the past year


- History of blood transfusion
- History of thrombocytopenia with grade 3 or 4 (repeated for leukopenia, anemia, and neutropenia)
- Prior ovarian cancer treatment, including number of prior lines of chemotherapy, number of prior platinum courses, any surgeries/procedures related to the study indication, number of surgeries, any radiotherapy prior to enrollment, response to last platinum-based therapy, PFI (months) after the last platinum-based therapy
- Histology and grade of disease at diagnosis and most recent biopsy, if additional biopsy performed
- BRCA and HRD status including:
  - o gBRCA-mut variant [BRCA1, BRCA2, Large rearrangement in BRCA1/2]
  - o tBRCA-mut variant [BRCA1, BRCA2]
  - BRCA status [BRCA-mut, gBRCA-mut and sBRCA-mut status within BRCA-mut; BRCA-wt; BRCA-unk]
  - o HRD status [HRD-pos, BRCA-mut and (BRCA-wt/BRCA-unk and HRD ≥42) within HRD-pos; HRD-neg; HRD-unk]
- Prior PARP treatment (yes, no)

Medical history will be coded using MedDRA v20.0 or later, and the number and percentage of patients experiencing at least 1 such diagnosis by MedDRA System Organ Class (SOC) and preferred term (PT) will be reported.

In addition, the following baseline subgroups will be presented for all patients, patients without prior PARP treatment and with prior PARP, respectively.

- BRCA status [BRCA-mut, BRCA-wt, BRCA-unk] by the response to the last platinum-based therapy
- HRD status [HRD-pos, HRD-neg, HRD-unk] by the response to the last platinum-based therapy

# 4.3. Efficacy Evaluation

4.3.1. Efficacy Variables for Primary and Key Secondary Analyses

The primary and key secondary efficacy analyses will be based on the investigator-assessed confirmed ORR per RECIST v1.1.

At each evaluation, the criteria in Table 4-1 were used to define each patient's overall response at that evaluation.


Table 4-1 Overall Response for Patients with Measureable Disease at Study Entry

| <b>Target Lesions</b> | Non-Target Lesions | New Lesions | Overall Response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/Non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-CR/Non-PD/Not evaluated | No | PR |
| SD | Non-CR/Non-PD/Not evaluated | No | SD |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

Abbreviations: CR = complete response; PD = progressive disease; PR = partial response; SD = stable disease.

As confirmed CR/PR is required, the best overall response (BOR) will be determined as shown in Table 4-2.

Given protocol scheduled tumor assessment interval is every 8 weeks ( $\pm 7$  days) from Cycle 1/Day 1 for 6 months and then every 12 weeks ( $\pm 7$  days) until progression. The minimum criteria for SD duration are at least 7 weeks from the date of first dose of study treatment.


Table 4-2: Best Overall Response when Confirmation of CR and PR Required

| Overall<br>Response First<br>Time Point | Overall Response Subsequent<br>Time Point (at least 4 weeks) | Best Overall Response |
|---|---|---|
| CR | CR | CR |
| CR | PR | SD provided minimum criteria for SD duration met, otherwise, PD |
| CR | SD | SD provided minimum criteria for SD duration met, otherwise, PD |
| CR | PD | SD provided minimum criteria for SD duration met, otherwise, PD |
| CR | NE | SD provided minimum criteria for SD duration met, otherwise, NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD provided minimum criteria for SD duration met, otherwise, NE |
| PR | PD | SD provided minimum criteria for SD duration met, otherwise, PD |
| PR | NE | SD provided minimum criteria for SD duration met, otherwise, NE |
| SD | SD | SD provided minimum criteria for SD duration met, otherwise, NE |
| SD | PD | SD provided minimum criteria for SD duration met, otherwise, PD |
| SD | NE | SD provided minimum criteria for SD duration met, otherwise, NE |
| NE | NE | NE |

Abbreviations: CR = complete response; NE = not evaluable; PD = progressive disease; PR = partial response; SD = stable disease.

For each patient, BOR will be determined based on the overall responses at all time points between the date of first dose and the date of first documented radiological disease progression, or the date of subsequent anti-cancer therapy, or the date of study discontinuation, whichever occurs first. Specifically:

- Day 1 can be determined from the "dose administration date" field on the "first dose" form.
- The date of radiological disease progression can be determined by selecting the earliest date from the "date of the radiological scan or assessment on which the response evaluation was based" field on the "evaluation of response (RECIST)" form where "overall response" = PD.
- Subsequent anti-cancer therapy can be determined by checking for any entries made on the "follow up anti-cancer therapy" form.


- The date of premature study discontinuation can be determined by using the "date of premature study discontinuation" field on the "premature study discontinuation" form. This date should be compared to the date on the "discontinuation of treatment" form where the primary reason for discontinuation is listed as "lost to follow up," "death," "sponsor decision to terminate study," or "patient withdrew consent." If these dates differ, select the earlier date.
- For each patient, select all "evaluation of response (RECIST)" forms meeting the following criteria:
  - The "date of the radiological scan or assessment on which the response evaluation was based" is after Day 1.
  - The "date of the radiological scan or assessment on which the response evaluation was based" is on or before the date of radiological disease progression, date that anti-cancer therapy first began, and the date of study discontinuation. If the patient did not experience radiological disease progression, begin anti-cancer therapy, or discontinue the study prematurely, select all forms after Day 1.

Patients with a BOR of either confirmed CR or PR are considered to have responded to treatment ("responders") for the primary efficacy variable (ORR). All other patients are considered to have not responded to treatment ("non-responders") for the primary efficacy variable.

The primary efficacy analysis will be testing the alternative hypothesis of  $ORR \ge 30\%$  will be tested against a null hypothesis of  $ORR \le 10\%$  in the HRD-positive patients who have received 3 or 4 prior lines of anti-cancer therapy and are platinum-sensitive to the last platinum-based therapy. Patients with prior PARP inhibitor treatment are excluded.

The key secondary efficacy analyses will be sequentially testing the alternative hypothesis of  $ORR \ge 25\%$  against a null hypothesis of  $ORR \le 10\%$  in:

- All patients who have received 3 or 4 prior lines of anti-cancer therapy and are platinum-sensitive to the last platinum-based therapy, regardless of HRD status (excluding patients with prior PARP treatment)
- All patients who have received 3 or 4 prior lines of anti-cancer therapy and are platinum-sensitive or platinum-resistant to the last platinum-based therapy, regardless of HRD status (excluding patients with prior PARP treatment)
- All patients treated in the study

The ORR and 2-sided 95% confidence interval along with a 1-sided p-value for testing the null hypothesis (one-sided alpha 0.025) based on the binomial distribution will be provided. The exact (Clopper-Pearson) method will be used to calculate 2-sided 95% CI. This can be programmed in SAS by appending the "/ BINOMIAL(EXACT)" option to the end of the appropriate "TABLE" statement.


The following subgroup analyses on ORR will be performed for the largest patient population achieving statistical significance among the sequential testing of primary and key secondary endpoints, and for all treated patients unless already available:

- Age categories [ $<65, \ge 65$ ]
- Primary tumor site [ovarian, primary peritoneal, fallopian tube]
- Response to last platinum-based therapy [platinum-sensitive, platinum-resistant, platinum-refractory, response-unknown]
- BRCA status [BRCA-mut, BRCA-wt, BRCA-unk]
- HRD status [HRD-pos, HRD-neg, HRD-unk]
- HRD-pos [BRCA-mut, (BRCA-wt/BRCA-unk and HRD score ≥42)]
- BRCA-mut [gBRCA-mut, sBRCA-mut]
- tBRCA-mut variant [BRCA1, BRCA2]
- gBRCA-mut variant [BRCA1, BRCA2, large rearrangement in BRCA1/2]
- Prior PARP treatment [yes, no]

### 4.3.2. Secondary Efficacy Variables

### 4.3.2.1. Duration of Response

For patients who responded to treatment, DOR (in months) is defined as the earliest date of initial response date of confirmed CR or PR to the earliest date of radiological PD or death, calculated as:

[Earliest date of radiological PD or death – Earliest of (Date of confirmed CR or PR) + 1] / 30.4375

Table 4-3 provides a summary of the censoring rules used in DOR analysis.

Table 4-3: Censoring Rules used in Duration of Response Analysis

| Situation | Date of Event or Censoring | Outcome |
|---|---|---|
| Start of subsequent anti-cancer therapy prior to a documented radiological progression or death | Date of last radiological tumor assessment prior to or on the date of initiation of the subsequent anti-cancer therapy | Censored |
| Free of radiological progression and no subsequent anti-cancer therapy started and no death | Date of last radiological tumor assessment | Censored |
| Documented radiological progression or death after 2 or more consecutive missing radiological assessments | Date of last radiological tumor assessment prior to the missed radiological assessment | Censored |
| Documented radiological progression or death | Earliest date of documented radiological progression or death | Event |

Details about defining CR, PR, PD, and end of study can be found in Section 4.3.1.


For each of the patient populations in the primary and key secondary endpoints, a time-to-event analysis of DOR will be performed respectively using KM methods including quartile estimates and 2-sided 95% CIs. A figure will be produced.

The same subgroup analyses performed for ORR will be performed for DOR.

#### 4.3.2.2. Disease Control Rate

Patients who achieved a best overall response rate of CR, PR, or SD (SD must have met the 7-week criteria described in Section 4.3.1) will be considered "responders" for this endpoint. All other patients will be considered "non-responders" for this endpoint. Details about defining best overall response rate can be found in Section 4.3.1.

For each of the patient populations in the primary and key secondary endpoints, the DCR and 2-sided 95% CI will be provided respectively. The exact (Clopper-Pearson) method will be used to calculate 95% CI. This can be programmed in SAS by appending the "/ BINOMIAL(EXACT)" option to the end of the appropriate "TABLE" statement.

### 4.3.2.3. Progression-Free Survival

Progressive disease (PD) will be determined based on RECIST criteria as defined in Section 4.3.1.

PFS (in months) is defined as the time from the date of first dose to the earlier date of radiological PD or death from any cause, calculated as:

[Earlier of (Date of radiological PD or death) – First dose date + 1] / 30.4375

Table 4-4 provides a summary of the censoring rules used in PFS analysis.

Table 4-4: Censoring Rules used in Progression-Free Survival Analysis

| Situation | Date of Event or Censoring | Outcome |
|---|---|---|
| No baseline tumor assessments | First dose date | Censored |
| No post-baseline tumor assessments and no death | First dose date | Censored |
| Start of subsequent anti-cancer therapy without a prior documented radiological progression or death | Date of last post-baseline radiological tumor assessment prior to or on the date of initiation of the subsequent anti-cancer therapy | Censored |
| Free of radiological progression and no subsequent anti-cancer therapy started and no death | Date of last post-baseline radiological tumor assessment | Censored |
| Documented radiological progression or death after 2 or more consecutive missing radiological assessments | Date of last post-baseline radiological tumor assessment prior to the missed radiological assessment | Censored |
| Documented radiological progression or death | Earliest date of radiological PD or death | Event |

For each of the patient populations in the primary and key secondary endpoints, a time-to-event analysis of PFS will be performed respectively using KM methods including quartile estimates and 2-sided 95% CIs. A figure will be produced.


### 4.3.2.4. Time to First Subsequent Therapy

TFST (in months) is defined as the date of first dose of study treatment in the current study to the earlier date of first dose of first subsequent therapy or death, calculated as:

[Earlier of (First dose of first subsequent therapy or death) – First dose date + 1] / 30.4375

Patients who are alive without a subsequent therapy will be censored on the last contact date.

For each of the patient populations in the primary and key secondary endpoints, a time-to-event analysis of TFST will be performed respectively using KM methods including quartile estimates and 2-sided 95% CIs. A figure will be produced.

#### 4 3 2 5 Overall Survival

Overall survival (in months) is defined as the time from the date of the first dose to the date of death for any cause, calculated as:

Patients who are known to be alive will be censored at the last contact date.

For each of the patient populations in the primary and key secondary endpoints, a time-to-event analysis of OS will be performed respectively using KM methods including quartile estimates and 2-sided 95% CIs. A figure will be produced.

#### 4.3.2.6. Pharmacokinetic Evaluations

Details of the population PK and intensive PK analyses, including combined analyses of the ECG variables and PK parameters, will be contained in a separate analysis plan.

## 4.4. Safety Analyses

Safety analyses will be conducted using the Safety population.

#### 4.4.1. Study Treatment Exposure

Extent of treatment will be summarized as follows:

- Number and percent of patients beginning 1, 2, 3, ..., 12, and >12 cycles.
- Number of cycles started summarized as a continuous variable.
- Overall treatment exposure (months), defined as the [last dose date first dose date + 1] / 30.4375, will be summarized and graphed both as a continuous and time-to-event variable.
- Time on study (months), defined as the [last visit date or date of death first dose date + 1] / 30.4375, will be summarized and graphed both as a continuous and time-to-event variable.

Intensity of study treatment:

• The total number of capsules consumed is the sum of the number of capsules dispensed less the sum of the number of capsules returned by the patient during the study. The sum of the daily doses consumed (mg) is the total number of capsules consumed multiplying by 100 mg. Unused capsules not returned will be assumed to have been consumed.


- Dose intensity (mg/day), defined as sum of the daily doses actually consumed divided by overall treatment exposure (converted to days), will be summarized as a continuous variable.
- Relative dose intensity (%), defined as dose intensity (mg/day) divided by intended dose intensity (mg/day), where intended dose intensity is 300 mg/day, will be summarized as a continuous variable.

Dose reductions and dose interruptions by cycle:

- Number and percentage of patients with a dose reduction, defined as the dose consumed is less than the dose prescribed, for any reason and due to an AE.
- Number and percentage of patients with a dose interruption, defined as the dose consumed is 0 mg, for any reason and due to an AE.

Dosing information for each patient will be presented in a data listing.

### 4.4.2. Study Treatment Compliance

Patient compliance with the study drug will be assessed via pill counts during the study.

For each cycle, study drug compliance (%) will be defined on the patient level by the dosing compliance ratio: the number of capsules consumed (the number of capsules dispensed less the number of capsules returned by the patient) divided by the number of capsules prescribed per protocol for a patieint in a cycle.

- Number of capsules dispensed per cycle is 93 capsules in a bottle throughout the trial. If the prescribed dose level at a cycle is unknown, assume both number of capsules prescribed and number of capsules dispensed at this cycle is 0. Otherwise:
  - Number of capsules prescribed for 300 mg/day per cycle is calculated by
     3 capsules per day multiplied by the actual treatment duration (day) in the cycle
  - Number of capsules prescribed for 200 mg/day per cycle is calculated by
     2 capsules per day multiplied by the actual treatment duration (day) in the cycle
  - Number of capsules prescribed for 100 mg/day per cycle is calculated by
     1 capsule per day multiplied by the actual treatment duration (day) in the cycle
  - The calculated number of capsules prescribed for a cycle will be capped at the maximum number of 93 capsules
- The treatment duration in a cycle *n* is calculated by the start date of dose prescribed at next cycle *n*+*I* minus the start date of dose prescribed at cycle *n*. If a patient discontinued study treatment during the cycle *n*, the treatment duration is calculated by the date of the last study dose minus the start date of dose prescribed at cycle *n*. The relevant data are in the eCRF pages: First Dose, Study Medication, and Discontinuation of Treatment.
  - If the treatment duration for a cycle can not be derived due to missing date, assume 28 days
  - o If the number of returned capsules is missing in a cycle, assume the number of capsules consumed to be the prescribed number of capsules/day (eg, 3/2/1 capsules per day) multiplied by the treatment duration in that cycle


- Any dose reduction in the middle of a cycle will not impact the compliance calculation in the current cycle. It will be taken into account for the compliance calculation at the next cycle as the reduced dose level will become the prescribed dose for that patient at the start of the next cycle.
- For any patients still ongoing with treatment at the time of analysis, compliance will be calculated up to and including the most recently completed cycle.

The overall study drug compliance (%) on the patient level is the total number of capsules consumed by a patient in all cycles divided by the total number of capsules prescribed per protocol for a patient in all cycles during the study.

A patient is evaluated as compliant if the patient has taken 80% to 120% of the prescribed capsules during the study. Study drug compliance rate (%) and the proportions of patients (<80%, 80%-120%, >120%) will be summarized.

#### 4.4.3. Adverse Events

#### 4.4.3.1. Overview

All AEs will be classified using MedDRA v20.0 or later. The severity of the toxicities will be graded according to the NCI CTCAE v4.03. Any AEs leading to death or discontinuation of study treatment, events classified as NCI CTCAE v4.03 Grade 3 or higher, study treatment-related events, and SAEs will be presented.

Any TEAEs will be defined as:

- Any new AE (one that was not seen prior to the start of treatment) that occurs for the first time after at least 1 dose of study treatment has been administered; or,
- A preexisting condition (one that was seen prior to the start of treatment) that worsens in severity (according to the CTCAE grade) after at least 1 dose of study treatment has been administered.
- Note: If the start date is missing for an AE and the actual start date cannot be determined from a partial date, the AE will be considered treatment-emergent.

All AEs will be collected from the time of signing the main ICF through the EOT visit. New SAEs (including deaths) will be collected for 30 days after the EOT visit. Any AEs recorded in the database that occur from the time of informed consent to first dose will be listed only and not included in safety analyses. Pre-existing conditions will be recorded in the eCRF on the Medical History or appropriate page.

Related TEAEs are defined as TEAEs considered likely related or related to treatment as judged by the Investigator. Any AEs for which the relationship to study drug is missing will be considered as related to study treatment.

The number and percentage of patients reporting a TEAE will be summarized by SOC, PT, toxicity grade, and relationship to study drug.

The toxicity grade of AEs as assessed by the investigator will be graded using NCI CTCAE v4.03. Within the same MedDRA PT, only the most severe AE for each patient will be counted in tabulations by severity. Within a MedDRA SOC, patients with more than 1 MedDRA PT will be counted only once for the most severe AE reported.


The relationship of each AE to the study drug will be summarized as assessed by the Investigator. All AEs for which the relationship to study drug is missing will be considered as related. Within the same MedDRA PT, only the AE with the highest ranked relationship to treatment for each patient will be counted in tabulations by relationship to treatment. Within a MedDRA SOC, patients with more than 1 MedDRA PT will be counted only once for the AE that is most related to treatment. The imputation for a missing relationship will take place prior to determining the most related AE within a SOC or PT for a given patient.

A high-level overview of AEs will be presented in a summary table. This table will include the number and percentage of patients for the following categories: any TEAE, any related TEAE, any grade  $\geq 3$  TEAE, any treatment-related grade  $\geq 3$  TEAE, any treatment-emergent serious adverse events (SAEs), any treatment-related serious TEAE, any AE leading to study drug interruption, any AE leading to study drug reduction, any AE leading to study drug withdrawal, any TEAE leading to death, and any pregnancies.

All AE tables will be summarized on the SAF population by 3-4 prior lines,  $\geq$ 5 prior lines, and Overall. Subgroup analyses of TEAEs will be conducted in the following subgroups on the SAF respectively by 3-4 prior lines,  $\geq$ 5 prior lines, and Overall:

- Age ( $<65 \text{ vs} \ge 65 \text{ years}$ )
- Primary tumor site (ovarian, peritoneal, fallopian tube)
- Response to last platinum-based therapy (platinum-sensitive, platinum-resistant, platinum-refractory, response-unknown)
- Patients with prior PARP treatment

The following lists the AE tables to be displayed; those designated with an '\*' will be produced for the subgroups described above.

- Overview of AEs\*
- TEAE by SOC and PT\*
- TEAE by PT (sorted by frequency)\*
- Related TEAE by SOC and PT
- Treatment-emergent SAEs by SOC and PT\*
- Related treatment-emergent SAEs by SOC and PT
- TEAE by SOC, PT, and maximum grade
- Related TEAE by SOC, PT, and maximum grade
- Grade ≥3 TEAEs by SOC and PT\*
- Grade ≥3 TEAEs by PT (sorted by frequency)\*
- Related Grade ≥3 TEAEs by SOC and PT
- TEAEs resulting in death by SOC and PT
- TEAEs resulting in study drug dose interruption by SOC and PT
- TEAEs resulting in study drug dose reduction by SOC and PT
- TEAEs resulting in study drug withdrawal by SOC and PT\*


- TEAEs of special interest (AESI) and other grouped events in Section 4.4.3.2, by the grouped event and PT within each group
  - All TEAEs\*
  - o Grade ≥3 TEAE\*
  - o SAEs
  - o TEAE resulting in dose interruption
  - o TEAE resulting in dose reduction
  - o TEAE resulting in study drug withdrawal
  - o Grade ≥3 TEAE resulting in study drug withdrawal
- Non-serious TEAEs ≥5% by SOC and PT (required by ClinicalTrials.gov)

Tables structured as listings will be provided for the following:

- Deaths
- SAEs
- TEAEs resulting in study drug interruption
- TEAEs resulting in study drug dose reduction
- TEAEs resulting in study drug withdrawn
- AESI and other grouped events
- Mapping of AE reported term to PT
- Patients developing MDS/AML; this listing will include the following:
  - Age and weight of patients with documented MDS/AML
  - o Number of previous chemotherapy regimens
  - Types of previous chemotherapies
  - o Time from last platinum therapy to start of study drug
  - o Prior history of myelosuppression
  - Myelosuppression AESIs on study
  - o Fluorescence in situ hybridization (FISH) result if available

Adverse event summaries will be ordered in terms of decreasing frequency for SOC (alphabetically for SOCs with the same number of AEs reported), and decreasing frequency for PT within SOC (alphabetically for PTs with the same number of AEs reported within a SOC).

# 4.4.3.2. Adverse Events of Special Interest

In the latest protocol amendment v8.0, the Adverse Events of Special Interest (AESIs) for this study are MDS, AML, secondary cancers (new malignancies other than MDS/AML), pneumonitis, and embryo-fetal toxicity.


#### 4.4.3.3. Other Adverse Events of Interest

In addition to AESIs, other AEs such as myelosuppression and hyptertension are also grouped for analysis. Table 4-5 outlines all the grouped events including AESIs with the criteria of mapping MedDRA PTs for each group using Standardized MedDRA Queries (SMQs), High Level Terms (HLTs), and/or PTs. A complete list of grouped events is provided in the Appendix (Section 7.1).

For TEAEs of special interest and other grouped events, the following analyses will be performed:

- Tabulations of all TEAEs, Grade ≥3 TEAEs, SAEs, TEAEs leading to dose interruption, dose reduction and withdrawal of study drug will be presented.
- A summary of all myelosuppression events and myelosuppression events ≥Grade 3 in severity will be produced to display the incidence of these events amongst patients with and without a prior history of myelosuppression.
- Tabulations of the thrombocytopenia event will be summarized by baseline platelet cutoffs.
- Tabulations of the anemia event will be summarized by baseline hemoglobin level.
- Tabulations of the thrombocytopenia, anemia, leukopenia, and neutropenia event will be summarized based on prior history of thrombocytopenia, anemia, leukopenia, and neutropenia event, respectively.
- Tabulations of all the AESI and other grouped events and ≥Grade 3 events for the subgroups described in the analysis of all TEAEs.
- A summary tabulation for patients who experienced thrombocytopenia event and who did and did not receive platelet transfusion (World Health Organization [WHO] drug preferred terms of platelets or platelets concentrated).
- A summary tabulation for patients who experienced anemia event and who did and did not receive red blood cell transfusion (WHO drug preferred terms of blood cells, packed human; red blood cells; red blood cells concentration; blood transfusion, auxiliary products) or who did and did not receive erythropoietin.
- A summary tabulation for patients who experienced neutropenia event and who did and did not receive colony stimulating factors (WHO drug preferred terms of filgrastim or granulocyte colony stimulating factor).
- A summary tabulation and a figure of time to first onset for each grouped event.
- The incidence of COVID-19 related AEs and SAEs will be summarized as part of the safety reporting summaries along with COVID-19-related as reasons for treatment discontinuation.
- A listing of all patients with COVID-19 assessments and symptom assessments will be produced and will include the following:
  - Treatment sequence
  - o Patient number
  - o COVID-19 case diagnosis


- o COVID-19 test performed
- o Result of the COVID-19 test
- Assessments and symptom assessments performed
- Results of the assessments and symptom assessments.

**Table 4-5:** Adverse Events of Special Interest and Other Grouped Events

| Group Term | MedDRA V18.1 Criteria for Selection of Preferred Terms <sup>1</sup> |
|---|---|
| Thrombocytopenia events | Haematopoietic thrombocytopenia SMQ (Broad) |
| Anemia events | Haematopoietic erythropenia SMQ (Broad) |
| Leukopenia events | Haematopoietic leukopenia SMQ (Broad) |
| Neutropenia events | Selected PTs related to neutropenia in the Haematopoietic leukopenia SMQ (Broad) |
| Pancytopenia events | Haematopoietic cytopenias SMQ (Broad) |
| AESI (MDS/AML events) | MedDRA PTs associated with MDS/AML |
| AESI (new malignancies other than MDS/AML) | Malignant tumor SMQ (other than MDS/AML) |
| AESI (pneumonitis) | Lower respiratory tract inflammatory and immunologic conditions (HLT) |
| AESI (embryo-fetal toxicity) | Pregnancy and neonatal topics SMQ |
| Hypertension events | Hypertension SMQ |

Abbreviations: AESI = adverse event of special interest; AML = acute myelogenous leukemia; HLT = high-level term; MDS = myelodysplastic syndrome; MedDRA = medical dictionary for regulatory activities; PT = preferred term; SMQ = Standardized MedDRA Query.

#### 4.4.3.4. Examination of Adverse Events Controlling for Duration of Drug Exposure

Since patients' duration of exposure to study drug will vary, AEs will also be presented as rates normalized for cumulative exposure. Total duration of exposure will be calculated as the last treatment date – first treatment date + 1.

In these tables, incidence rates per patient-exposure year (PEY) will be calculated as the number of patients experiencing an event in the numerator, and the total exposure time in PEY in the denominator. PEY is defined as follows: for each patient with the AE, the exposure-years will be the time of exposure to the drug in years at the time of first occurrence of the AE; for patients without the AE, the exposure-years will be defined as their total exposure in years on the study. For recurring events, the first occurrence of an AE (by MedDRA preferred term) will be reported.

The US Food and Drug Administration (FDA) guidance recommends examining AE incidence by cumulative exposure time (as discussed above), but notes that it is necessary to assume a constant risk of AEs across time for such analyses. If there is not a constant risk for a given AE, the incidence per PEY analysis would be biased. Therefore, a second method will be used to summarize AEs occurring by duration of exposure to study treatment within specific reporting intervals as defined by cycles of therapy. The number of patients on study—that is patients who


<sup>&</sup>lt;sup>1</sup> The list of preferred terms for each group is provided in the Appendix (Section 7.1).

have not withdrawn from the study, at the start of the reporting interval (number at risk)—will be used as the denominator for incidence and prevalence calculations.

Reporting of Incidence by Cycle: For incidence rates by cycle, the specific AE will be assigned to the relevant time period if the start date of the AE occurs within the period. For recurrent events during a reporting interval, the first event occurrence is reported. For events that recur in more than 1 reporting interval (event start date is in different reporting intervals), the event will be reported in the first applicable reporting interval. In addition, incidence adjusted for exposure on a per-interval basis will be performed. This analysis will calculate the cumulative exposure in patient-months up to the beginning of each interval, and divide the total number of patients with first incidence of the specific event in the interval by this cumulative exposure. Incidence of AESIs and the potentially bothersome gastrointestinal events of nausea and vomiting will be analyzed using these methods, for any severity event as well as for  $\geq$ Grade 3 events.

Reporting of Prevalence by Cycle: For prevalence rates by cycle, the specific AE will be assigned to the relevant time period if the AE occurs within the period, regardless of the interval in which the event started. For events that recur in more than 1 reporting interval (event occurs in different reporting intervals), the event will be reported in each applicable reporting interval. In addition, prevalence adjusted for exposure on a per-interval basis will be performed. This analysis will calculate the cumulative exposure in patient-months up to the beginning of each interval, and divide the total number of patients with any occurrence of the specific event in the interval by this cumulative exposure. Prevalence of AESIs and the gastrointestinal events of nausea and vomiting will be analyzed using these methods, for any severity event as well as for >Grade 3 events.

#### 4.4.3.5. Examination of Duration of Adverse Events

The duration of AESIs by category and the gastrointestinal events of nausea and vomiting will be calculated on a per-patient basis as the sum of the durations of each discrete episode of occurrence. The duration in days of overlapping occurrences will be calculated as the first start date to the last stop date +1. The average duration over patients for these events of any severity and of  $\geq$ Grade 3 severity will be summarized with descriptive statistics. Ongoing events will be censored at the time of the analysis cut-off date.

As individual events of long duration may be clinically relevant, the incidence of anemia events of  $\geq$ 28 days in duration for events of any severity and for events of  $\geq$ Grade 3 severity will be tabulated. In addition, events of  $\geq$ Grade 2 hematologic toxicities (defined as thrombocytopenia, leukopenia, neutropenia, or pancytopenia events)  $\geq$ 28 days with any grade anemia  $\geq$ 28 days will be summarized. Note that these durations are for specific instances of the event, and not based on cumulative time with the event. Incidence categories of 0, 1, 2, 3, and 4 or more will be summarized.

### 4.4.4. Laboratory Data

Laboratory assessments will be performed locally at each center's laboratory by means of their established methods. All laboratory values will be converted to SI units and classified as normal, low, or high based on normal ranges supplied by the local laboratories. Laboratory assessments will be assigned to cycles based on the start date of the cycle based on exposure data.

Hematologic and chemistry laboratory results will be graded according to the cut points defined in the NCI CTCAE v4.03 severity grade. Laboratory results will be summarized by maximum


CTCAE grade as available. For platelet count decrease, an additional category for CTCAE v4.03 will be included for values that are  $<\!10,\!000/\mu L$ . Continuous results will be analyzed using change from baseline and shift values.

Change from baseline will be summarized and analyzed according to the largest increase, decrease, and at EOT, irrespective of scheduled or unscheduled visit. Graphical line mean changes over time may be provided, but due to the varying visits, no repeated measures analysis will be performed.

Shift from baseline to the smallest, largest, and EOT will be reported using number and percentage of patients. Baseline and post-baseline results will be categorized as low, normal, or high relative to the normal range, or by CTCAE grade as applicable.

A listing of potential Hy's Law cases (patients with AST or ALT  $>3 \times$  upper limit of normal [ULN] in combination with bilirubin  $>2 \times$  ULN and ALP within normal range or  $\le 1.5 \times$  ULN) will be also presented. Additionally, a Hy's Law (DILI) plot will be produced which plots peak ALT and peak total bilirubin in 1 panel and peak AST and peak total bilirubin in a second panel.

A distribution boxplot of liver function test (albumin, ALT, AST, alkaline phosphatase, total bilirubin, direct bilirubin and GGT) and selected hematology and other chemistry laboratory test values over time will be presented. A side panel will be added to the plot to show the distribution of maximum values.

A by-patient listing of all laboratory data will be provided, with laboratory reference ranges and abnormal values highlighted, and including center, patient identifier, and visit.

# 4.4.5. Vital Signs and Physical Examination

Summaries of vital signs parameters (systolic and diastolic blood pressures, pulse rate, and temperature) and weight will be presented by visit. Summary statistics will be produced for both observed and change from baseline values, for each parameter.

Change from baseline will be summarized and analyzed according to the largest increase, decrease, and at the end of treatment, irrespective of scheduled or unscheduled visit. Graphical line mean changes over time may be provided, but due to the varying visits no repeated measures analysis will be performed.

Vital sign measurements will be presented for each patient in a data listing.

The number and percentage of patients experiencing at least 1 abnormal result at the baseline physical examination will be summarized by body system. Subsequent symptom-targeted physical examination findings will be presented for each patient in a data listing.

All physical examination findings will be presented in a data listing.

### 4.4.6. Electrocardiogram

All patients will undergo a single ECG assessment at the screening visit. A subset of approximately 12 patients will undergo intensive, triplicate ECG monitoring to coincide with PK evaluation on Cycle 1/Day 1 and all other assessments in the study. The average of each of the triplicate measures will be used for analysis.

Any ECG findings that were assessed as clinically significant and were reported as an AE or SAE will be summarized in the tables and listings.


Electrocardiogram results will be summarized descriptively. Baseline will be defined as the average of the closest triplicate (if triplicates were collected) readings prior to dosing on the first day that study drug is administered.

Electrocardiogram measurements including PR interval, QT interval, RR interval, and QRS complex will be collected.

QTc will be used for the data analysis and interpretation. Commonly used techniques including Bazett's (QTcB) and Fridericia's (QTcF) methods are applied. QTcF will be used for the primary QT evaluation. A summary of the number and percentage of patients with QTc interval exceeding some predefined upper limit (eg, >450 ms, >480 ms, >500 ms) will be provided. A summary of the number and percentage of patients with change from baseline in QTc interval exceeding some predefined upper limit (eg, >30 ms, >60 ms) will be provided. A separate summary will be provided which summarizes the change from baseline to the most extreme high or low value at any time during treatment. Change from baseline will be summarized and analyzed according to the largest increase, decrease, and at EOT, irrespective of scheduled or unscheduled visit. Graphical line mean changes over time may be provided.

No values will be imputed for missing data except for averaging of triplicate measurements. If 1 or 2 of the triplicate measurements for an ECG parameter are missing, the average of the remaining 2 measurements or the single measurement will be used in analyses. If all triplicate measurements are missing at a time point for an ECG parameter, no values will be imputed for this time point and no analyses related to this time point will be performed. If the triplicate is not good because of an artifact, then if the triplicate is repeated within about  $\pm 15$  minutes, it can be used at that nominal time. Patients who have data on other days or unscheduled ECGs but not at the scheduled time points will be included in the categorical tables but not the statistical analyses.

All ECG data for each patient will be provided in a data listing.

### 4.4.7. Concomitant Medications

All medications will be coded using the September 2017 or later version of the WHO Drug Dictionary (WHODD). Medication start and stop dates will be compared to the date of first dose of study drug to allow medications to be classified as either Prior only, both Prior and Concomitant, or Concomitant only. Medications starting after the treatment withdrawal date will be listed but will not be classified or summarized.

Medications that start and stop prior to the date of first dose of study drug will be classified as Prior only. If a medication starts before the date of first dose of study drug and stops on or after the date of first dose of study drug, then the medication will be classified as both Prior and Concomitant. Medications will be classified as Concomitant only if they have a start date on or after the date of first dose of study drug. Concomitant medication will be summarized by ATC level 3 and PT in frequency tables by treatment. Patients with more than 1 medication in a given ATC level and PT will be counted only once in that category.

If medication start and/or stop dates are missing or partial, the dates will be compared as far as possible with the date of first dose of study drug. Medications will be assumed to be Concomitant only, unless there is clear evidence (through comparison of partial dates) to suggest that the medication started prior to the first dose of study drug. If there is clear evidence to suggest that the medication started prior to the first dose of study drug, the medication will be assumed to be both Prior and Concomitant, unless there is clear evidence to suggest that the


medication stopped prior to the first dose of study drug. If there is clear evidence to suggest that the medication stopped prior to the first dose of study drug, the medication will be assumed to be Prior only. The following lists the concomitant medication tables to be displayed:

- Number and percentage with at least 1 prior medication by ATC level 3 and PT
- Number and percentage with at least 1 concomitant medication by ATC level 3 and PT
- Number and percentage with at least 1 prior and concomitant medication by ATC level 3 and PT

The use of concomitant medications will be included in a by-patient data listing.


## 5. CHANGES TO PLANNED ANALYSES

As of this date, there have been no changes between the protocol-defined statistical analyses and those presented in this SAP.

If any modifications in the experimental design, dosages, parameters, patient selection, or any other sections of the protocol are indicated or required, the Investigator will consult with the Sponsor before such changes are instituted. Modifications will be accomplished through formal amendments to this protocol by the Sponsor and approval from the appropriate Institutional Review Board (IRB) or Independent Ethics Committee (IEC).


## 6. REFERENCES

- Fong, P.C., et al., Inhibition of poly(ADP-ribose) polymerase in tumors from BRCA mutation carriers. N Engl J Med, 2009. 361(2): p. 123-34.
- Audeh, M.W., et al., Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with BRCA1 or BRCA2 mutations and recurrent ovarian cancer: a proof-of-concept trial. Lancet, 2010. 376(9737): p. 245-51.
- Gelmon, K.A., et al., Olaparib in patients with recurrent high-grade serous or poorly differentiated ovarian carcinoma or triple-negative breast cancer: a phase 2, multicentre, open-label, non-randomised study. Lancet Oncol, 2011. 12(9): p. 852-61.
- Kummar, S., et al., A phase I study of veliparib in combination with metronomic cyclophosphamide in adults with refractory solid tumors and lymphomas. Clin Cancer Res, 2012. 18(6): p. 1726-34.
- Ledermann, J., et al., Olaparib maintenance therapy in platinum-sensitive relapsed ovarian cancer. N Engl J Med, 2012. 366(15): p. 1382-92.
- Ledermann, J., et al., Olaparib maintenance therapy in patients with platinum-sensitive relapsed serous ovarian cancer: a preplanned retrospective analysis of outcomes by BRCA status in a randomised phase 2 trial. Lancet Oncol, 2014. 15(8): p. 852-61.
- Sandhu, S.K., et al., The poly(ADP-ribose) polymerase inhibitor niraparib (MK4827) in BRCA mutation carriers and patients with sporadic cancer: a phase 1 dose-escalation trial. Lancet Oncol, 2013. 14(9): p. 882-92.
- US Federal Register. International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D 0174]. Federal Register Volume 63, Number, pages 49583 49598. September 16, 1998.


# 7. APPENDIX

# 7.1. MedDRA Preferred Terms for Adverse Events of Special Groups


| AE Category<br>MedDRA Level | Preferred Terms | SMQ<br>Scope |
|---|---|---|
| | Primary myelofibrosis | Broad |
| | Scan bone marrow abnormal | Broad |
| MDS/AML Event: | | |
| MedDRA PTs as listed | Myelodysplastic syndrome | NA |
| | Myelodysplastic syndrome transformation | NA |
| | Myelodysplastic syndrome unclassifiable | NA |
| | Acute myeloid leukaemia | NA |
| | Acute myeloid leukaemia recurrent | NA |
| | Blast crisis in myelogenous leukaemia | NA |
| | Myeloid leukaemia | NA |
| New malignancies other than MDS/AML | See Section 7.2 | |
| Malignant Tumours (SMQ) [20000194] | | |
| Pneumonitis Event: | | |
| Lower respiratory tract inflammatory and | Pneumonitis | NA |
| immunologic conditions (HLT) | Acute interstitial pneumonitis | NA |
| Embryo-fetal toxicity | See Section 7.3 | |
| Pregnancy and neonatal topics (SMQ) [20000185] | | |
| Hypertension Event: | See Section 7.4 | |
| Hypertension SMQ [20000147] | | |

Abbreviations: AE = adverse event; AML = acute myelogenous leukemia; HLT = high-level term; MDS = myelodysplastic syndrome; MedDRA = medical dictionary for regulatory activities; PT = preferred term; SMQ = Standardized MedDRA Query.


<sup>\*</sup> Preferred terms are included in the Neutropenia Event.

# 7.2. SMQ Terms for Malignant Tumors

SMQ Export: 20.1 - English 1/8/2018 2:20:21 PM

Include Inactive PT: No

Term Attributes: Name, Code, Level, Scope, Category, Weight, Status, Addition Version, Last Modified Version

Malignant tumours (SMQ) [20000194]

Haematological malignant tumours (SMQ) [20000227]

| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| Name | Code | Level | Scope | y | t | Status | Version | Version |
| | 1006853 | | Narro | | | | | |
| 5q minus syndrome | 2 | PT | W | A | 0 | Active | 11.1 | 20.0 |
| | 1006739 | | Narro | | | | | |
| Acute biphenotypic leukaemia | 9 | PT | W | A | 0 | Active | 10.1 | 20.0 |
| | 1000083 | | Narro | | | | | |
| Acute leukaemia | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006093 | | Narro | | | | | |
| Acute leukaemia in remission | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000084 | | Narro | | | | | |
| Acute lymphocytic leukaemia | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000084 | | Narro | | | | | |
| Acute lymphocytic leukaemia (in remission) | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006362 | | Narro | | | | | |
| Acute lymphocytic leukaemia recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007686 | | Narro | | | | | |
| Acute lymphocytic leukaemia refractory | 6 | PT | W | A | 0 | Active | 18.1 | 20.0 |
| | 1000086 | | Narro | | | | | |
| Acute megakaryocytic leukaemia | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005719 | | Narro | | | | | |
| Acute megakaryocytic leukaemia (in remission) | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000087 | | Narro | | | | | |
| Acute monocytic leukaemia | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000087 | | Narro | | | | | |
| Acute monocytic leukaemia (in remission) | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000088 | | Narro | | | | | |
| Acute myeloid leukaemia (in remission) | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1000089 | | Narro | | | | | |
| Acute myelomonocytic leukaemia | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000101 | | Narro | | | | | |
| Acute promyelocytic leukaemia | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007347 | | Narro | | | | | |
| Acute undifferentiated leukaemia | 9 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1000141 | | Narro | | | | | |
| Adult T-cell lymphoma/leukaemia | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000141 | | Narro | | | | | |
| Adult T-cell lymphoma/leukaemia recurrent | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000141 | | Narro | | | | | |
| Adult T-cell lymphoma/leukaemia refractory | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000141 | | Narro | | | | | |
| Adult T-cell lymphoma/leukaemia stage I | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000141 | | Narro | | | | | |
| Adult T-cell lymphoma/leukaemia stage II | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000142 | | Narro | | | | | |
| Adult T-cell lymphoma/leukaemia stage III | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000142 | | Narro | | | | | |
| Adult T-cell lymphoma/leukaemia stage IV | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000166 | | Narro | | | | | |
| Aleukaemic leukaemia | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000222 | | Narro | | | | | |
| Anaplastic large cell lymphoma T- and null-cell types | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Anaplastic large cell lymphoma T- and null-cell types | 1000222 | | Narro | | | | | |
| recurrent | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Anaplastic large cell lymphoma T- and null-cell types | 1000223 | | Narro | | | | | |
| refractory | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Anaplastic large cell lymphoma T- and null-cell types | 1000223 | | Narro | | | | | |
| stage I | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Anaplastic large cell lymphoma T- and null-cell types | 1000223 | | Narro | | | | | |
| stage II | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Anaplastic large cell lymphoma T- and null-cell types | 1000223 | | Narro | | | | | |
| stage III | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| Anaplastic large cell lymphoma T- and null-cell types | 1000223 | | Narro | | | | | |
| stage IV | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007347 | | Narro | | | | | |
| Anaplastic large-cell lymphoma | 8 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1000241 | | Narro | | | | | |
| Angiocentric lymphoma | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000241 | | Narro | | | | | |
| Angiocentric lymphoma recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000241 | | Narro | | | | | |
| Angiocentric lymphoma refractory | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000241 | | Narro | | | | | |
| Angiocentric lymphoma stage I | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000241 | | Narro | | | | | |
| Angiocentric lymphoma stage II | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000241 | | Narro | | | | | |
| Angiocentric lymphoma stage III | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000241 | | Narro | | | | | |
| Angiocentric lymphoma stage IV | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000244 | | Narro | | | | | |
| Angioimmunoblastic T-cell lymphoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000245 | | Narro | | | | | |
| Angioimmunoblastic T-cell lymphoma recurrent | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000245 | | Narro | | | | | |
| Angioimmunoblastic T-cell lymphoma refractory | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000245 | | Narro | | | | | |
| Angioimmunoblastic T-cell lymphoma stage I | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000245 | | Narro | | | | | |
| Angioimmunoblastic T-cell lymphoma stage II | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000245 | | Narro | | | | | |
| Angioimmunoblastic T-cell lymphoma stage III | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000245 | | Narro | | | | | |
| Angioimmunoblastic T-cell lymphoma stage IV | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000389 | | Narro | | | | | |
| B precursor type acute leukaemia | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1000389 | | Narro | | | | | |
| B-cell lymphoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000390 | | Narro | | | | | |
| B-cell lymphoma recurrent | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000390 | | Narro | | | | | |
| B-cell lymphoma refractory | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000390 | | Narro | | | | | |
| B-cell lymphoma stage I | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000390 | | Narro | | | | | |
| B-cell lymphoma stage II | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000390 | | Narro | | | | | |
| B-cell lymphoma stage III | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000390 | | Narro | | | | | |
| B-cell lymphoma stage IV | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007348 | | Narro | | | | | |
| B-cell prolymphocytic leukaemia | 0 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1000390 | | Narro | | | | | |
| B-cell small lymphocytic lymphoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000391 | | Narro | | | | | |
| B-cell small lymphocytic lymphoma recurrent | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000391 | | Narro | | | | | |
| B-cell small lymphocytic lymphoma refractory | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000391 | | Narro | | | | | |
| B-cell small lymphocytic lymphoma stage I | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000391 | | Narro | | | | | |
| B-cell small lymphocytic lymphoma stage II | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000391 | | Narro | | | | | |
| B-cell small lymphocytic lymphoma stage III | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000391 | | Narro | | | | | |
| B-cell small lymphocytic lymphoma stage IV | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| · | 1000391 | | Narro | | | | | |
| B-cell type acute leukaemia | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000392 | | Narro | | | | | |
| B-cell unclassifiable lymphoma high grade | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1000392 | | Narro | | | | | |
| B-cell unclassifiable lymphoma low grade | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005028 | | Narro | | | | | |
| Blast crisis in myelogenous leukaemia | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007546 | | Narro | | | | | |
| Blastic plasmacytoid dendritic cell neoplasia | 0 | PT | W | A | 0 | Active | 17.1 | 20.0 |
| | 1004955 | | Narro | | | | | |
| Bone marrow leukaemic cell infiltration | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004955 | | Narro | | | | | |
| Bone marrow tumour cell infiltration | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006718 | | Narro | | | | | |
| Burkitt's leukaemia | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000659 | | Narro | | | | | |
| Burkitt's lymphoma | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000659 | | Narro | | | | | |
| Burkitt's lymphoma recurrent | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000659 | | Narro | | | | | |
| Burkitt's lymphoma refractory | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000660 | | Narro | | | | | |
| Burkitt's lymphoma stage I | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000660 | | Narro | | | | | |
| Burkitt's lymphoma stage II | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000660 | | Narro | | | | | |
| Burkitt's lymphoma stage III | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000660 | | Narro | | | | | |
| Burkitt's lymphoma stage IV | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006623 | | Narro | | | | | |
| Central nervous system leukaemia | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000795 | | Narro | | | | | |
| Central nervous system lymphoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000858 | | Narro | | | | | |
| Chloroma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000858 | | Narro | | | | | |
| Chloroma (in remission) | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006585 | | Narro | | | | | |
| Chronic eosinophilic leukaemia | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000894 | | Narro | | | | | |
| Chronic leukaemia | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006104 | | Narro | | | | | |
| Chronic leukaemia in remission | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000895 | | Narro | | | | | |
| Chronic lymphocytic leukaemia | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000895 | | Narro | | | | | |
| Chronic lymphocytic leukaemia (in remission) | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000896 | | Narro | | | | | |
| Chronic lymphocytic leukaemia recurrent | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000896 | | Narro | | | | | |
| Chronic lymphocytic leukaemia refractory | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000896 | | Narro | | | | | |
| Chronic lymphocytic leukaemia stage 0 | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000896 | | Narro | | | | | |
| Chronic lymphocytic leukaemia stage 1 | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000896 | | Narro | | | | | |
| Chronic lymphocytic leukaemia stage 2 | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000896 | | Narro | | | | | |
| Chronic lymphocytic leukaemia stage 3 | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000896 | | Narro | | | | | |
| Chronic lymphocytic leukaemia stage 4 | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005871 | | Narro | | | | | |
| Chronic lymphocytic leukaemia transformation | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000901 | | Narro | | | | | |
| Chronic myeloid leukaemia | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000901 | | Narro | | | | | |
| Chronic myeloid leukaemia (in remission) | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007508 | | Narro | | | | | |
| Chronic myeloid leukaemia recurrent | 1 | PT | W | A | 0 | Active | 17.1 | 20.0 |
| | 1006823 | | Narro | | | | | |
| Chronic myeloid leukaemia transformation | 2 | PT | W | A | 0 | Active | 11.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1000901 | | Narro | | | | | |
| Chronic myelomonocytic leukaemia | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000901 | | Narro | | | | | |
| Chronic myelomonocytic leukaemia (in remission) | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007395 | | Narro | | | | | |
| Composite lymphoma | 7 | PT | W | A | 0 | Active | 16.1 | 20.0 |
| | 1007994 | | Narro | | | | | |
| Cutaneous lymphoma | 5 | PT | W | A | 0 | Active | 20.1 | 20.1 |
| | 1001281 | | Narro | | | | | |
| Diffuse large B-cell lymphoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001282 | | Narro | | | | | |
| Diffuse large B-cell lymphoma recurrent | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001282 | | Narro | | | | | |
| Diffuse large B-cell lymphoma refractory | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001282 | | Narro | | | | | |
| Diffuse large B-cell lymphoma stage I | 3 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1001282 | | Narro | | | | | |
| Diffuse large B-cell lymphoma stage II | 4 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1001282 | | Narro | | | | | |
| Diffuse large B-cell lymphoma stage III | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001282 | | Narro | | | | | |
| Diffuse large B-cell lymphoma stage IV | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005495 | | Narro | | | | | |
| Disseminated large cell lymphoma | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1008020 | | Narro | | | | | |
| Double hit lymphoma | 2 | PT | W | A | 0 | Active | 20.1 | 20.1 |
| | 1007348 | | Narro | | | | | |
| Enteropathy-associated T-cell lymphoma | 1 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1001495 | | Narro | | | | | |
| Eosinophilic leukaemia | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007144 | | Narro | | | | | |
| Epstein-Barr virus associated lymphoma | 1 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1001524 | | Narro | | | | | |
| Erythraemic myelosis (in remission) | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1001528 | | Narro | | | | | |
| Erythroleukaemia | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Extranodal marginal zone B-cell lymphoma (MALT | 1006185 | | Narro | | | | | |
| type) | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Extranodal marginal zone B-cell lymphoma (MALT | 1001582 | | Narro | | | | | |
| type) recurrent | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Extranodal marginal zone B-cell lymphoma (MALT | 1001582 | | Narro | | | | | |
| type) refractory | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Extranodal marginal zone B-cell lymphoma (MALT | 1001582 | | Narro | | | | | |
| type) stage I | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Extranodal marginal zone B-cell lymphoma (MALT | 1001582 | | Narro | | | | | |
| type) stage II | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Extranodal marginal zone B-cell lymphoma (MALT | 1001582 | | Narro | | | | | |
| type) stage III | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Extranodal marginal zone B-cell lymphoma (MALT | 1001582 | | Narro | | | | | |
| type) stage IV | 8 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1006195 | | Narro | | | | | |
| Follicle centre lymphoma diffuse small cell lymphoma | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma diffuse small cell lymphoma | 1001689 | | Narro | | | | | |
| recurrent | 7 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma diffuse small cell lymphoma | 1001689 | | Narro | | | | | |
| refractory | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma diffuse small cell lymphoma | 1001689 | | Narro | | | | | |
| stage I | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma diffuse small cell lymphoma | 1001690 | | Narro | | | | | |
| stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma diffuse small cell lymphoma | 1001690 | | Narro | | | | | |
| stage III | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma diffuse small cell lymphoma | 1001690 | | Narro | | | | | |
| stage IV | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006117 | | Narro | | | | | |
| Follicle centre lymphoma, follicular grade I, II, III | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma, follicular grade I, II, III | 1001690 | | Narro | | | | | |
| recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| Follicle centre lymphoma, follicular grade I, II, III | 1001690 | | Narro | | | | | |
| refractory | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma, follicular grade I, II, III stage | 1001690 | | Narro | | | | | |
| I | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma, follicular grade I, II, III stage | 1001690 | | Narro | | | | | |
| II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma, follicular grade I, II, III stage | 1001690 | | Narro | | | | | |
| III | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Follicle centre lymphoma, follicular grade I, II, III stage | 1001691 | | Narro | | | | | |
| IV | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007533 | | Narro | | | | | |
| Follicular dendritic cell sarcoma | 2 | PT | w | A | 0 | Active | 17.1 | 20.0 |
| | 1001797 | | Narro | | | | | |
| Gastrointestinal lymphoma | 3 | PT | w | A | 0 | Active | 10.0 | 20.1 |
| | 1006647 | | Narro | | | | | |
| Haematological malignancy | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001905 | | Narro | | | | | |
| Hairy cell leukaemia | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007740 | | Narro | | | | | |
| Hairy cell leukaemia recurrent | 3 | PT | W | Α | 0 | Active | 19.0 | 20.0 |
| | 1006695 | | Narro | | | | | |
| Hepatosplenic T-cell lymphoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002006 | | Narro | | | | | |
| High grade B-cell lymphoma Burkitt-like lymphoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| High grade B-cell lymphoma Burkitt-like lymphoma | 1002007 | | Narro | | | | | |
| recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| High grade B-cell lymphoma Burkitt-like lymphoma | 1002007 | | Narro | | | | | |
| refractory | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| High grade B-cell lymphoma Burkitt-like lymphoma | 1002007 | | Narro | | | | | |
| stage I | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| High grade B-cell lymphoma Burkitt-like lymphoma | 1002007 | | Narro | | | | | |
| stage II | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| High grade B-cell lymphoma Burkitt-like lymphoma | 1002007 | | Narro | | | | | |
| stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| High grade B-cell lymphoma Burkitt-like lymphoma | 1002007 | | Narro | | | | | |
| stage IV | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1008021 | | Narro | | | | | |
| High-grade B-cell lymphoma | 5 | PT | W | A | 0 | Active | 20.1 | 20.1 |
| | 1006878 | | Narro | | | | | |
| Histiocytic medullary reticulosis | 5 | PT | W | A | 0 | Active | 12.0 | 20.0 |
| | 1007687 | | Narro | | | | | |
| Histiocytic sarcoma | 6 | PT | w | A | 0 | Active | 18.1 | 20.0 |
| | 1002020 | | Narro | | | | | |
| Hodgkin's disease | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte depletion stage I site | 1002020 | | Narro | | | | | |
| unspecified | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte depletion stage I | 1002020 | | Narro | | | | | |
| subdiaphragm | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte depletion stage I | 1002021 | | Narro | | | | | |
| supradiaphragm | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte depletion stage II site | 1002021 | | Narro | | | | | |
| unspecified | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte depletion stage II | 1002021 | | Narro | | | | | |
| subdiaphragm | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte depletion stage II | 1002021 | | Narro | | | | | |
| supradiaphragm | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002021 | | Narro | | | | | |
| Hodgkin's disease lymphocyte depletion type recurrent | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002021 | | Narro | | | | | |
| Hodgkin's disease lymphocyte depletion type refractory | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002021 | | Narro | | | | | |
| Hodgkin's disease lymphocyte depletion type stage III | 7 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1002021 | | Narro | | | | | |
| Hodgkin's disease lymphocyte depletion type stage IV | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte depletion type stage | 1002021 | | Narro | | | | | |
| unspecified | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance stage I site | 1002022 | | Narro | | | | | |
| unspec | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| Hodgkin's disease lymphocyte predominance stage I subdiaphragm | 1002022<br>1 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance stage I supradiaphragm | 1002022 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance stage II site unspec | 1002022 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance stage II subdiaphragm | 1002022<br>4 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance stage II supradiaphragm | 1002022<br>5 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance type recurrent | 1002022<br>7 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance type refractory | 1002022<br>8 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance type stage III | 1002022<br>9 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance type stage IV | 1002023<br>0 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease lymphocyte predominance type stage unspecified | 1002023<br>1 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease mixed cellularity recurrent | 1002023 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease mixed cellularity refractory | 1002023<br>4 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease mixed cellularity stage I site unspecified | 1002023<br>5 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease mixed cellularity stage I subdiaphragmatic | 1002023<br>6 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease mixed cellularity stage I supradiaphragmatic | 1002023<br>7 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease mixed cellularity stage II subdiaphragmatic | 1002023<br>8 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Hodgkin's disease mixed cellularity stage II supradiaphragmatic | 1002023 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002024 | | Narro | | | | | |
| Hodgkin's disease mixed cellularity stage III | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002024 | | Narro | | | | | |
| Hodgkin's disease mixed cellularity stage IV | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002024 | | Narro | | | | | |
| Hodgkin's disease mixed cellularity stage unspecified | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002024 | | Narro | | | | | |
| Hodgkin's disease nodular sclerosis | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002024 | | Narro | | | | | |
| Hodgkin's disease nodular sclerosis recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002024 | | Narro | | | | | |
| Hodgkin's disease nodular sclerosis refractory | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007353 | | Narro | | | | | |
| Hodgkin's disease nodular sclerosis stage I | 5 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007353 | | Narro | | | | | |
| Hodgkin's disease nodular sclerosis stage II | 4 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1002025 | | Narro | | | | | |
| Hodgkin's disease nodular sclerosis stage III | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002025 | | Narro | | | | | |
| Hodgkin's disease nodular sclerosis stage IV | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002026 | | Narro | | | | | |
| Hodgkin's disease recurrent | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002026 | | Narro | | | | | |
| Hodgkin's disease refractory | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002026 | | Narro | | | | | |
| Hodgkin's disease stage I | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002026 | | Narro | | | | | |
| Hodgkin's disease stage II | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002027 | | Narro | | | | | |
| Hodgkin's disease stage III | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006159 | | Narro | | | | | |
| Hodgkin's disease stage IV | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002027 | | Narro | | | | | |
| Hodgkin's disease unclassifiable | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1005357 | | Narro | | | | | |
| Immunoblastic lymphoma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002270 | | Narro | | | | | |
| Intestinal T-cell lymphoma recurrent | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002270 | | Narro | | | | | |
| Intestinal T-cell lymphoma refractory | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002270 | | Narro | | | | | |
| Intestinal T-cell lymphoma stage I | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002270 | | Narro | | | | | |
| Intestinal T-cell lymphoma stage II | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002271 | | Narro | | | | | |
| Intestinal T-cell lymphoma stage III | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002271 | | Narro | | | | | |
| Intestinal T-cell lymphoma stage IV | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002324 | | Narro | | | | | |
| Juvenile chronic myelomonocytic leukaemia | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007828 | | Narro | | | | | |
| Leptomeningeal myelomatosis | 2 | PT | W | A | 0 | Active | 19.1 | 20.0 |
| | 1002428 | | Narro | | | | | |
| Leukaemia | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002429 | | Narro | | | | | |
| Leukaemia basophilic | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005318 | | Narro | | | | | |
| Leukaemia cutis | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002429 | | Narro | | | | | |
| Leukaemia granulocytic | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006122 | | Narro | | | | | |
| Leukaemia in remission | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002430 | | Narro | | | | | |
| Leukaemia monocytic | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006248 | | Narro | | | | | |
| Leukaemia recurrent | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007756 | | Narro | | | | | |
| Leukaemic cardiac infiltration | 3 | PT | W | A | 0 | Active | 19.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006936 | | Narro | | | | | |
| Leukaemic infiltration | 0 | PT | W | A | 0 | Active | 12.1 | 20.0 |
| | 1006711 | | Narro | | | | | |
| Leukaemic infiltration extramedullary | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006743 | | Narro | | | | | |
| Leukaemic infiltration gingiva | 1 | PT | W | A | 0 | Active | 10.1 | 20.0 |
| | 1005867 | | Narro | | | | | |
| Leukaemic infiltration hepatic | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007585 | | Narro | | | | | |
| Leukaemic infiltration ovary | 3 | PT | W | A | 0 | Active | 18.0 | 20.0 |
| | 1005236 | | Narro | | | | | |
| Leukaemic infiltration pulmonary | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006935 | | Narro | | | | | |
| Leukaemic infiltration renal | 9 | PT | W | A | 0 | Active | 12.1 | 20.0 |
| | 1002432 | | Narro | | | | | |
| Leukaemic lymphoma | 5 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1005923 | | Narro | | | | | |
| Leukaemic retinopathy | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002522 | | Narro | | | | | |
| Lymphangiosarcoma | 3 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1005313 | | Narro | | | | | |
| Lymphangiosis carcinomatosa | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002527 | | Narro | | | | | |
| Lymphocytic leukaemia | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005217 | | Narro | | | | | |
| Lymphocytic lymphoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002530 | | Narro | | | | | |
| Lymphoid leukaemia (in remission) | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002531 | | Narro | | | | | |
| Lymphoma | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002531 | | Narro | | | | | |
| Lymphoma AIDS related | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005170 | | Narro | | | | | |
| Lymphoma cutis | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006434 | | Narro | | | | | |
| Lymphoma transformation | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002534 | | Narro | | | | | |
| Lymphoplasmacytoid lymphoma/immunocytoma | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Lymphoplasmacytoid lymphoma/immunocytoma | 1002534 | | Narro | | | | | |
| recurrent | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Lymphoplasmacytoid lymphoma/immunocytoma | 1002534 | | Narro | | | | | |
| refractory | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Lymphoplasmacytoid lymphoma/immunocytoma stage | 1002534 | | Narro | | | | | |
| I | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Lymphoplasmacytoid lymphoma/immunocytoma stage | 1002534 | | Narro | | | | | |
| II | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Lymphoplasmacytoid lymphoma/immunocytoma stage | 1002534 | | Narro | | | | | |
| III | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Lymphoplasmacytoid lymphoma/immunocytoma stage | 1002535 | | Narro | | | | | |
| IV | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002558 | | Narro | | | | | |
| Malignant histiocytosis | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006124 | | Narro | | | | | |
| Malignant lymphoid neoplasm | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002563 | | Narro | | | | | |
| Malignant lymphoma unclassifiable high grade | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002563 | | Narro | | | | | |
| Malignant lymphoma unclassifiable low grade | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002563 | | Narro | | | | | |
| Malignant mast cell neoplasm | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002653 | | Narro | | | | | |
| Malignant neoplasm of thymus | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002670 | | Narro | | | | | |
| Malignant splenic neoplasm | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006127 | | Narro | | | | | |
| Mantle cell lymphoma | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002680 | | Narro | | | | | |
| Mantle cell lymphoma recurrent | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002680 | | Narro | | | | | |
| Mantle cell lymphoma refractory | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002680 | | Narro | | | | | |
| Mantle cell lymphoma stage I | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002680 | | Narro | | | | | |
| Mantle cell lymphoma stage II | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002680 | | Narro | | | | | |
| Mantle cell lymphoma stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002680 | | Narro | | | | | |
| Mantle cell lymphoma stage IV | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007659 | | Narro | | | | | |
| Marginal zone lymphoma | 6 | PT | W | Α | 0 | Active | 18.1 | 20.0 |
| | 1007753 | | Narro | | | | | |
| Marginal zone lymphoma recurrent | 3 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1007753 | | Narro | | | | | |
| Marginal zone lymphoma refractory | 4 | PT | W | Α | 0 | Active | 19.0 | 20.0 |
| | 1007752 | | Narro | | | | | |
| Marginal zone lymphoma stage I | 9 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1007753 | | Narro | | | | | |
| Marginal zone lymphoma stage II | 0 | PT | W | Α | 0 | Active | 19.0 | 20.0 |
| , | 1007753 | | Narro | | | | | |
| Marginal zone lymphoma stage III | 1 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| 3 1 | 1007753 | | Narro | | | | | |
| Marginal zone lymphoma stage IV | 2 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1005645 | | Narro | | | | | |
| Mastocytic leukaemia | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002694 | | Narro | | | | | |
| Mature B-cell type acute leukaemia | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| V 1 | 1005166 | | Narro | | 1 | | | |
| Metastases to bone marrow | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002745 | | Narro | | | | | |
| Metastases to lymph nodes | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| <b>7</b> 1 | 1005168 | | Narro | | † | | | |
| Metastases to spleen | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007154 | | Narro | | | | | |
| Metastatic lymphoma | 1 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1007998 | | Narro | | | | | |
| Minimal residual disease | 7 | PT | W | A | 0 | Active | 20.1 | 20.1 |
| | 1006129 | | Narro | | | | | |
| Monocytic leukaemia in remission | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002848 | | Narro | | | | | |
| Mycosis fungoides | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002850 | | Narro | | | | | |
| Mycosis fungoides recurrent | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002850 | | Narro | | | | | |
| Mycosis fungoides refractory | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002850 | | Narro | | | | | |
| Mycosis fungoides stage I | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002850 | | Narro | | | | | |
| Mycosis fungoides stage II | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002850 | | Narro | | | | | |
| Mycosis fungoides stage III | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002850 | | Narro | | | | | |
| Mycosis fungoides stage IV | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005114 | | Narro | | | | | |
| Myeloblastoma | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006130 | | Narro | | | | | |
| Myeloid leukaemia in remission | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002881 | | Narro | | | | | |
| Natural killer-cell leukaemia | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005897 | | Narro | | | | | |
| Natural killer-cell lymphoblastic lymphoma | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002895 | | Narro | | | | | |
| Neonatal leukaemia | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002946 | | Narro | | | | | |
| Nodal marginal zone B-cell lymphoma | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002946 | | Narro | | | | | |
| Nodal marginal zone B-cell lymphoma recurrent | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002946 | | Narro | | | | | |
| Nodal marginal zone B-cell lymphoma refractory | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002946 | | Narro | | | | | |
| Nodal marginal zone B-cell lymphoma stage I | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002946 | | Narro | | | | | |
| Nodal marginal zone B-cell lymphoma stage II | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002946 | | Narro | | | | | |
| Nodal marginal zone B-cell lymphoma stage III | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002946 | | Narro | | | | | |
| Nodal marginal zone B-cell lymphoma stage IV | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1008020 | | Narro | | | | | |
| Nodular lymphocyte predominant Hodgkin lymphoma | 1 | PT | W | A | 0 | Active | 20.1 | 20.1 |
| | 1002954 | | Narro | | | | | |
| Non-Hodgkin's lymphoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007153 | | Narro | | | | | |
| Non-Hodgkin's lymphoma metastatic | 5 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1002960 | | Narro | | | | | |
| Non-Hodgkin's lymphoma recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002960 | | Narro | | | | | |
| Non-Hodgkin's lymphoma refractory | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002960 | | Narro | | | | | |
| Non-Hodgkin's lymphoma stage I | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002960 | | Narro | | | | | |
| Non-Hodgkin's lymphoma stage II | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002960 | | Narro | | | | | |
| Non-Hodgkin's lymphoma stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002960 | | Narro | | | | | |
| Non-Hodgkin's lymphoma stage IV | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006187 | | Narro | | | | | |
| Non-Hodgkin's lymphoma transformed recurrent | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1006390 | | Narro | | | | | |
| aggressive | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1002960 | | Narro | | | | | |
| aggressive recurrent | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| Non-Hodgkin's lymphoma unspecified histology | 1002961 | | Narro | | | | | |
| aggressive refractory | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1002961 | | Narro | | | | | |
| aggressive stage I | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1002961 | | Narro | | | | | |
| aggressive stage II | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1002961 | | Narro | | | | | |
| aggressive stage III | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1002961 | | Narro | | | | | |
| aggressive stage IV | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1006585 | | Narro | | | | | |
| indolent | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1002962 | | Narro | | | | | |
| indolent stage I | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1002962 | | Narro | | | | | |
| indolent stage II | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1002962 | | Narro | | | | | |
| indolent stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Non-Hodgkin's lymphoma unspecified histology | 1002962 | | Narro | | | | | |
| indolent stage IV | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007532 | | Narro | | | | | |
| Ocular lymphoma | 4 | PT | W | A | 0 | Active | 17.1 | 20.0 |
| | 1003462 | | Narro | | | | | |
| Peripheral T-cell lymphoma unspecified | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003462 | | Narro | | | | | |
| Peripheral T-cell lymphoma unspecified recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003462 | | Narro | | | | | |
| Peripheral T-cell lymphoma unspecified refractory | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003462 | | Narro | | | | | |
| Peripheral T-cell lymphoma unspecified stage I | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003462 | 1 | Narro | | | | | |
| Peripheral T-cell lymphoma unspecified stage II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003462 | | Narro | | | | | |
| Peripheral T-cell lymphoma unspecified stage III | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| Name | | | Scope | Categor | Weigh | | Addition<br>Version | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | Code | Level | | y | t | Status | | Version |
| | 1003463 | | Narro | | | | | |
| Peripheral T-cell lymphoma unspecified stage IV | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003522 | | Narro | | | | | |
| Plasma cell leukaemia | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006040 | | Narro | | | | | |
| Plasma cell leukaemia in remission | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003522 | | Narro | | | | | |
| Plasma cell myeloma | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007313 | | Narro | | | | | |
| Plasma cell myeloma in remission | 2 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1007313 | | Narro | | | | | |
| Plasma cell myeloma recurrent | 3 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1006503 | | Narro | | | | | |
| Plasmablastic lymphoma | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003548 | | Narro | | | | | |
| Plasmacytoma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003652 | | Narro | | | | | |
| Precursor B-lymphoblastic lymphoma | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006091 | | Narro | | | | | |
| Precursor B-lymphoblastic lymphoma recurrent | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006091 | | Narro | | | | | |
| Precursor B-lymphoblastic lymphoma refractory | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003653 | | Narro | | | | | |
| Precursor B-lymphoblastic lymphoma stage I | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003653 | | Narro | | | | | |
| Precursor B-lymphoblastic lymphoma stage II | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003653 | | Narro | | | | | |
| Precursor B-lymphoblastic lymphoma stage III | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003653 | | Narro | | | | | |
| Precursor B-lymphoblastic lymphoma stage IV | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| - | 1003654 | | Narro | | | | | |
| Precursor T-lymphoblastic lymphoma/leukaemia | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Precursor T-lymphoblastic lymphoma/leukaemia | 1003654 | | Narro | | | | | |
| recurrent | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |


| Name | Code | Level | Scope | Categor<br>y | Weigh<br>t | Status | Addition<br>Version | Last Modified<br>Version |
|---|---|---|---|---|---|---|---|---|
| refractory | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003654 | | Narro | | | | | |
| Precursor T-lymphoblastic lymphoma/leukaemia stage I | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Precursor T-lymphoblastic lymphoma/leukaemia stage | 1003654 | | Narro | | | | | |
| II | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Precursor T-lymphoblastic lymphoma/leukaemia stage | 1003655 | | Narro | | | | | |
| III | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Precursor T-lymphoblastic lymphoma/leukaemia stage | 1003655 | | Narro | | | | | |
| IV 3 1 3 1 | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007599 | | Narro | | | | | |
| Primary cardiac lymphoma | 3 | PT | w | A | 0 | Active | 18.0 | 20.0 |
| | 1006585 | | Narro | | | | | |
| Primary effusion lymphoma | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007897 | | Narro | | | | | |
| Primary gastrointestinal follicular lymphoma | 2 | PT | W | A | 0 | Active | 20.0 | 20.0 |
| | 1003671 | | Narro | | | | | |
| Primary mediastinal large B-cell lymphoma | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003671 | | Narro | | | | | |
| Primary mediastinal large B-cell lymphoma recurrent | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003671 | | Narro | | | | | |
| Primary mediastinal large B-cell lymphoma refractory | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003671 | | Narro | | | | | |
| Primary mediastinal large B-cell lymphoma stage I | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003671 | | Narro | | | | | |
| Primary mediastinal large B-cell lymphoma stage II | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003671 | | Narro | | | | | |
| Primary mediastinal large B-cell lymphoma stage III | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003671 | | Narro | | | | | |
| Primary mediastinal large B-cell lymphoma stage IV | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003688 | | Narro | | | | | |
| Prolymphocytic leukaemia | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005872 | | Narro | | | | | |
| Richter's syndrome | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006211 | | Narro | | | | | |
| Splenic marginal zone lymphoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004165 | | Narro | | | | | |
| Splenic marginal zone lymphoma recurrent | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004165 | | Narro | | | | | |
| Splenic marginal zone lymphoma refractory | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004165 | | Narro | | | | | |
| Splenic marginal zone lymphoma stage I | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004165 | | Narro | | | | | |
| Splenic marginal zone lymphoma stage II | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004165 | | Narro | | | | | |
| Splenic marginal zone lymphoma stage III | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004165 | | Narro | | | | | |
| Splenic marginal zone lymphoma stage IV | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004297 | | Narro | | | | | |
| T-cell chronic lymphocytic leukaemia | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| , i | 1004297 | | Narro | | | | | |
| T-cell lymphoma | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004297 | | Narro | | | | | |
| T-cell lymphoma recurrent | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004298 | | Narro | | | | | |
| T-cell lymphoma refractory | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004298 | | Narro | | | | | |
| T-cell lymphoma stage I | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004298 | | Narro | | | | | |
| T-cell lymphoma stage II | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004298 | | Narro | | | | | |
| T-cell lymphoma stage III | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004298 | | Narro | | | | | |
| T-cell lymphoma stage IV | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004298 | | Narro | | | | | |
| T-cell prolymphocytic leukaemia | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004298 | | Narro | | | | | |
| T-cell type acute leukaemia | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1004298 | | Narro | | | | | |
| T-cell unclassifiable lymphoma high grade | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004299 | | Narro | | | | | |
| T-cell unclassifiable lymphoma low grade | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005510 | | Narro | | | | | |
| Thymic cancer metastatic | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006103 | | Narro | | | | | |
| Thymoma malignant | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004367 | | Narro | | | | | |
| Thymoma malignant recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007261 | | Narro | | | | | |
| Thyroid B-cell lymphoma | 3 | PT | W | A | 0 | Active | 15.1 | 20.0 |
| | 1007910 | | Narro | | | | | |
| Transformation to acute myeloid leukaemia | 7 | PT | W | A | 0 | Active | 20.0 | 20.0 |
| | 1008020 | | Narro | | | | | |
| Triple hit lymphoma | 0 | PT | W | A | 0 | Active | 20.1 | 20.1 |
| | 1004780 | | Narro | | | | | |
| Waldenstrom's macroglobulinaemia | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004780 | | Narro | | | | | |
| Waldenstrom's macroglobulinaemia recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004780 | | Narro | | | | | |
| Waldenstrom's macroglobulinaemia refractory | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004780 | | Narro | | | | | |
| Valdenstrom's macroglobulinaemia stage I | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004780 | | Narro | | | | | |
| Waldenstrom's macroglobulinaemia stage II | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| Name | Code | Level | Scope | Categor | Weigh<br>t | Status | Addition<br>Version | Last Modified<br>Version |
|---|---|---|---|---|---|---|---|---|
| | 1004780 | | Narro | | | | | |
| Waldenstrom's macroglobulinaemia stage III | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004780 | | Narro | | | | | |
| Waldenstrom's macroglobulinaemia stage IV | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| haematological malignant tumours (SMQ) [20000 | 228] | | | | | | | |
| Name | Code | Level | Scope | Categor | Weigh<br>t | Status | Addition<br>Version | Last Modified<br>Version |
| | 1007102 | | Narro | J | | | , 6151011 | 7 61 51 611 |
| Abdominal wall neoplasm malignant | 3 | PT | W | A | 0 | Active | 14.0 | 20.0 |
| 1 5 | 1007336 | | Narro | | | | | |
| Acinar cell carcinoma of pancreas | 3 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1007336 | | Narro | | | | | |
| Acinic cell carcinoma of salivary gland | 9 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1000058 | | Narro | | | | | |
| Acral lentiginous melanoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000058 | | Narro | | | | | |
| Acral lentiginous melanoma stage I | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000058 | | Narro | | | | | |
| Acral lentiginous melanoma stage II | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000058 | | Narro | | | | | |
| Acral lentiginous melanoma stage III | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| A continued disconnection of the IV | 1000058 | DT | Narro | | | A -4: | 10.0 | 20.0 |
| Acral lentiginous melanoma stage IV | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Adenocarcinoma | 1000114 | PT | Narro<br>w | A | 0 | Active | 10.0 | 20.0 |
| Adenocaremonia | 1000115 | 1 1 | Narro | A | 0 | Active | 10.0 | 20.0 |
| Adenocarcinoma gastric | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Additional gustife | 1007335 | 1.1 | Narro | 11 | 0 | Tictive | 10.0 | 20.0 |
| Adenocarcinoma of appendix | 9 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1000116 | | Narro | | <u> </u> | - 1001.0 | - 3.0 | |
| Adenocarcinoma of colon | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006806 | | Narro | | 1 | | | |
| Adenocarcinoma of salivary gland | 8 | PT | W | A | 0 | Active | 11.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1000119 | | Narro | | | | | |
| Adenocarcinoma of the cervix | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005274 | | Narro | | | | | |
| Adenocarcinoma pancreas | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005323 | | Narro | | | | | |
| Adenoid cystic carcinoma | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007805 | | Narro | | | | | |
| Adenoid cystic carcinoma of external auditory canal | 7 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1007337 | | Narro | | | | | |
| Adenoid cystic carcinoma of salivary gland | 0 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1000124 | | Narro | | | | | |
| Adenosquamous carcinoma of the cervix | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007397 | | Narro | | | | | |
| Adenosquamous carcinoma of vagina | 8 | PT | W | A | 0 | Active | 16.1 | 20.0 |
| | 1006887 | | Narro | | | | | |
| Adenosquamous cell carcinoma | 3 | PT | W | A | 0 | Active | 12.0 | 20.0 |
| • | 1000124 | | Narro | | | | | |
| Adenosquamous cell lung cancer | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000124 | | Narro | | | | | |
| Adenosquamous cell lung cancer recurrent | 7 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1000124 | | Narro | | | | | |
| Adenosquamous cell lung cancer stage 0 | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000124 | | Narro | | | | | |
| Adenosquamous cell lung cancer stage I | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000125 | | Narro | | | | | |
| Adenosquamous cell lung cancer stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000125 | | Narro | | | | | |
| Adenosquamous cell lung cancer stage III | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000125 | | Narro | | | | | |
| Adenosquamous cell lung cancer stage IV | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007315 | | Narro | | | | | |
| Adrenal gland cancer | 2 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1005509 | | Narro | | | | | |
| Adrenal gland cancer metastatic | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1000138 | | Narro | | | | | |
| Adrenocortical carcinoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000143 | | Narro | | | | | |
| Aesthesioneuroblastoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006586 | | Narro | | | | | |
| Alveolar rhabdomyosarcoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000188 | | Narro | | | | | |
| Alveolar soft part sarcoma | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000188 | | Narro | | | | | |
| Alveolar soft part sarcoma metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000188 | | Narro | | | | | |
| Alveolar soft part sarcoma recurrent | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006142 | | Narro | | | | | |
| Anal cancer | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005509 | | Narro | | | | | |
| Anal cancer metastatic | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000213 | | Narro | | | | | |
| Anal cancer recurrent | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000213 | | Narro | | | | | |
| Anal cancer stage 0 | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000213 | | Narro | | | | | |
| Anal cancer stage I | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000213 | | Narro | | | | | |
| Anal cancer stage II | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000213 | | Narro | | | | | |
| Anal cancer stage III | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000213 | | Narro | | | | | |
| Anal cancer stage IV | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007335 | | Narro | | | | | |
| Anal squamous cell carcinoma | 8 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1000222 | | Narro | | | | | |
| Anaplastic astrocytoma | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007312 | | Narro | | | | | |
| Anaplastic meningioma | 7 | PT | W | A | 0 | Active | 16.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007312 | | Narro | | | | | |
| Anaplastic oligodendroglioma | 8 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1000224 | | Narro | | | | | |
| Anaplastic thyroid cancer | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007312 | | Narro | | | | | |
| Angiocentric glioma | 9 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1000247 | | Narro | | | | | |
| Angiosarcoma | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000247 | | Narro | | | | | |
| Angiosarcoma metastatic | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005770 | | Narro | | | | | |
| Angiosarcoma non-metastatic | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000248 | | Narro | | | | | |
| Angiosarcoma recurrent | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006620 | | Narro | | | | | |
| Apocrine breast carcinoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007336 | | Narro | | | | | |
| Appendix cancer | 0 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1000357 | | Narro | | | | | |
| Astrocytoma | 1 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1006097 | | Narro | | | | | |
| Astrocytoma malignant | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006590 | | Narro | | | | | |
| Atypical teratoid/rhabdoid tumour of CNS | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000414 | | Narro | | | | | |
| Basal cell carcinoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000417 | | Narro | | | | | |
| Basosquamous carcinoma | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000417 | | Narro | | | | | |
| Basosquamous carcinoma of skin | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000458 | | Narro | | | | | |
| Bile duct adenocarcinoma | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000458 | | Narro | | | | | |
| Bile duct adenosquamous carcinoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1000459 | | Narro | | | | | |
| Bile duct cancer | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000459 | | Narro | | | | | |
| Bile duct cancer recurrent | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005938 | | Narro | | | | | |
| Bile duct cancer stage 0 | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005937 | | Narro | | | | | |
| Bile duct cancer stage I | 3 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1005937 | | Narro | | | | | |
| Bile duct cancer stage II | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005937 | | Narro | | | | | |
| Bile duct cancer stage III | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005937 | | Narro | | | | | |
| Bile duct cancer stage IV | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000463 | | Narro | | | | | |
| Bile duct squamous cell carcinoma | 3 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| • | 1005511 | | Narro | | | | | |
| Biliary cancer metastatic | 1 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1007306 | | Narro | | | | | |
| Biphasic mesothelioma | 2 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1000498 | | Narro | | | | | |
| Bladder adenocarcinoma recurrent | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000498 | | Narro | | | | | |
| Bladder adenocarcinoma stage 0 | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000498 | | Narro | | | | | |
| Bladder adenocarcinoma stage I | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000498 | | Narro | | | | | |
| Bladder adenocarcinoma stage II | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000499 | | Narro | | | | | |
| Bladder adenocarcinoma stage III | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000499 | | Narro | | | | | |
| Bladder adenocarcinoma stage IV | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000499 | 1 | Narro | 1 | | | | |
| Bladder adenocarcinoma stage unspecified | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1000500 | | Narro | | | | | |
| Bladder cancer | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000500 | | Narro | | | | | |
| Bladder cancer recurrent | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000500 | | Narro | | | | | |
| Bladder cancer stage 0, with cancer in situ | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000500 | | Narro | | | | | |
| Bladder cancer stage 0, without cancer in situ | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000500 | | Narro | | | | | |
| Bladder cancer stage I, with cancer in situ | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000500 | | Narro | | | | | |
| Bladder cancer stage I, without cancer in situ | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000501 | | Narro | | | | | |
| Bladder cancer stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000501 | | Narro | | | | | |
| Bladder cancer stage III | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000501 | | Narro | | | | | |
| Bladder cancer stage IV | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000507 | | Narro | | | | | |
| Bladder squamous cell carcinoma recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000507 | | Narro | | | | | |
| Bladder squamous cell carcinoma stage 0 | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000507 | | Narro | | | | | |
| Bladder squamous cell carcinoma stage I | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000507 | | Narro | | | | | |
| Bladder squamous cell carcinoma stage II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000507 | | Narro | | | | | |
| Bladder squamous cell carcinoma stage III | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000508 | | Narro | | | | | |
| Bladder squamous cell carcinoma stage IV | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000508 | | Narro | | | | | |
| Bladder squamous cell carcinoma stage unspecified | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000508 | | Narro | | | | | |
| Bladder transitional cell carcinoma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007166 | | Narro | | | | | |
| Bladder transitional cell carcinoma metastatic | 4 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1006675 | | Narro | | | | | |
| Bladder transitional cell carcinoma recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006674 | | Narro | | | | | |
| Bladder transitional cell carcinoma stage 0 | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006675 | | Narro | | | | | |
| Bladder transitional cell carcinoma stage I | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006675 | | Narro | | | | | |
| Bladder transitional cell carcinoma stage II | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006675 | | Narro | | | | | |
| Bladder transitional cell carcinoma stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006675 | | Narro | | | | | |
| Bladder transitional cell carcinoma stage IV | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000594 | | Narro | | | | | |
| Bone cancer | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005510 | | Narro | | | | | |
| Bone cancer metastatic | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007310 | | Narro | | | | | |
| Bone giant cell tumour malignant | 6 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1000600 | | Narro | | | | | |
| Bone sarcoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000605 | | Narro | | | | | |
| Bowen's disease | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005509 | | Narro | | | | | |
| Brain cancer metastatic | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000613 | | Narro | | | | | |
| Brain neoplasm malignant | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007385 | | Narro | | | | | |
| Brain sarcoma | 7 | PT | W | A | 0 | Active | 16.1 | 20.0 |
| | 1000614 | | Narro | | | | | |
| Brain stem glioma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007281 | | Narro | | | | | |
| Breast angiosarcoma | 3 | PT | W | A | 0 | Active | 15.1 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007281 | | Narro | | | | | |
| Breast angiosarcoma metastatic | 4 | PT | w | A | 0 | Active | 15.1 | 20.0 |
| | 1000618 | | Narro | | | | | |
| Breast cancer | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005765 | | Narro | | | | | |
| Breast cancer female | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000618 | | Narro | | | | | |
| Breast cancer in situ | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006102 | | Narro | | | | | |
| Breast cancer male | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005511 | | Narro | | | | | |
| Breast cancer metastatic | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000619 | | Narro | | | | | |
| Breast cancer recurrent | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000619 | | Narro | | | | | |
| Breast cancer stage I | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000620 | | Narro | | | | | |
| Breast cancer stage II | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000620 | | Narro | | | | | |
| Breast cancer stage III | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000620 | | Narro | | | | | |
| Breast cancer stage IV | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| <u> </u> | 1006858 | | Narro | | | | | |
| Breast sarcoma | 2 | PT | W | Α | 0 | Active | 11.1 | 20.0 |
| | 1006858 | | Narro | | | | | |
| Breast sarcoma metastatic | 3 | PT | w | A | 0 | Active | 11.1 | 20.0 |
| | 1006858 | | Narro | | | | | |
| Breast sarcoma recurrent | 4 | PT | W | A | 0 | Active | 11.1 | 20.0 |
| | 1000641 | | Narro | | | | | |
| Bronchial carcinoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005835 | | Narro | | | | | |
| Bronchioloalveolar carcinoma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005942 | | Narro | | | | | |
| Buschke-Lowenstein's tumour | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006530 | | Narro | | | | | |
| Cancer in remission | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000727 | | Narro | | | | | |
| Carcinoid tumour | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000727 | | Narro | | | | | |
| Carcinoid tumour of the appendix | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000727 | | Narro | | | | | |
| Carcinoid tumour of the caecum | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005011 | | Narro | | | | | |
| Carcinoid tumour of the duodenum | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000727 | | Narro | | | | | |
| Carcinoid tumour of the gastrointestinal tract | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005500 | | Narro | | | | | |
| Carcinoid tumour of the pancreas | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000728 | | Narro | | | | | |
| Carcinoid tumour of the prostate | 0 | PT | w | Α | 0 | Active | 10.0 | 20.0 |
| 1 | 1005281 | | Narro | | | | | |
| Carcinoid tumour of the small bowel | 9 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1000728 | | Narro | | | | | |
| Carcinoid tumour of the stomach | 1 | PT | w | Α | 0 | Active | 10.0 | 20.0 |
| | 1000728 | | Narro | | | | | |
| Carcinoid tumour pulmonary | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| · | 1007743 | | Narro | | | | | |
| Carcinoma ex-pleomorphic adenoma | 5 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1006145 | | Narro | | | | | |
| Carcinoma in situ | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000736 | | Narro | | | | | |
| Carcinoma in situ of eye | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1000738 | | Narro | | | | | |
| Carcinoma in situ of penis | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| ^ | 1000739 | | Narro | | | | | |
| Carcinoma in situ of skin | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000740 | | Narro | | | | | |
| Carcinoma in situ of trachea | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006102 | | Narro | | | | | |
| Cardiac neoplasm malignant | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007716 | | Narro | | | | | |
| Central nervous system melanoma | 0 | PT | W | A | 0 | Active | 18.1 | 20.0 |
| | 1007313 | | Narro | | | | | |
| Central nervous system neuroblastoma | 0 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005509 | | Narro | | | | | |
| Cervix cancer metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000834 | | Narro | | | | | |
| Cervix carcinoma | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000834 | | Narro | | | | | |
| Cervix carcinoma recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006180 | | Narro | | | | | |
| Cervix carcinoma stage 0 | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000834 | | Narro | | | | | |
| Cervix carcinoma stage I | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000834 | | Narro | | | | | |
| Cervix carcinoma stage II | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000834 | | Narro | | | | | |
| Cervix carcinoma stage III | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000834 | | Narro | | | | | |
| Cervix carcinoma stage IV | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000859 | | Narro | | | | | |
| Cholangiocarcinoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007786 | | Narro | | | | | |
| Cholangiosarcoma | 1 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1000873 | | Narro | | | | | |
| Chondrosarcoma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000873 | | Narro | | | | | |
| Chondrosarcoma metastatic | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000873 | | Narro | | | | | |
| Chondrosarcoma recurrent | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000874 | | Narro | | | | | |
| Chordoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1000875 | | Narro | | | | | |
| Choriocarcinoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000877 | | Narro | | | | | |
| Choroid melanoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006747 | | Narro | | | | | |
| Choroid plexus carcinoma | 8 | PT | W | A | 0 | Active | 10.1 | 20.0 |
| | 1007490 | | Narro | | | | | |
| Clear cell carcinoma of cervix | 9 | PT | W | A | 0 | Active | 17.1 | 20.0 |
| | 1000925 | | Narro | | | | | |
| Clear cell endometrial carcinoma | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007325 | | Narro | | | | | |
| Clear cell renal cell carcinoma | 1 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007314 | | Narro | | | | | |
| Clear cell sarcoma of soft tissue | 0 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1000925 | | Narro | | | | | |
| Clear cell sarcoma of the kidney | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| <u> </u> | 1006585 | | Narro | | | | | |
| CNS germinoma | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000994 | | Narro | | | | | |
| Colon cancer | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005511 | | Narro | | | | | |
| Colon cancer metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000995 | | Narro | | | | | |
| Colon cancer recurrent | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006352 | | Narro | | | | | |
| Colon cancer stage 0 | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1000995 | | Narro | | | | | |
| Colon cancer stage I | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000995 | | Narro | | | | | |
| Colon cancer stage II | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000995 | | Narro | | | | | |
| Colon cancer stage III | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1000995 | | Narro | | | | | |
| Colon cancer stage IV | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1005236 | | Narro | | | | | |
| Colorectal adenocarcinoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006145 | | Narro | | | | | |
| Colorectal cancer | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005235 | | Narro | | | | | |
| Colorectal cancer metastatic | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001003 | | Narro | | | | | |
| Colorectal cancer recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001003 | | Narro | | | | | |
| Colorectal cancer stage I | 2 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1001003 | | Narro | | | | | |
| Colorectal cancer stage II | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001003 | | Narro | | | | | |
| Colorectal cancer stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001003 | | Narro | | | | | |
| Colorectal cancer stage IV | 5 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1001003 | | Narro | | | | | |
| Colorectal carcinoma stage 0 | 8 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1006585 | | Narro | | | | | |
| Congenital fibrosarcoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007349 | | Narro | | | | | |
| Congenital malignant neoplasm | 2 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007347 | | Narro | | | | | |
| Congenital retinoblastoma | 0 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1006638 | | Narro | | | | | |
| Conjunctival melanoma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005491 | | Narro | | | | | |
| Cystadenocarcinoma ovary | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| • | 1007313 | | Narro | | | | | |
| Dedifferentiated liposarcoma | 5 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| • | 1005707 | | Narro | | | | | |
| Dermatofibrosarcoma protuberans | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| • | 1007357 | | Narro | 1 | 1 | | | |
| Dermatofibrosarcoma protuberans metastatic | 4 | PT | W | A | 0 | Active | 16.1 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007244 | | Narro | | | | | |
| Desmoplastic melanoma | 9 | PT | w | A | 0 | Active | 15.1 | 20.0 |
| | 1007306 | | Narro | | | | | |
| Desmoplastic mesothelioma | 3 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1006458 | | Narro | | | | | |
| Desmoplastic small round cell tumour | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007336 | | Narro | | | | | |
| Ductal adenocarcinoma of pancreas | 4 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005501 | | Narro | | | | | |
| Ear neoplasm malignant | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006968 | | Narro | | | | | |
| Eccrine carcinoma | 0 | PT | w | A | 0 | Active | 12.1 | 20.0 |
| | 1006586 | | Narro | | | | | |
| Embryonal rhabdomyosarcoma | 8 | PT | w | Α | 0 | Active | 10.0 | 20.0 |
| • | 1006112 | | Narro | | | | | |
| Endocrine neoplasm malignant | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001472 | | Narro | | | | | |
| Endometrial adenocarcinoma | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001473 | | Narro | | | | | |
| Endometrial cancer | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001473 | | Narro | | | | | |
| Endometrial cancer metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001473 | | Narro | | | | | |
| Endometrial cancer recurrent | 6 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1001473 | | Narro | | | | | |
| Endometrial cancer stage 0 | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001473 | | Narro | | | | | |
| Endometrial cancer stage I | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001473 | | Narro | | | | | |
| Endometrial cancer stage II | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001474 | | Narro | | 1 | | | |
| Endometrial cancer stage III | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001474 | | Narro | | 1 | | | |
| Endometrial cancer stage IV | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1005764 | | Narro | | | | | |
| Endometrial sarcoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006706 | | Narro | | | | | |
| Endometrial sarcoma metastatic | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006706 | | Narro | | | | | |
| Endometrial sarcoma recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004839 | | Narro | | | | | |
| Endometrial stromal sarcoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007686 | | Narro | | | | | |
| Endotheliomatosis | 8 | PT | W | A | 0 | Active | 18.1 | 20.0 |
| | 1001496 | | Narro | | | | | |
| Ependymoma malignant | 8 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1007311 | | Narro | | | | | |
| Epididymal cancer | 5 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005743 | | Narro | | | | | |
| Epiglottic carcinoma | 8 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1007306 | | Narro | | | | | |
| Epithelioid mesothelioma | 4 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1001509 | | Narro | | | | | |
| Epithelioid sarcoma | 9 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1001510 | | Narro | | | | | |
| Epithelioid sarcoma metastatic | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1001510 | | Narro | | | | | |
| Epithelioid sarcoma recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001556 | | Narro | | | | | |
| Ewing's sarcoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1001556 | | Narro | | | | | |
| Ewing's sarcoma metastatic | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1001556 | | Narro | | | | | |
| Ewing's sarcoma recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1001578 | | Narro | | | | | |
| Extragonadal primary embryonal carcinoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007305 | | Narro | | | | | |
| Extragonadal primary germ cell tumour | 5 | PT | W | A | 0 | Active | 16.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007305 | | Narro | | | | | |
| Extragonadal primary germ cell tumour mixed | 6 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1001580 | | Narro | | | | | |
| Extragonadal primary germ cell tumour mixed stage I | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001580 | | Narro | | | | | |
| Extragonadal primary germ cell tumour mixed stage II | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001580 | | Narro | | | | | |
| Extragonadal primary germ cell tumour mixed stage III | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006184 | | Narro | | | | | |
| Extragonadal primary malignant teratoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006184 | | Narro | | | | | |
| Extragonadal primary non-seminoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001580 | | Narro | | | | | |
| Extragonadal primary non-seminoma stage I | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001580 | | Narro | | | | | |
| Extragonadal primary non-seminoma stage II | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001580 | | Narro | | | | | |
| Extragonadal primary non-seminoma stage III | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001581 | | Narro | | | | | |
| Extragonadal primary non-seminoma stage IV | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007305 | | Narro | | | | | |
| Extragonadal primary seminoma (pure) | 7 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1001581 | | Narro | | | | | |
| Extragonadal primary seminoma (pure) stage I | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001581 | | Narro | | | | | |
| Extragonadal primary seminoma (pure) stage II | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001581 | | Narro | | | | | |
| Extragonadal primary seminoma (pure) stage III | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001581 | | Narro | | | | | |
| Extragonadal primary seminoma (pure) stage IV | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006822 | | Narro | | | | | |
| Extramammary Paget's disease | 3 | PT | W | A | 0 | Active | 11.0 | 20.0 |
| | 1001583 | | Narro | | | | | |
| Extraocular retinoblastoma | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1001575 | | Narro | | | | | |
| Extra-osseous Ewing's sarcoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001576 | | Narro | | | | | |
| Extra-osseous Ewing's sarcoma metastatic | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001576 | | Narro | | | | | |
| Extra-osseous Ewing's sarcoma recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001584 | | Narro | | | | | |
| Extraskeletal chondrosarcoma metastatic | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001584 | | Narro | | | | | |
| Extraskeletal chondrosarcoma recurrent | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007313 | | Narro | | | | | |
| Extraskeletal myxoid chondrosarcoma | 4 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1001584 | | Narro | | | | | |
| Extraskeletal osteosarcoma | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001584 | | Narro | | | | | |
| Extraskeletal osteosarcoma metastatic | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001585 | | Narro | | | | | |
| Extraskeletal osteosarcoma recurrent | 2 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1001618 | | Narro | | | | | |
| Fallopian tube cancer | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001618 | | Narro | | | | | |
| Fallopian tube cancer metastatic | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1001618 | | Narro | | | | | |
| Fallopian tube cancer stage I | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1001618 | | Narro | | | | | |
| Fallopian tube cancer stage II | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| <del>-</del> | 1001618 | | Narro | | | | | |
| Fallopian tube cancer stage III | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1001618 | | Narro | | | | | |
| Fallopian tube cancer stage IV | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007315 | | Narro | | | | | |
| Familial medullary thyroid cancer | 3 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1006115 | | Narro | | | | | |
| Female reproductive tract carcinoma in situ | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1001663 | | Narro | | | | | |
| Fibrosarcoma | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001663 | | Narro | | | | | |
| Fibrosarcoma metastatic | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001693 | | Narro | | | | | |
| Follicular thyroid cancer | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005828 | | Narro | | | | | |
| Gallbladder adenocarcinoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007306 | | Narro | | | | | |
| Gallbladder adenosquamous carcinoma | 7 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1001761 | | Narro | | | | | |
| Gallbladder cancer | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006687 | | Narro | | | | | |
| Gallbladder cancer metastatic | 9 | PT | w | Α | 0 | Active | 10.0 | 20.0 |
| | 1001761 | | Narro | | | | | |
| Gallbladder cancer recurrent | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005931 | | Narro | | | | | |
| Gallbladder cancer stage 0 | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005931 | | Narro | | | | | |
| Gallbladder cancer stage I | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005828 | | Narro | | | | | |
| Gallbladder cancer stage II | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| <u> </u> | 1005828 | | Narro | | | | | |
| Gallbladder cancer stage III | 2 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1005828 | | Narro | | | | | |
| Gallbladder cancer stage IV | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| <u> </u> | 1007306 | | Narro | | | | | |
| Gallbladder squamous cell carcinoma | 8 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| • | 1001770 | | Narro | | | | | |
| Ganglioglioma | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001770 | | Narro | | | | | |
| Ganglioneuroblastoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001775 | | Narro | | | | | |
| Gastric cancer | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1001776 | | Narro | | | | | |
| Gastric cancer recurrent | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001776 | | Narro | | | | | |
| Gastric cancer stage 0 | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001776 | | Narro | | | | | |
| Gastric cancer stage I | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001776 | | Narro | | | | | |
| Gastric cancer stage II | 4 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1001776 | | Narro | | | | | |
| Gastric cancer stage III | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006196 | | Narro | | | | | |
| Gastric cancer stage IV | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005500 | | Narro | | | | | |
| Gastric sarcoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005170 | | Narro | | | | | |
| Gastrinoma malignant | 9 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1007755 | | Narro | | | | | |
| Gastroenteropancreatic neuroendocrine tumour disease | 9 | PT | W | Α | 0 | Active | 19.0 | 20.0 |
| - | 1005354 | | Narro | | | | | |
| Gastrointestinal cancer metastatic | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001794 | | Narro | | | | | |
| Gastrointestinal carcinoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006116 | | Narro | | | | | |
| Gastrointestinal carcinoma in situ | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007716 | | Narro | | | | | |
| Gastrointestinal melanoma | 7 | PT | W | A | 0 | Active | 18.1 | 20.0 |
| | 1007165 | | Narro | | | | | |
| Gastrointestinal stromal cancer | 3 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1006287 | | Narro | | | | | |
| Gastrooesophageal cancer | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007311 | | Narro | | | | | |
| Genital cancer male | 6 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007312 | | Narro | 1 | | | | |
| Genital cancer male in situ | 4 | PT | W | A | 0 | Active | 16.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1001816 | | Narro | | | | | |
| Genital neoplasm malignant female | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007716 | | Narro | | | | | |
| Genitourinary melanoma | 6 | PT | W | A | 0 | Active | 18.1 | 20.0 |
| | 1006118 | | Narro | | | | | |
| Germ cell cancer | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006897 | | Narro | | | | | |
| Germ cell cancer metastatic | 1 | PT | W | A | 0 | Active | 12.0 | 20.0 |
| | 1006198 | | Narro | | | | | |
| Gestational trophoblastic tumour | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006780 | | Narro | | | | | |
| Gingival cancer | 7 | PT | W | A | 0 | Active | 11.0 | 20.0 |
| | 1001833 | | Narro | | | | | |
| Glioblastoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001833 | | Narro | | | | | |
| Glioblastoma multiforme | 7 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1001833 | | Narro | | | | | |
| Glioma | 8 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1006625 | | Narro | | | | | |
| Gliomatosis cerebri | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006860 | | Narro | | | | | |
| Glioneuronal tumour | 1 | PT | W | A | 0 | Active | 11.1 | 20.0 |
| | 1001834 | | Narro | | | | | |
| Gliosarcoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001839 | | Narro | | | | | |
| Glottis carcinoma | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001840 | | Narro | | | | | |
| Glucagonoma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001882 | | Narro | | | | | |
| Haemangiopericytoma | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1001882 | | Narro | | | | | |
| Haemangiopericytoma of meninges | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006782 | | Narro | | | | | |
| Head and neck cancer | 1 | PT | W | A | 0 | Active | 11.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007154 | | Narro | | | | | |
| Head and neck cancer metastatic | 0 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1007153 | | Narro | | | | | |
| Head and neck cancer stage I | 9 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1007153 | | Narro | | | | | |
| Head and neck cancer stage II | 8 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1007153 | | Narro | | | | | |
| Head and neck cancer stage III | 7 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1007153 | | Narro | | | | | |
| Head and neck cancer stage IV | 6 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1006738 | | Narro | | | | | |
| Hepatic angiosarcoma | 8 | PT | W | A | 0 | Active | 10.1 | 20.0 |
| | 1007306 | | Narro | | | | | |
| Hepatic cancer | 9 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005511 | | Narro | | | | | |
| Hepatic cancer metastatic | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007307 | | Narro | | | | | |
| Hepatic cancer recurrent | 0 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005931 | | Narro | | | | | |
| Hepatic cancer stage I | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005931 | | Narro | | | | | |
| Hepatic cancer stage II | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005932 | | Narro | | | | | |
| Hepatic cancer stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005932 | | Narro | | | | | |
| Hepatic cancer stage IV | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007307 | | Narro | | | | | |
| Hepatobiliary cancer | 3 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007307 | | Narro | | | | | |
| Hepatobiliary cancer in situ | 4 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1006200 | | Narro | | | | | |
| Hepatoblastoma | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1001982 | | Narro | | | | | |
| Hepatoblastoma recurrent | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007307 | | Narro | | | | | |
| Hepatocellular carcinoma | 1 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1006543 | | Narro | | | | | |
| HER-2 positive breast cancer | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006689 | | Narro | | | | | |
| HER-2 positive gastric cancer | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006794 | | Narro | | | | | |
| Hereditary leiomyomatosis renal cell carcinoma | 4 | PT | W | A | 0 | Active | 11.0 | 20.0 |
| | 1006794 | | Narro | | | | | |
| Hereditary papillary renal carcinoma | 3 | PT | W | A | 0 | Active | 11.0 | 20.0 |
| | 1007308 | | Narro | | | | | |
| Hidradenocarcinoma | 8 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007693 | | Narro | | | | | |
| Hormone refractory breast cancer | 5 | PT | W | A | 0 | Active | 18.1 | 20.0 |
| | 1007111 | | Narro | | | | | |
| Hormone-dependent prostate cancer | 9 | PT | W | A | 0 | Active | 14.0 | 20.0 |
| | 1006290 | | Narro | | | | | |
| Hormone-refractory prostate cancer | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006613 | | Narro | | | | | |
| Huerthle cell carcinoma | 6 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1002104 | | Narro | | | | | |
| Hypopharyngeal cancer | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002104 | | Narro | | | | | |
| Hypopharyngeal cancer recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002104 | | Narro | | | | | |
| Hypopharyngeal cancer stage 0 | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002104 | | Narro | | | | | |
| Hypopharyngeal cancer stage I | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002104 | | Narro | | | | | |
| Hypopharyngeal cancer stage II | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002104 | | Narro | | | | | |
| Hypopharyngeal cancer stage III | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002104 | | Narro | | | | | |
| Hypopharyngeal cancer stage IV | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| Immune reconstitution inflammatory syndrome | 1007279 | | Narro | | | | | |
| associated Kaposi's sarcoma | 6 | PT | w | A | 0 | Active | 15.1 | 20.0 |
| | 1002197 | | Narro | | | | | |
| Inflammatory carcinoma of breast recurrent | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002197 | | Narro | | | | | |
| Inflammatory carcinoma of breast stage III | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002197 | | Narro | | | | | |
| Inflammatory carcinoma of breast stage IV | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002198 | | Narro | | | | | |
| Inflammatory carcinoma of the breast | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007314 | | Narro | | | | | |
| Inflammatory malignant fibrous histiocytoma | 2 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1006791 | | Narro | | | | | |
| Inflammatory myofibroblastic tumour | 7 | PT | w | A | 0 | Active | 11.0 | 20.0 |
| | 1005192 | | Narro | | | | | |
| Intestinal adenocarcinoma | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1008031 | | Narro | | | | | |
| Intestinal metastasis | 1 | PT | w | A | 0 | Active | 20.1 | 20.1 |
| | 1007375 | | Narro | | | | | |
| Intracranial germ cell tumour | 1 | PT | W | A | 0 | Active | 16.1 | 20.0 |
| | 1002277 | | Narro | | | | | |
| Intracranial meningioma malignant | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007354 | | Narro | | | | | |
| Intraductal papillary breast neoplasm | 0 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007336 | | Narro | | | | | |
| Intraductal papillary-mucinous carcinoma of pancreas | 5 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007309 | | Narro | | | | | |
| Intraductal proliferative breast lesion | 4 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1006125 | | Narro | | | | | |
| Intraocular melanoma | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007571 | | Narro | | | | | |
| Invasive breast carcinoma | 3 | PT | W | A | 0 | Active | 18.0 | 20.0 |
| | 1007309 | | Narro | | | | | |
| Invasive ductal breast carcinoma | 5 | PT | W | A | 0 | Active | 16.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007309 | | Narro | | | | | |
| Invasive lobular breast carcinoma | 6 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1007309 | | Narro | | | | | |
| Invasive papillary breast carcinoma | 8 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1007308 | | Narro | | | | | |
| Iris melanoma | 6 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1002328 | | Narro | | | | | |
| Kaposi's sarcoma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002328 | | Narro | | | | | |
| Kaposi's sarcoma AIDS related | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002328 | | Narro | | | | | |
| Kaposi's sarcoma classical type | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007332 | | Narro | | | | | |
| Keratinising squamous cell carcinoma of nasopharynx | 4 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1002334 | | Narro | | | | | |
| Keratoacanthoma | 7 | PT | W | A | 0 | Active | 13.1 | 20.0 |
| | 1007878 | | Narro | | | | | |
| Langerhans cell sarcoma | 2 | PT | w | A | 0 | Active | 20.0 | 20.0 |
| | 1002377 | | Narro | | | | | |
| Large cell lung cancer | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006973 | | Narro | | | | | |
| Large cell lung cancer metastatic | 0 | PT | w | A | 0 | Active | 13.0 | 20.0 |
| | 1002377 | | Narro | | | | | |
| Large cell lung cancer recurrent | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002377 | | Narro | | | | | |
| Large cell lung cancer stage 0 | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002377 | | Narro | | | | | |
| Large cell lung cancer stage I | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002377 | | Narro | | | | | |
| Large cell lung cancer stage II | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002377 | | Narro | | | | | |
| Large cell lung cancer stage III | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002378 | | Narro | | | | | |
| Large cell lung cancer stage IV | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002382 | | Narro | | | | | |
| Laryngeal cancer | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007090 | | Narro | | | | | |
| Laryngeal cancer metastatic | 2 | PT | w | A | 0 | Active | 14.0 | 20.0 |
| | 1002382 | | Narro | | | | | |
| Laryngeal cancer recurrent | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002382 | | Narro | | | | | |
| Laryngeal cancer stage 0 | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002383 | | Narro | | | | | |
| Laryngeal cancer stage I | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002383 | | Narro | | | | | |
| Laryngeal cancer stage II | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002383 | | Narro | | | | | |
| Laryngeal cancer stage III | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002383 | | Narro | | | | | |
| Laryngeal cancer stage IV | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002385 | | Narro | | | | | |
| Laryngeal squamous cell carcinoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002418 | | Narro | | | | | |
| Leiomyosarcoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1002419 | | Narro | | | | | |
| Leiomyosarcoma metastatic | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002419 | | Narro | | | | | |
| Leiomyosarcoma recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002421 | | Narro | | | | | |
| Lentigo maligna | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002422 | | Narro | | | | | |
| Lentigo maligna recurrent | 0 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1002422 | | Narro | | | | | |
| Lentigo maligna stage I | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002422 | | Narro | | | | | |
| Lentigo maligna stage II | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002422 | | Narro | | | | | |
| Lentigo maligna stage III | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002422 | | Narro | | | | | |
| Lentigo maligna stage IV | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002440 | | Narro | | | | | |
| Leydig cell tumour of the testis | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002452 | | Narro | | | | | |
| Linitis plastica | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006152 | | Narro | | | | | |
| Lip and/or oral cavity cancer | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002453 | | Narro | | | | | |
| Lip and/or oral cavity cancer recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002453 | | Narro | | | | | |
| Lip and/or oral cavity cancer stage 0 | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002453 | | Narro | | | | | |
| Lip and/or oral cavity cancer stage I | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002453 | | Narro | | | | | |
| Lip and/or oral cavity cancer stage II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002453 | | Narro | | | | | |
| Lip and/or oral cavity cancer stage III | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002454 | | Narro | | | | | |
| Lip and/or oral cavity cancer stage IV | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002455 | | Narro | | | | | |
| Lip neoplasm malignant stage unspecified | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006405 | | Narro | | | | | |
| Lip squamous cell carcinoma | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002462 | | Narro | | | | | |
| Liposarcoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002462 | | Narro | | | | | |
| Liposarcoma metastatic | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002463 | | Narro | | | | | |
| Liposarcoma recurrent | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007309 | | Narro | | | | | |
| Lobular breast carcinoma in situ | 9 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1002503 | | Narro | | | | | |
| Lung adenocarcinoma | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002503 | | Narro | | | | | |
| Lung adenocarcinoma recurrent | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002503 | | Narro | | | | | |
| Lung adenocarcinoma stage 0 | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002503 | | Narro | | | | | |
| Lung adenocarcinoma stage I | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002503 | | Narro | | | | | |
| Lung adenocarcinoma stage II | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002503 | | Narro | | | | | |
| Lung adenocarcinoma stage III | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002503 | | Narro | | | | | |
| Lung adenocarcinoma stage IV | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005001 | | Narro | | | | | |
| Lung cancer metastatic | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002506 | | Narro | | | | | |
| Lung carcinoma cell type unspecified recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002506 | | Narro | | | | | |
| Lung carcinoma cell type unspecified stage 0 | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002506 | | Narro | | | | | |
| Lung carcinoma cell type unspecified stage I | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002506 | | Narro | | | | | |
| Lung carcinoma cell type unspecified stage II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002506 | | Narro | | | | | |
| Lung carcinoma cell type unspecified stage III | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002507 | | Narro | | | | | |
| Lung carcinoma cell type unspecified stage IV | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006204 | | Narro | | | | | |
| Lung infiltration malignant | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005846 | | Narro | | | | | |
| Lung neoplasm malignant | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007153 | | Narro | | | | | |
| Lung squamous cell carcinoma metastatic | 3 | PT | w | A | 0 | Active | 14.1 | 20.0 |
| | 1002512 | | Narro | | | | | |
| Lung squamous cell carcinoma recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002512 | | Narro | | | | | |
| Lung squamous cell carcinoma stage 0 | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002512 | | Narro | | | | | |
| Lung squamous cell carcinoma stage I | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002512 | | Narro | | | | | |
| Lung squamous cell carcinoma stage II | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002512 | | Narro | | | | | |
| Lung squamous cell carcinoma stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002512 | | Narro | | | | | |
| Lung squamous cell carcinoma stage IV | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006123 | | Narro | | | | | |
| Malignant anorectal neoplasm | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007244 | | Narro | | | | | |
| Malignant blue naevus | 8 | PT | W | A | 0 | Active | 15.1 | 20.0 |
| | 1007434 | | Narro | | | | | |
| Malignant connective tissue neoplasm | 0 | PT | W | A | 0 | Active | 17.0 | 20.0 |
| | 1006123 | | Narro | | | | | |
| Malignant cranial nerve neoplasm | 8 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| - | 1002555 | | Narro | | | | | |
| Malignant fibrous histiocytoma | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1002555 | | Narro | | | | | |
| Malignant fibrous histiocytoma metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1002555 | | Narro | | | | | |
| Malignant fibrous histiocytoma of bone | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1002556 | | Narro | | | | | |
| Malignant fibrous histiocytoma recurrent | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| , | 1007441 | | Narro | | | | | |
| Malignant genitourinary tract neoplasm | 9 | PT | W | A | 0 | Active | 17.0 | 20.0 |
| • • | 1007314 | | Narro | | | | | |
| Malignant giant cell fibrous histiocytoma | 1 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1006544 | | Narro | | | | | |
| Malignant glioma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002556 | | Narro | | | | | |
| Malignant haemangiopericytoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002556 | | Narro | | | | | |
| Malignant haemangiopericytoma metastatic | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002557 | | Narro | | | | | |
| Malignant haemangiopericytoma recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002559 | | Narro | | | | | |
| Malignant hydatidiform mole | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007814 | | Narro | | | | | |
| Malignant joint neoplasm | 5 | PT | W | A | 0 | Active | 19.1 | 20.0 |
| | 1006124 | | Narro | | | | | |
| Malignant mediastinal neoplasm | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002565 | | Narro | | | | | |
| Malignant melanoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002565 | | Narro | | | | | |
| Malignant melanoma in situ | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006370 | | Narro | | | | | |
| Malignant melanoma of eyelid | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002565 | | Narro | | | | | |
| Malignant melanoma of sites other than skin | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002566 | | Narro | | | | | |
| Malignant melanoma stage I | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002566 | | Narro | | | | | |
| Malignant melanoma stage II | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002567 | | Narro | | | | | |
| Malignant melanoma stage III | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002567 | | Narro | | | | | |
| Malignant melanoma stage IV | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007775 | | Narro | | | | | |
| Malignant meningioma metastatic | 8 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1006152 | | Narro | | | | | |
| Malignant mesenchymoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002567 | | Narro | | | | | |
| Malignant mesenchymoma metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002567 | | Narro | | | | | |
| Malignant mesenchymoma recurrent | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006736 | | Narro | | | | | |
| Malignant mesenteric neoplasm | 9 | PT | W | A | 0 | Active | 10.1 | 20.0 |
| | 1006126 | | Narro | | | | | |
| Malignant middle ear neoplasm | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006205 | | Narro | | | | | |
| Malignant muscle neoplasm | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002569 | | Narro | | | | | |
| Malignant neoplasm of ampulla of Vater | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005727 | | Narro | | | | | |
| Malignant neoplasm of auricular cartilage | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002583 | | Narro | | | | | |
| Malignant neoplasm of choroid | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002586 | | Narro | | | | | |
| Malignant neoplasm of conjunctiva | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002587 | | Narro | | | | | |
| Malignant neoplasm of cornea | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002591 | | Narro | | | | | |
| Malignant neoplasm of eye | 0 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| - | 1006369 | | Narro | | | | | |
| Malignant neoplasm of eyelid | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002599 | | Narro | | | | | |
| Malignant neoplasm of islets of Langerhans | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002603 | | Narro | | | | | |
| Malignant neoplasm of lacrimal duct | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002603 | | Narro | | | | | |
| Malignant neoplasm of lacrimal gland | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002618 | | Narro | | | | | |
| Malignant neoplasm of orbit | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1002632 | | Narro | | | | | |
| Malignant neoplasm of paraurethral glands | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| <u> </u> | 1002635 | | Narro | | | | | |
| Malignant neoplasm of placenta | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002635 | | Narro | | | | | |
| Malignant neoplasm of pleura | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007243 | | Narro | | | | | |
| Malignant neoplasm of pleura metastatic | 2 | PT | W | A | 0 | Active | 15.1 | 20.0 |
| | 1002642 | | Narro | | | | | |
| Malignant neoplasm of renal pelvis | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002643 | | Narro | | | | | |
| Malignant neoplasm of retina | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006812 | | Narro | | | | | |
| Malignant neoplasm of seminal vesicle | 4 | PT | W | A | 0 | Active | 11.0 | 20.0 |
| | 1002647 | | Narro | | | | | |
| Malignant neoplasm of spermatic cord | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002647 | | Narro | | | | | |
| Malignant neoplasm of spinal cord | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002653 | | Narro | | | | | |
| Malignant neoplasm of thorax | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007305 | | Narro | | | | | |
| Malignant neoplasm of unknown primary site | 9 | PT | W | Α | 0 | Active | 16.0 | 20.0 |
| | 1002661 | | Narro | | | | | |
| Malignant neoplasm of uterine adnexa | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007730 | | Narro | | | | | |
| Malignant neoplasm papilla of Vater | 3 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1005139 | | Narro | | | | | |
| Malignant neoplasm progression | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006126 | | Narro | | | | | |
| Malignant nervous system neoplasm | 8 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1006205 | | Narro | | | | | |
| Malignant nipple neoplasm | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005312 | | Narro | | | | | |
| Malignant nipple neoplasm female | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005312 | | Narro | | | | | |
| Malignant nipple neoplasm male | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002665 | | Narro | | | | | |
| Malignant oligodendroglioma | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002666 | | Narro | | | | | |
| Malignant ovarian cyst | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002666 | | Narro | | | | | |
| Malignant palate neoplasm | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005494 | | Narro | | | | | |
| Malignant pericardial neoplasm | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006126 | | Narro | | | | | |
| Malignant peritoneal neoplasm | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002667 | | Narro | | | | | |
| Malignant pituitary tumour | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007869 | | Narro | | | | | |
| Malignant polyp | 5 | PT | W | A | 0 | Active | 19.1 | 20.0 |
| | 1006127 | | Narro | | | | | |
| Malignant respiratory tract neoplasm | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007308 | | Narro | | | | | |
| Malignant sweat gland neoplasm | 7 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1006491 | | Narro | | | | | |
| Malignant transformation | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006127 | | Narro | | | | | |
| Malignant urinary tract neoplasm | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007624 | | Narro | | | | | |
| Marjolin's ulcer | 8 | PT | W | A | 0 | Active | 18.0 | 20.0 |
| | 1007987 | | Narro | | | | | |
| Maternal cancer in pregnancy | 7 | PT | W | A | 0 | Active | 20.1 | 20.1 |
| | 1002709 | | Narro | | | | | |
| Medullary carcinoma of breast | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002710 | | Narro | | | | | |
| Medullary thyroid cancer | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002710 | | Narro | | | | | |
| Medulloblastoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006659 | | Narro | | | | | |
| Medulloblastoma recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006660 | | Narro | | | | | |
| Melanoma recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002719 | | Narro | | | | | |
| Meningioma malignant | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002740 | | Narro | | | | | |
| Mesothelioma malignant | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002741 | | Narro | | | | | |
| Mesothelioma malignant recurrent | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007310 | | Narro | | | | | |
| Metaplastic breast carcinoma | 0 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1002745 | | Narro | | | | | |
| Metastases to abdominal cavity | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005166 | | Narro | | | | | |
| Metastases to abdominal wall | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002745 | | Narro | | | | | |
| Metastases to adrenals | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006219 | | Narro | | | | | |
| Metastases to biliary tract | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004972 | | Narro | | | | | |
| Metastases to bladder | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002745 | | Narro | | | | | |
| Metastases to bone | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002745 | | Narro | | | | | |
| Metastases to breast | 4 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1005928 | | Narro | | | | | |
| Metastases to central nervous system | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005166 | | Narro | | | | | |
| Metastases to chest wall | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005166 | | Narro | | | | | |
| Metastases to diaphragm | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005166 | | Narro | | | | | |
| Metastases to Eustachian tube | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004972 | | Narro | | | | | |
| Metastases to eye | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004972 | | Narro | | | | | |
| Metastases to fallopian tube | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005166 | | Narro | | | | | |
| Metastases to gallbladder | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006219 | | Narro | | | | | |
| Metastases to gastrointestinal tract | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004971 | | Narro | | | | | |
| Metastases to heart | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002745 | | Narro | | | | | |
| Metastases to kidney | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005166 | | Narro | | | | | |
| Metastases to larynx | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002745 | | Narro | | | | | |
| Metastases to liver | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002745 | | Narro | | | | | |
| Metastases to lung | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005169 | | Narro | | | | | |
| Metastases to meninges | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005166 | | Narro | | | | | |
| Metastases to mouth | 9 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1004973 | | Narro | | | | | |
| Metastases to muscle | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005167 | | Narro | | | | | |
| Metastases to nasal sinuses | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002746 | | Narro | | | | | |
| Metastases to neck | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006128 | | Narro | | | | | |
| Metastases to nervous system | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1005167 | | Narro | | | | | |
| Metastases to oesophagus | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002746 | | Narro | | | | | |
| Metastases to ovary | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| • | 1004972 | | Narro | | | | | |
| Metastases to pancreas | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| • | 1007091 | | Narro | | | | | |
| Metastases to pelvis | 3 | PT | W | A | 0 | Active | 14.0 | 20.0 |
| • | 1005167 | | Narro | | | | | |
| Metastases to penis | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1005167 | | Narro | | | | | |
| Metastases to perineum | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005167 | | Narro | | | | | |
| Metastases to peripheral nervous system | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005830 | | Narro | | | | | |
| Metastases to peripheral vascular system | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005167 | | Narro | | | | | |
| Metastases to peritoneum | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005167 | | Narro | | | | | |
| Metastases to pharynx | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004972 | | Narro | | | | | |
| Metastases to pituitary gland | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004972 | | Narro | | | | | |
| Metastases to placenta | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002746 | | Narro | | | | | |
| Metastases to pleura | 3 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| • | 1005167 | | Narro | | | | | |
| Metastases to prostate | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005167 | | Narro | | | | | |
| Metastases to rectum | 9 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1006128 | | Narro | | | | | |
| Metastases to reproductive organ | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005168 | | Narro | | | | | |
| Metastases to retroperitoneum | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005168 | | Narro | | | | | |
| Metastases to salivary gland | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002746 | | Narro | | | | | |
| Metastases to skin | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006219 | | Narro | | | | | |
| Metastases to soft tissue | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007826 | | Narro | | | | | |
| Metastases to spinal cord | 7 | PT | w | A | 0 | Active | 19.1 | 20.0 |
| - | 1002746 | | Narro | | | | | |
| Metastases to spine | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1004971 | | Narro | | | | | |
| Metastases to stomach | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005168 | | Narro | | | | | |
| Metastases to testicle | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1002746 | | Narro | | | | | |
| Metastases to the mediastinum | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006160 | | Narro | | | | | |
| Metastases to the respiratory system | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005168 | | Narro | | | | | |
| Metastases to thorax | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004972 | | Narro | | | | | |
| Metastases to thyroid | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007747 | | Narro | | | | | |
| Metastases to tonsils | 6 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1005168 | | Narro | | | | | |
| Metastases to trachea | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005625 | | Narro | | | | | |
| Metastases to urinary tract | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| · | 1004972 | | Narro | | | | | |
| Metastases to uterus | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007555 | | Narro | | | | | |
| Metastases to vagina | 5 | PT | W | A | 0 | Active | 18.0 | 20.0 |
| | 1006219 | | Narro | | | | | |
| Metastasis | 4 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1005830 | | Narro | | | | | |
| Metastatic bronchial carcinoma | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006811 | | Narro | | | | | |
| Metastatic carcinoid tumour | 5 | PT | W | A | 0 | Active | 11.0 | 20.0 |
| | 1005735 | | Narro | | | | | |
| Metastatic carcinoma of the bladder | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007153 | | Narro | | 1 | | | |
| Metastatic choriocarcinoma | 2 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1006391 | | Narro | | 1 | | | |
| Metastatic gastric cancer | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006315 | | Narro | | | | | |
| Metastatic glioma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007524 | | Narro | | | | | |
| Metastatic glucagonoma | 5 | PT | W | A | 0 | Active | 17.1 | 20.0 |
| | 1002748 | | Narro | | | | | |
| Metastatic malignant melanoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006128 | | Narro | | | | | |
| Metastatic neoplasm | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007770 | | Narro | | | | | |
| Metastatic nervous system neoplasm | 3 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1006811 | | Narro | | | | | |
| Metastatic ocular melanoma | 7 | PT | W | A | 0 | Active | 11.0 | 20.0 |
| | 1005051 | | Narro | | | | | |
| Metastatic renal cell carcinoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006688 | | Narro | | | | | |
| Metastatic salivary gland cancer | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006356 | | Narro | | | | | |
| Metastatic squamous cell carcinoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006811 | | Narro | | | | | |
| Metastatic uterine cancer | 6 | PT | W | A | 0 | Active | 11.0 | 20.0 |
| | 1007961 | | Narro | | | | | |
| Microsatellite instability cancer | 8 | PT | W | A | 0 | Active | 20.1 | 20.1 |
| | 1007788 | | Narro | | | | | |
| Mismatch repair cancer syndrome | 8 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1007674 | | Narro | | | | | |
| Mixed adenoneuroendocrine carcinoma | 8 | PT | W | A | 0 | Active | 18.1 | 20.0 |
| | 1002776 | | Narro | | | | | |
| Mixed hepatocellular cholangiocarcinoma | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007313 | | Narro | | | | | |
| Mixed-type liposarcoma | 6 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1007336 | | Narro | | | | | |
| Mucinous adenocarcinoma of appendix | 1 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007310 | | Narro | | | | | |
| Mucinous breast carcinoma | 1 | PT | w | A | 0 | Active | 16.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007336 | | Narro | | | | | |
| Mucinous cystadenocarcinoma of pancreas | 6 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005491 | | Narro | | | | | |
| Mucinous cystadenocarcinoma ovary | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002807 | | Narro | | | | | |
| Mucinous endometrial carcinoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005726 | | Narro | | | | | |
| Mucoepidermoid carcinoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007337 | | Narro | | | | | |
| Mucoepidermoid carcinoma of salivary gland | 1 | PT | W | Α | 0 | Active | 16.0 | 20.0 |
| | 1007767 | | Narro | | | | | |
| Musculoskeletal cancer | 5 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1006694 | | Narro | | | | | |
| Myxofibrosarcoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007313 | | Narro | | | | | |
| Myxoid liposarcoma | 7 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| , | 1007905 | | Narro | | | | | |
| Naevoid melanoma | 4 | PT | W | Α | 0 | Active | 20.0 | 20.0 |
| | 1002872 | | Narro | | | | | |
| Nasal cavity cancer | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1002876 | | Narro | | | | | |
| Nasal sinus cancer | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006130 | | Narro | | | | | |
| Nasopharyngeal cancer | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007910 | | Narro | | | | | |
| Nasopharyngeal cancer metastatic | 4 | PT | W | A | 0 | Active | 20.0 | 20.0 |
| | 1002878 | | Narro | | | | | |
| Nasopharyngeal cancer recurrent | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1002878 | | Narro | | | | | |
| Nasopharyngeal cancer stage 0 | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| · - | 1002878 | | Narro | | | | | |
| Nasopharyngeal cancer stage I | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002879 | | Narro | | | | | |
| Nasopharyngeal cancer stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002879 | | Narro | | | | | |
| Nasopharyngeal cancer stage III | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002879 | | Narro | | | | | |
| Nasopharyngeal cancer stage IV | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004979 | | Narro | | | | | |
| Neonatal neuroblastoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002899 | | Narro | | | | | |
| Neoplasm malignant | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002914 | | Narro | | | | | |
| Nephroblastoma | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002926 | | Narro | | | | | |
| Neuroblastoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006659 | | Narro | | | | | |
| Neuroblastoma recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007310 | | Narro | | | | | |
| Neuroendocrine breast tumour | 3 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005727 | | Narro | | | | | |
| Neuroendocrine carcinoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007154 | | Narro | | | | | |
| Neuroendocrine carcinoma metastatic | 2 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1007834 | | Narro | | | | | |
| Neuroendocrine carcinoma of the bladder | 1 | PT | W | A | 0 | Active | 19.1 | 20.0 |
| | 1002926 | | Narro | | | | | |
| Neuroendocrine carcinoma of the skin | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005239 | | Narro | | | | | |
| Neuroendocrine tumour | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007817 | | Narro | | | | | |
| Neuroendocrine tumour of the lung | 4 | PT | W | A | 0 | Active | 19.1 | 20.0 |
| | 1007817 | | Narro | | | | | |
| Neuroendocrine tumour of the lung metastatic | 5 | PT | W | A | 0 | Active | 19.1 | 20.0 |
| | 1006152 | | Narro | | | | | |
| Neurofibrosarcoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002927 | | Narro | | | | | |
| Neurofibrosarcoma metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1002927 | | Narro | | | | | |
| Neurofibrosarcoma recurrent | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002948 | | Narro | | | | | |
| Nodular melanoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006587 | | Narro | | | | | |
| Nongerminomatous germ cell tumour of the CNS | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007332 | | Narro | | | | | |
| Jonkeratinising carcinoma of nasopharynx | 5 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1006187 | | Narro | | | | | |
| Non-renal cell carcinoma of kidney | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006187 | | Narro | | | | | |
| Non-small cell lung cancer | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005951 | | Narro | | | | | |
| Non-small cell lung cancer metastatic | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002951 | | Narro | | | | | |
| Non-small cell lung cancer recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1002951 | | Narro | | | | | |
| Non-small cell lung cancer stage 0 | 6 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1002951 | | Narro | | | | | |
| Non-small cell lung cancer stage I | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002951 | | Narro | | | | | |
| Non-small cell lung cancer stage II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002951 | | Narro | | | | | |
| Non-small cell lung cancer stage III | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002952 | | Narro | | | | | |
| Non-small cell lung cancer stage IIIA | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002952 | | Narro | | | | | |
| Non-small cell lung cancer stage IIIB | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1002952 | | Narro | | | | | |
| Non-small cell lung cancer stage IV | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| <u> </u> | 1007829 | | Narro | | | | | |
| NUT midline carcinoma | 5 | PT | W | A | 0 | Active | 19.1 | 20.0 |
| | 1005509 | | Narro | | | | | |
| Ocular cancer metastatic | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1005741 | | Narro | | | | | |
| Ocular haemangiopericytoma | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003013 | | Narro | | | | | |
| Oesophageal adenocarcinoma | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003014 | | Narro | | | | | |
| Oesophageal adenocarcinoma recurrent | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003014 | | Narro | | | | | |
| Oesophageal adenocarcinoma stage 0 | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003014 | | Narro | | | | | |
| Oesophageal adenocarcinoma stage I | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003014 | | Narro | | | | | |
| Oesophageal adenocarcinoma stage II | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003014 | | Narro | | | | | |
| Oesophageal adenocarcinoma stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003014 | | Narro | | | | | |
| Oesophageal adenocarcinoma stage IV | 5 | PT | w | Α | 0 | Active | 10.0 | 20.0 |
| | 1005510 | | Narro | | | | | |
| Oesophageal cancer metastatic | 2 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1003015 | | Narro | | | | | |
| Oesophageal carcinoma | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003015 | | Narro | | | | | |
| Oesophageal carcinoma recurrent | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003016 | | Narro | | | | | |
| Oesophageal carcinoma stage 0 | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006153 | | Narro | | | | | |
| Oesophageal squamous cell carcinoma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005852 | | Narro | | | | | |
| Oesophageal squamous cell carcinoma metastatic | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003018 | | Narro | | | | | |
| Oesophageal squamous cell carcinoma recurrent | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003018 | | Narro | | | | | |
| Desophageal squamous cell carcinoma stage 0 | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| <del>-</del> | 1003018 | | Narro | | | | | |
| Oesophageal squamous cell carcinoma stage I | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1003019 | | Narro | | | | | |
| Oesophageal squamous cell carcinoma stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003019 | | Narro | | | | | |
| Oesophageal squamous cell carcinoma stage III | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003019 | | Narro | | | | | |
| Oesophageal squamous cell carcinoma stage IV | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007057 | | Narro | | | | | |
| Oestrogen receptor positive breast cancer | 7 | PT | W | A | 0 | Active | 13.1 | 20.0 |
| | 1007313 | | Narro | | | | | |
| Oligoastrocytoma | 1 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1003028 | | Narro | | | | | |
| Oligodendroglioma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007333 | | Narro | | | | | |
| Optic glioma | 8 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005509 | | Narro | | | | | |
| Oral cavity cancer metastatic | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| , | 1003109 | | Narro | | | | | |
| Oropharyngeal cancer | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003109 | | Narro | | | | | |
| Oropharyngeal cancer recurrent | 8 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1003109 | | Narro | | | | | |
| Oropharyngeal cancer stage 0 | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003110 | | Narro | | | | | |
| Oropharyngeal cancer stage I | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003110 | | Narro | | | | | |
| Oropharyngeal cancer stage II | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003110 | | Narro | | | | | |
| Oropharyngeal cancer stage III | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006409 | | Narro | | | | | |
| Oropharyngeal cancer stage IV | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1003110 | | Narro | | | | | |
| Oropharyngeal lymphoepithelioma | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003111 | | Narro | | | | | |
| Oropharyngeal squamous cell carcinoma | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1003129 | | Narro | | | | | |
| Osteosarcoma | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003129 | | Narro | | | | | |
| Osteosarcoma metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003129 | | Narro | | | | | |
| Osteosarcoma recurrent | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005510 | | Narro | | | | | |
| Otic cancer metastatic | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003312 | | Narro | | | | | |
| Ovarian cancer | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005752 | | Narro | | | | | |
| Ovarian cancer metastatic | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006669 | | Narro | | | | | |
| Ovarian cancer recurrent | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007090 | | Narro | | | | | |
| Ovarian cancer stage I | 5 | PT | W | A | 0 | Active | 14.0 | 20.0 |
| | 1007090 | | Narro | | | | | |
| Ovarian cancer stage II | 6 | PT | W | A | 0 | Active | 14.0 | 20.0 |
| | 1007090 | | Narro | | | | | |
| Ovarian cancer stage III | 7 | PT | W | Α | 0 | Active | 14.0 | 20.0 |
| | 1007090 | | Narro | | | | | |
| Ovarian cancer stage IV | 8 | PT | W | A | 0 | Active | 14.0 | 20.0 |
| | 1007326 | | Narro | | | | | |
| Ovarian clear cell carcinoma | 8 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1003314 | | Narro | | | | | |
| Ovarian dysgerminoma stage I | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003314 | | Narro | | | | | |
| Ovarian dysgerminoma stage II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003315 | | Narro | | | | | |
| Ovarian dysgerminoma stage III | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003315 | | Narro | | | | | |
| Ovarian dysgerminoma stage IV | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005275 | | Narro | | | | | |
| Ovarian dysgerminoma stage unspecified | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1005626 | | Narro | | | | | |
| Ovarian embryonal carcinoma | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007326 | | Narro | | | | | |
| Ovarian endometrioid carcinoma | 9 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1006132 | | Narro | | | | | |
| Ovarian epithelial cancer | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003315 | | Narro | | | | | |
| Ovarian epithelial cancer metastatic | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003316 | | Narro | | | | | |
| Ovarian epithelial cancer recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003316 | | Narro | | | | | |
| Ovarian epithelial cancer stage I | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003316 | | Narro | | | | | |
| Ovarian epithelial cancer stage II | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003316 | | Narro | | | | | |
| Ovarian epithelial cancer stage III | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003316 | | Narro | | | | | |
| Ovarian epithelial cancer stage IV | 4 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1006189 | | Narro | | | | | |
| Ovarian germ cell cancer | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006189 | | Narro | | | | | |
| Ovarian germ cell cancer stage I | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1006189 | | Narro | | | | | |
| Ovarian germ cell cancer stage II | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006189 | | Narro | | | | | |
| Ovarian germ cell cancer stage III | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006189 | | Narro | | | | | |
| Ovarian germ cell cancer stage IV | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007326 | | Narro | | | | | |
| Ovarian germ cell choriocarcinoma | 2 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1003318 | | Narro | | | | | |
| Ovarian germ cell choriocarcinoma stage I | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| - | 1003318 | | Narro | | | | | |
| Ovarian germ cell choriocarcinoma stage II | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1003319 | | Narro | | | | | |
| Ovarian germ cell choriocarcinoma stage III | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003319 | | Narro | | | | | |
| Ovarian germ cell choriocarcinoma stage IV | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003319 | | Narro | | | | | |
| Ovarian germ cell embryonal carcinoma stage I | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003320 | | Narro | | | | | |
| Ovarian germ cell embryonal carcinoma stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003320 | | Narro | | | | | |
| Ovarian germ cell embryonal carcinoma stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003320 | | Narro | | | | | |
| Ovarian germ cell embryonal carcinoma stage IV | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007326 | | Narro | | | | | |
| Ovarian germ cell endodermal sinus tumour | 3 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1003321 | | Narro | | | | | |
| Ovarian germ cell endodermal sinus tumour stage I | 8 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1003321 | | Narro | | | | | |
| Ovarian germ cell endodermal sinus tumour stage II | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003322 | | Narro | | | | | |
| Ovarian germ cell endodermal sinus tumour stage III | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003322 | | Narro | | | | | |
| Ovarian germ cell endodermal sinus tumour stage IV | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1007326 | | Narro | | | | | |
| Ovarian germ cell polyembryoma | 4 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1003322 | | Narro | | | | | |
| Ovarian germ cell polyembryoma stage I | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003322 | | Narro | | | | | |
| Ovarian germ cell polyembryoma stage II | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003323 | | Narro | | | | | |
| Ovarian germ cell polyembryoma stage III | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003323 | | Narro | | | | | |
| Ovarian germ cell polyembryoma stage IV | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007326 | | Narro | | | | | |
| Ovarian germ cell teratoma | 5 | PT | W | A | 0 | Active | 16.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1003323 | | Narro | | | | | |
| Ovarian germ cell teratoma stage I | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003324 | | Narro | | | | | |
| Ovarian germ cell teratoma stage II | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003324 | | Narro | | | | | |
| Ovarian germ cell teratoma stage III | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003324 | | Narro | | | | | |
| Ovarian germ cell teratoma stage IV | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007325 | | Narro | | | | | |
| Ovarian germ cell tumour mixed | 9 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005737 | | Narro | | | | | |
| Ovarian granulosa-theca cell tumour | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003326 | | Narro | | | | | |
| Ovarian low malignant potential tumour | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006585 | | Narro | | | | | |
| Ovarian stromal cancer | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003336 | | Narro | | | | | |
| Paget's disease of nipple | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003336 | | Narro | | | | | |
| Paget's disease of penis | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003336 | | Narro | | | | | |
| Paget's disease of the vulva | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003357 | | Narro | | | | | |
| Pancoast's tumour | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003360 | | Narro | | | | | |
| Pancreatic carcinoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003361 | | Narro | | | | | |
| Pancreatic carcinoma metastatic | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003361 | | Narro | | | | | |
| Pancreatic carcinoma recurrent | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005932 | | Narro | | | | | |
| Pancreatic carcinoma stage 0 | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005932 | | Narro | | | | | |
| Pancreatic carcinoma stage I | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1005932 | | Narro | | | | | |
| Pancreatic carcinoma stage II | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005932 | | Narro | | | | | |
| Pancreatic carcinoma stage III | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005932 | | Narro | | | | | |
| Pancreatic carcinoma stage IV | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006751 | | Narro | | | | | |
| Pancreatic neuroendocrine tumour | 7 | PT | W | A | 0 | Active | 10.1 | 20.0 |
| | 1006890 | | Narro | | | | | |
| Pancreatic neuroendocrine tumour metastatic | 9 | PT | W | A | 0 | Active | 12.0 | 20.0 |
| | 1005500 | | Narro | | | | | |
| Pancreatic sarcoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007336 | | Narro | | | | | |
| Pancreatoblastoma | 7 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007849 | | Narro | | | | | |
| Papillary renal cell carcinoma | 3 | PT | w | A | 0 | Active | 19.1 | 20.0 |
| | 1003370 | | Narro | | | | | |
| Papillary serous endometrial carcinoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| • | 1003370 | | Narro | | | | | |
| Papillary thyroid cancer | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003379 | | Narro | | | | | |
| Paraganglion neoplasm malignant | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006190 | | Narro | | | | | |
| Paranasal sinus and nasal cavity malignant neoplasm | 9 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| Paranasal sinus and nasal cavity malignant neoplasm | 1003385 | | Narro | | | | | |
| recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Paranasal sinus and nasal cavity malignant neoplasm | 1003385 | | Narro | | | | | |
| stage 0 | 6 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| Paranasal sinus and nasal cavity malignant neoplasm | 1003385 | | Narro | 1 | 1 | | | |
| stage I | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Paranasal sinus and nasal cavity malignant neoplasm | 1003385 | | Narro | | | | | |
| stage II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Paranasal sinus and nasal cavity malignant neoplasm | 1003385 | | Narro | 1 | 1 | | | |
| stage III | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| Paranasal sinus and nasal cavity malignant neoplasm | 1003386 | | Narro | | | | | |
| stage IV | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003396 | | Narro | | | | | |
| Parathyroid tumour malignant | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003429 | | Narro | | | | | |
| Penile cancer | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005963 | | Narro | | | | | |
| Penile squamous cell carcinoma | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003432 | | Narro | | | | | |
| Penis carcinoma metastatic | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003433 | | Narro | | | | | |
| Penis carcinoma recurrent | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003433 | | Narro | | | | | |
| Penis carcinoma stage I | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1003433 | | Narro | | | | | |
| Penis carcinoma stage II | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003433 | | Narro | | | | | |
| Penis carcinoma stage III | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003433 | | Narro | | | | | |
| Penis carcinoma stage IV | 5 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1007306 | | Narro | | | | | |
| Pericardial mesothelioma malignant | 6 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| <u> </u> | 1003448 | | Narro | | | | | |
| Pericardial mesothelioma malignant recurrent | 0 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1003459 | | Narro | | | | | |
| Peripheral nerve sheath tumour malignant | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006134 | | Narro | | | | | |
| Peripheral neuroepithelioma of bone | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| • | 1003460 | 1 | Narro | 1 | 1 | | | |
| Peripheral neuroepithelioma of bone metastatic | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| 1 1 | 1003460 | | Narro | | | | | |
| Peripheral neuroepithelioma of bone recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005764 | | Narro | | 1 | | | |
| Peripheral neuroepithelioma of soft tissue | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007310 | | Narro | | | | | |
| Peripheral primitive neuroectodermal bone tumour | 7 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| Peripheral primitive neuroectodermal tumour of soft | 1007314 | | Narro | | | | | |
| tissue | 4 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1006897 | | Narro | | | | | |
| Peritoneal carcinoma metastatic | 4 | PT | w | A | 0 | Active | 12.0 | 20.0 |
| | 1005655 | | Narro | | | | | |
| Peritoneal mesothelioma malignant | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003467 | | Narro | | | | | |
| Peritoneal mesothelioma malignant recurrent | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005194 | | Narro | | | | | |
| Peritoneal sarcoma | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005171 | | Narro | | | | | |
| Phaeochromocytoma malignant | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003481 | | Narro | | | | | |
| Pharyngeal cancer | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005510 | | Narro | | | | | |
| Pharyngeal cancer metastatic | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003481 | | Narro | | | | | |
| Pharyngeal cancer recurrent | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003481 | | Narro | | | | | |
| Pharyngeal cancer stage 0 | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003481 | | Narro | | | | | |
| Pharyngeal cancer stage I | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003481 | | Narro | | | | | |
| Pharyngeal cancer stage II | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003481 | | Narro | | | | | |
| Pharyngeal cancer stage III | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003481 | | Narro | | | | | |
| Pharyngeal cancer stage IV | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007561 | | Narro | | | | | |
| Pilomatrix carcinoma | 4 | PT | w | A | 0 | Active | 18.0 | 20.0 |
| | 1003505 | | Narro | | | | | |
| Pineal germinoma | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006153 | | Narro | | | | | |
| Pineal parenchymal neoplasm malignant | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005048 | | Narro | | | | | |
| Pinealoblastoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005510 | | Narro | | | | | |
| Pituitary cancer metastatic | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005783 | | Narro | | | | | |
| Pituitary neoplasm malignant recurrent | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007313 | | Narro | | | | | |
| Pleomorphic liposarcoma | 8 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007314 | | Narro | | | | | |
| Pleomorphic malignant fibrous histiocytoma | 3 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1003560 | | Narro | | | | | |
| Pleural mesothelioma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005951 | | Narro | | | | | |
| Pleural mesothelioma malignant | 8 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003560 | | Narro | | | | | |
| Pleural mesothelioma malignant recurrent | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005195 | | Narro | | | | | |
| Pleural sarcoma | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007660 | | Narro | | | | | |
| Poorly differentiated thyroid carcinoma | 3 | PT | w | A | 0 | Active | 18.1 | 20.0 |
| | 1006360 | | Narro | | | | | |
| Porocarcinoma | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003633 | | Narro | | | | | |
| Postcricoid cancer | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005784 | | Narro | | | | | |
| Primitive neuroectodermal tumour | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006891 | | Narro | | | | | |
| Primitive neuroectodermal tumour metastatic | 0 | PT | w | A | 0 | Active | 12.0 | 20.0 |
| | 1006086 | | Narro | | | | | |
| Prostate cancer | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003690 | | Narro | | | | | |
| Prostate cancer metastatic | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1003691 | | Narro | | | | | |
| Prostate cancer recurrent | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003691 | | Narro | | | | | |
| Prostate cancer stage 0 | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003691 | | Narro | | | | | |
| Prostate cancer stage I | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003691 | | Narro | | | | | |
| Prostate cancer stage II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003691 | | Narro | | | | | |
| Prostate cancer stage III | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003692 | | Narro | | | | | |
| Prostate cancer stage IV | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005180 | | Narro | | | | | |
| Pseudosarcoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003773 | | Narro | | | | | |
| Queyrat erythroplasia | 2 | PT | W | A | 0 | Active | 17.0 | 20.0 |
| | 1003801 | | Narro | | | | | |
| Rectal adenocarcinoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003803 | | Narro | | | | | |
| Rectal cancer | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005509 | | Narro | | | | | |
| Rectal cancer metastatic | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003804 | | Narro | | | | | |
| Rectal cancer recurrent | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003804 | | Narro | | | | | |
| Rectal cancer stage 0 | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003804 | | Narro | | | | | |
| Rectal cancer stage I | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003804 | | Narro | | | | | |
| Rectal cancer stage II | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| <del>-</del> | 1003805 | | Narro | | | | | |
| Rectal cancer stage III | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| - | 1003805 | | Narro | | | | | |
| Rectal cancer stage IV | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1003808 | | Narro | | | | | |
| Rectosigmoid cancer | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006972 | | Narro | | | | | |
| Rectosigmoid cancer metastatic | 8 | PT | W | A | 0 | Active | 13.0 | 20.0 |
| | 1003809 | | Narro | | | | | |
| Rectosigmoid cancer recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003809 | | Narro | | | | | |
| Rectosigmoid cancer stage 0 | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003809 | | Narro | | | | | |
| Rectosigmoid cancer stage I | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003809 | | Narro | | | | | |
| Rectosigmoid cancer stage II | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003809 | | Narro | | | | | |
| Rectosigmoid cancer stage III | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003809 | | Narro | | | | | |
| Rectosigmoid cancer stage IV | 9 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1003811 | | Narro | | | | | |
| Recurrent cancer | 1 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1007030 | | Narro | | | | | |
| Refractory cancer | 8 | PT | W | A | 0 | Active | 13.0 | 20.0 |
| | 1003838 | | Narro | | | | | |
| Renal cancer | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005001 | | Narro | | | | | |
| Renal cancer metastatic | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003839 | | Narro | | | | | |
| Renal cancer recurrent | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003839 | | Narro | | | | | |
| Renal cancer stage I | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1003839 | | Narro | | | | | |
| Renal cancer stage II | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003839 | | Narro | | | | | |
| Renal cancer stage III | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1003839 | | Narro | | | | | |
| Renal cancer stage IV | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1006794 | | Narro | | | | | |
| Renal cell carcinoma | 6 | PT | w | A | 0 | Active | 11.0 | 20.0 |
| | 1003841 | | Narro | | | | | |
| Renal cell carcinoma recurrent | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003841 | | Narro | | | | | |
| Renal cell carcinoma stage I | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003841 | | Narro | | | | | |
| Renal cell carcinoma stage II | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003841 | | Narro | | | | | |
| Renal cell carcinoma stage III | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003841 | | Narro | | | | | |
| Renal cell carcinoma stage IV | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003872 | | Narro | | | | | |
| Respiratory tract carcinoma in situ | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003887 | | Narro | | | | | |
| Retinal melanoma | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003891 | | Narro | | | | | |
| Retinoblastoma | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003897 | | Narro | | | | | |
| Retroperitoneal cancer | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006248 | | Narro | | | | | |
| Retroperitoneal neoplasm metastatic | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007333 | | Narro | | | | | |
| Rhabdoid tumour | 4 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1003901 | | Narro | | | | | |
| Rhabdoid tumour of the kidney | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1003902 | | Narro | | | | | |
| Rhabdomyosarcoma | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003902 | | Narro | | | | | |
| Rhabdomyosarcoma recurrent | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007313 | | Narro | | | | | |
| Round cell liposarcoma | 9 | PT | w | A | 0 | Active | 16.0 | 20.0 |
| | 1006193 | | Narro | | | | | |
| Salivary gland cancer | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1003939 | | Narro | | | | | |
| Salivary gland cancer recurrent | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003939 | | Narro | | | | | |
| Salivary gland cancer stage 0 | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003940 | | Narro | | | | | |
| Salivary gland cancer stage I | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003940 | | Narro | | | | | |
| Salivary gland cancer stage II | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003940 | | Narro | | | | | |
| Salivary gland cancer stage III | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003940 | | Narro | | | | | |
| Salivary gland cancer stage IV | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003949 | | Narro | | | | | |
| Sarcoma | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006859 | | Narro | | | | | |
| Sarcoma metastatic | 5 | PT | W | Α | 0 | Active | 11.1 | 20.0 |
| | 1003949 | | Narro | | | | | |
| Sarcoma of skin | 5 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1003949 | | Narro | | | | | |
| Sarcoma uterus | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007306 | | Narro | | | | | |
| Sarcomatoid mesothelioma | 5 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1003950 | | Narro | | | | | |
| Sarcomatosis | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1003974 | | Narro | | | | | |
| Scrotal cancer | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006878 | | Narro | | | | | |
| Sebaceous carcinoma | 4 | PT | W | A | 0 | Active | 12.0 | 20.0 |
| | 1003980 | | Narro | | | | | |
| Second primary malignancy | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| <u> </u> | 1003995 | | Narro | | | | | |
| Seminoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007336 | | Narro | | | | | |
| Serous cystadenocarcinoma of pancreas | 8 | PT | W | A | 0 | Active | 16.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1005491 | | Narro | | | | | |
| Serous cystadenocarcinoma ovary | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005726 | | Narro | | | | | |
| Signet-ring cell carcinoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005510 | | Narro | | | | | |
| Sinus cancer metastatic | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007289 | | Narro | | | | | |
| Skin angiosarcoma | 1 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1004080 | | Narro | | | | | |
| Skin cancer | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005511 | | Narro | | | | | |
| Skin cancer metastatic | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007731 | | Narro | | | | | |
| Skin squamous cell carcinoma metastatic | 4 | PT | W | A | 0 | Active | 19.0 | 20.0 |
| | 1004105 | | Narro | | | | | |
| Small cell carcinoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004105 | | Narro | | | | | |
| Small cell carcinoma of the cervix | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004106 | | Narro | | | | | |
| Small cell lung cancer | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004106 | | Narro | | | | | |
| Small cell lung cancer extensive stage | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004106 | | Narro | | | | | |
| Small cell lung cancer limited stage | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005951 | | Narro | | | | | |
| Small cell lung cancer metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004107 | | Narro | | | | | |
| Small cell lung cancer recurrent | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007337 | | Narro | | | | | |
| Small intestine adenocarcinoma | 3 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1005418 | | Narro | | | | | |
| Small intestine carcinoma | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004112 | | Narro | | | | | |
| Small intestine carcinoma metastatic | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1004112 | | Narro | | | | | |
| Small intestine carcinoma recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005936 | | Narro | | | | | |
| Small intestine carcinoma stage 0 | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005936 | | Narro | | | | | |
| Small intestine carcinoma stage I | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005937 | | Narro | | | | | |
| Small intestine carcinoma stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005937 | | Narro | | | | | |
| Small intestine carcinoma stage III | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005937 | | Narro | | | | | |
| Small intestine carcinoma stage IV | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004112 | | Narro | | | | | |
| Small intestine leiomyosarcoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007533 | | Narro | | | | | |
| Soft tissue sarcoma | 3 | PT | W | A | 0 | Active | 17.1 | 20.0 |
| | 1006934 | | Narro | | | | | |
| Solid pseudopapillary tumour of the pancreas | 5 | PT | W | A | 0 | Active | 12.1 | 20.0 |
| | 1007311 | | Narro | | | | | |
| Spermatocytic seminoma | 8 | PT | W | Α | 0 | Active | 16.0 | 20.0 |
| | 1004158 | | Narro | | | | | |
| Spinal meningioma malignant | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004906 | | Narro | | | | | |
| Spindle cell sarcoma | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007930 | | Narro | | | | | |
| Squamous cell breast carcinoma | 7 | PT | W | A | 0 | Active | 20.0 | 20.0 |
| | 1004182 | | Narro | | | | | |
| Squamous cell carcinoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006012 | | Narro | | | | | |
| Squamous cell carcinoma of head and neck | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004182 | | Narro | | | | | |
| Squamous cell carcinoma of lung | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006647 | | Narro | | | | | |
| Squamous cell carcinoma of pharynx | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1004183 | | Narro | | | | | |
| Squamous cell carcinoma of skin | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004184 | | Narro | | | | | |
| Squamous cell carcinoma of the cervix | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004184 | | Narro | | | | | |
| Squamous cell carcinoma of the hypopharynx | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004185 | | Narro | | | | | |
| Squamous cell carcinoma of the oral cavity | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004186 | | Narro | | | | | |
| Squamous cell carcinoma of the tongue | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004186 | | Narro | | | | | |
| Squamous cell carcinoma of the vagina | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| • | 1004187 | | Narro | | | | | |
| Squamous cell carcinoma of the vulva | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004188 | | Narro | | | | | |
| Squamous endometrial carcinoma | 3 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1005949 | | Narro | | | | | |
| Stewart-Treves syndrome | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004254 | | Narro | | | | | |
| Superficial spreading melanoma stage I | 9 | PT | W | Α | 0 | Active | 10.0 | 20.0 |
| | 1004255 | | Narro | | | | | |
| Superficial spreading melanoma stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004255 | | Narro | | | | | |
| Superficial spreading melanoma stage III | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004255 | | Narro | | | | | |
| Superficial spreading melanoma stage IV | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004255 | | Narro | | | | | |
| Superficial spreading melanoma stage unspecified | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004286 | | Narro | | | | | |
| Synovial sarcoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1004286 | | Narro | | | | | |
| Synovial sarcoma metastatic | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004286 | | Narro | | | | | |
| Synovial sarcoma recurrent | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1005510 | | Narro | | | | | |
| Testicular cancer metastatic | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006212 | | Narro | | | | | |
| Testicular choriocarcinoma | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006981 | | Narro | | | | | |
| Testicular choriocarcinoma recurrent | 2 | PT | W | A | 0 | Active | 13.0 | 20.0 |
| | 1004330 | | Narro | | | | | |
| Testicular choriocarcinoma stage I | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004330 | | Narro | | | | | |
| Testicular choriocarcinoma stage II | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004330 | | Narro | | | | | |
| Testicular choriocarcinoma stage III | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006212 | | Narro | | | | | |
| Testicular embryonal carcinoma | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004330 | | Narro | | | | | |
| Testicular embryonal carcinoma stage I | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004331 | | Narro | | | | | |
| Testicular embryonal carcinoma stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004331 | | Narro | | | | | |
| Testicular embryonal carcinoma stage III | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006137 | | Narro | | | | | |
| Testicular germ cell cancer | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006869 | | Narro | | | | | |
| Testicular germ cell cancer metastatic | 4 | PT | W | A | 0 | Active | 11.1 | 20.0 |
| | 1007311 | | Narro | | | | | |
| Testicular germ cell tumour mixed | 9 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1004333 | | Narro | | | | | |
| Testicular germ cell tumour mixed stage I | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004333 | | Narro | | | | | |
| Testicular germ cell tumour mixed stage II | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004333 | | Narro | | | | | |
| Testicular germ cell tumour mixed stage III | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1005734 | | Narro | | | | | |
| Testicular leiomyosarcoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007312 | | Narro | | | | | |
| Testicular malignant teratoma | 0 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1004333 | | Narro | | | | | |
| Testicular malignant teratoma stage I | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004334 | | Narro | | | | | |
| Testicular malignant teratoma stage II | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004334 | | Narro | | | | | |
| Testicular malignant teratoma stage III | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006212 | | Narro | | | | | |
| Testicular seminoma (pure) | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004335 | | Narro | | | | | |
| Testicular seminoma (pure) stage I | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004335 | | Narro | | | | | |
| Testicular seminoma (pure) stage II | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004335 | | Narro | | | | | |
| Testicular seminoma (pure) stage III | 2 | PT | w | Α | 0 | Active | 10.0 | 20.0 |
| | 1007312 | | Narro | | | | | |
| Testicular yolk sac tumour | 1 | PT | w | Α | 0 | Active | 16.0 | 20.0 |
| | 1004335 | | Narro | | | | | |
| Testicular yolk sac tumour stage I | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004335 | | Narro | | | | | |
| Testicular yolk sac tumour stage II | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| • | 1004335 | | Narro | | | | | |
| Testicular yolk sac tumour stage III | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| <del>-</del> | 1005764 | | Narro | | | | | |
| Testis cancer | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1006981 | | Narro | | | | | |
| Testis cancer recurrent | 3 | PT | W | A | 0 | Active | 13.0 | 20.0 |
| | 1004351 | | Narro | | | | | |
| Throat cancer | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006647 | | Narro | | | | | |
| Thyroid cancer | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| - | 1005510 | | Narro | | | | | |
| Thyroid cancer metastatic | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1007216 | | Narro | | | | | |
| Thyroid cancer recurrent | 2 | PT | w | A | 0 | Active | 15.0 | 20.0 |
| | 1007056 | | Narro | | | | | |
| Thyroid cancer stage 0 | 7 | PT | w | A | 0 | Active | 13.1 | 20.0 |
| | 1007102 | | Narro | | | | | |
| Thyroid cancer stage I | 7 | PT | w | A | 0 | Active | 14.0 | 20.0 |
| | 1007102 | | Narro | | | | | |
| Thyroid cancer stage II | 8 | PT | w | A | 0 | Active | 14.0 | 20.0 |
| | 1007102 | | Narro | | | | | |
| Thyroid cancer stage III | 9 | PT | w | A | 0 | Active | 14.0 | 20.0 |
| | 1007103 | | Narro | | | | | |
| Thyroid cancer stage IV | 0 | PT | w | A | 0 | Active | 14.0 | 20.0 |
| | 1005510 | | Narro | | | | | |
| Tongue cancer metastatic | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007125 | | Narro | | | | | |
| Tongue cancer recurrent | 1 | PT | W | A | 0 | Active | 14.1 | 20.0 |
| | 1005842 | | Narro | | | | | |
| Tongue carcinoma stage 0 | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005843 | | Narro | | | | | |
| Tongue carcinoma stage I | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005843 | | Narro | | | | | |
| Tongue carcinoma stage II | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005843 | | Narro | | | | | |
| Tongue carcinoma stage III | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1005843 | | Narro | | | | | |
| Tongue carcinoma stage IV | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004396 | | Narro | | | | | |
| Tongue neoplasm malignant stage unspecified | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004400 | | Narro | | | | | |
| Tonsil cancer | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007279 | | Narro | | | | | |
| Tonsil cancer metastatic | 2 | PT | w | A | 0 | Active | 15.1 | 20.0 |
| | 1004428 | | Narro | | | | | |
| Tracheal cancer | 5 | PT | w | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| Transitional cell cancer of renal pelvis and ureter | 1004440 | | Narro | | | | | |
| metastatic | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004440 | | Narro | | | | | |
| Transitional cell cancer of the renal pelvis and ureter | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Transitional cell cancer of the renal pelvis and ureter | 1004440 | | Narro | | | | | |
| localised | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| Transitional cell cancer of the renal pelvis and ureter | 1004441 | | Narro | | | | | |
| recurrent | 0 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| Transitional cell cancer of the renal pelvis and ureter | 1004441 | | Narro | | | | | |
| regional | 1 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004441 | | Narro | | | | | |
| Transitional cell carcinoma | 2 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1007108 | | Narro | | | | | |
| Transitional cell carcinoma metastatic | 0 | PT | w | A | 0 | Active | 14.0 | 20.0 |
| | 1007705 | | Narro | | | | | |
| Transitional cell carcinoma recurrent | 1 | PT | W | A | 0 | Active | 18.1 | 20.0 |
| | 1004442 | | Narro | | | | | |
| Transitional cell carcinoma urethra | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007556 | | Narro | | | | | |
| Triple negative breast cancer | 6 | PT | W | A | 0 | Active | 18.0 | 20.0 |
| | 1007310 | | Narro | | | | | |
| Tubular breast carcinoma | 4 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007696 | | Narro | | | | | |
| Tumour budding | 9 | PT | W | Α | 0 | Active | 18.1 | 20.0 |
| | 1007336 | | Narro | | | | | |
| Undifferentiated carcinoma of colon | 2 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| | 1007332 | | Narro | | | | | |
| Undifferentiated nasopharyngeal carcinoma | 8 | PT | W | A | 0 | Active | 16.0 | 20.0 |
| 1 2 0 | 1004551 | | Narro | | | | | |
| Undifferentiated sarcoma | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004639 | | Narro | | | | | |
| Ureteric cancer | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004639 | | Narro | | | | | |
| Ureteric cancer local | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1004639 | | Narro | | | | | |
| Ureteric cancer metastatic | 4 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004639 | | Narro | | | | | |
| Ureteric cancer recurrent | 6 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004639 | | Narro | | | | | |
| Ureteric cancer regional | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004643 | | Narro | | | | | |
| Urethral cancer | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004643 | | Narro | | | | | |
| Urethral cancer metastatic | 3 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004643 | | Narro | | | | | |
| Urethral cancer recurrent | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1007279 | | Narro | | | | | |
| Urethral melanoma metastatic | 3 | PT | W | A | 0 | Active | 15.1 | 20.0 |
| | 1005169 | | Narro | | | | | |
| Urinary bladder sarcoma | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006139 | | Narro | | | | | |
| Urinary tract carcinoma in situ | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004676 | | Narro | | | | | |
| Uterine cancer | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004677 | | Narro | | | | | |
| Uterine carcinoma in situ | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004679 | | Narro | | | | | |
| Uterine leiomyosarcoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006534 | | Narro | | | | | |
| Vaginal adenocarcinoma | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004688 | | Narro | | | | | |
| Vaginal cancer | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004688 | | Narro | | | | | |
| Vaginal cancer metastatic | 7 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004688 | | Narro | | | | | |
| Vaginal cancer recurrent | 9 | PT | w | A | 0 | Active | 10.0 | 20.0 |
| | 1004689 | | Narro | | | | | |
| Vaginal cancer stage 0 | 0 | PT | W | A | 0 | Active | 10.0 | 20.0 |


| | | | | Categor | Weigh | | Addition | Last Modified |
|---|---|---|---|---|---|---|---|---|
| | 1004689 | | Narro | | | | | |
| Vaginal cancer stage I | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004689 | | Narro | | | | | |
| Vaginal cancer stage II | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004689 | | Narro | | | | | |
| Vaginal cancer stage III | 3 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004689 | | Narro | | | | | |
| Vaginal cancer stage IVA | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004689 | | Narro | | | | | |
| Vaginal cancer stage IVB | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004774 | | Narro | | | | | |
| Vulval cancer | 1 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004774 | | Narro | | | | | |
| Vulval cancer metastatic | 2 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004774 | | Narro | | | | | |
| Vulval cancer recurrent | 4 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004774 | | Narro | | | | | |
| Vulval cancer stage 0 | 5 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004774 | | Narro | | | | | |
| Vulval cancer stage I | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004774 | | Narro | | | | | |
| Vulval cancer stage II | 7 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004774 | | Narro | | | | | |
| Vulval cancer stage III | 8 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1004774 | | Narro | | | | | |
| Vulval cancer stage IV | 9 | PT | W | A | 0 | Active | 10.0 | 20.0 |
| | 1006353 | | Narro | | | | | |
| Vulvar adenocarcinoma | 6 | PT | W | A | 0 | Active | 10.0 | 20.0 |


## 7.3. SMQ Terms for Pregnancy and Neonatal Topics

SMQ Export: 20.1 - English 1/8/2018 2:22:18 PM

Include Inactive PT: No

Term Attributes: Name, Code, Level, Scope, Category, Weight, Status, Addition Version, Last

Modified Version

Pregnancy and neonatal topics (SMQ) [20000185]

Congenital, familial and genetic disorders (SMQ) [20000077]


#### Foetal disorders (SMQ) [20000190]


# Lactation related topics (incl neonatal exposure through breast milk) (SMQ) [20000187] Functional lactation disorders (SMQ) [20000188]


Normal pregnancy conditions and outcomes (SMQ) [20000193]


|---|---|---|---|---|---|---|---|---|
| Alpha 1 foetoprotein normal | 10001782 | PT | Broad | A | 0 | Active | 14.0 | 14.0 |
| Breast engorgement | 10006240 | PT | Broad | A | 0 | Active | 14.0 | 14.0 |

Pregnancy, labour and delivery complications and risk factors (excl abortions and stillbirth) (SMQ) [20000186]


## 7.4. SMQ Terms for Hypertension

SMQ Export: 20.1 - English 1/8/2018 2:15:07 PM

Include Inactive PT: No

Term Attributes: Name, Code, Level, Scope, Category, Weight, Status, Addition Version, Last Modified Version

Hypertension (SMQ) [20000147]


# 7.5. List of Per-Protocol Chemotherapy Regimens in Preferred Term


| Agent Name in Preferred Term |
|------------------------------------------|
| ALTRETAMINE |
| ANETUMAB RAVTANSINE |
| ANTINEOPLASTIC AGENTS |
| BEVACIZUMAB |
| BEVACIZUMAB W/CARBOPLATIN* |
| CAPECITABINE |
| CARBOPLATIN* |
| CARBOPLATIN W/GEMCITABINE* |
| CARBOPLATIN W/GEMCITABINE HYDROCHLORIDE* |
| CARBOPLATIN W/PACLITAXEL* |
| CISPLATIN* |
| CISPLATIN W/DOCETAXEL* |
| CISPLATIN W/GEMCITABINE HYDROCHLORIDE* |
| CISPLATIN W/PACLITAXEL* |
| CYCLOPHOSPHAMIDE |
| DECITABINE |
| DOCETAXEL |
| DOXORUBICIN |
| DOXORUBICIN HYDROCHLORIDE |
| ETOPOSIDE |
| GEMCITABINE |
| GEMCITABINE HYDROCHLORIDE |
| IFOSFAMIDE |
| INVESTIGATIONAL DRUG |
| IRINOTECAN |
| IXABEPILONE |
| LIPOSOMAL DOXORUBICIN HYDROCHLORIDE |
| LURBINECTEDIN |
| MELPHALAN |
| METHOTREXATE |
| NINTEDANIB |
| NIRAPARIB |
| OLAPARIB |
| OMEPRAZOLE |
| OTHER ANTINEOPLASTIC AGENTS |
| OXALIPLATIN* |
| PACLITAXEL |
| PACLITAXEL ALBUMIN |


| Agent Name in Preferred Term |
|-----------------------------------------------|
| PACLITAXEL POLIGLUMEX |
| PACLITAXEL W/CARBOPLATIN* |
| PAZOPANIB |
| PEGYLATED LIPOSOMAL DOXORUBICIN |
| PEGYLATED LIPOSOMAL DOXORUBICIN HYDROCHLORIDE |
| PEMETREXED |
| PEMETREXED DISODIUM |
| PLATINUM COMPOUNDS* |
| PRALATREXATE |
| RUCAPARIB |
| TAXANES |
| TOPOTECAN |
| TRABECTEDIN |
| TRASTUZUMAB EMTANSINE |
| VELIPARIB |
| VINORELBINE |
| VINORELBINE TARTRATE |

<sup>\*</sup> Denotes platinum-based therapies.


### 8. STATISTICAL OUTPUT SHELLS

The list of statistical output and corresponding table/figure/listing shells are provided in a separate document.


#### 9. **REVISION HISTOR**

• The efficacy analyses were revised between versions 2.0 and 3.0 of the SAP in order to ensure consistency with the revised Protocol v3.2. Table, figure, and listing shells were modified to account for the revised analyses.

